CLINICAL TRIAL: NCT03653507
Title: A Phase 3, Global, Multi-Center, Double-Blind, Randomized, Efficacy Study of Zolbetuximab (IMAB362) Plus CAPOX Compared With Placebo Plus CAPOX as First-line Treatment of Subjects With Claudin (CLDN) 18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: A Study of Zolbetuximab (IMAB362) Plus CAPOX Compared With Placebo Plus CAPOX as First-line Treatment of Subjects With Claudin (CLDN) 18.2-positive, HER2-negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma (GLOW).
Acronym: GLOW
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8951-CL-0302; 2018-000519-26 (EudraCT Number); CTR20190261 (Registry Identifier: ChinaDrugTrials.org.cn); jRCT2080224166 (Registry Identifier: jRCT); 2024-511648-16-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06048081 (Available)
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma or Cancer; Locally Advanced Unresectable Gastric Adenocarcinoma or Cancer; Metastatic Gastric Adenocarcinoma or Cancer; Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: CLDN 18.2; gastroesophageal junction cancer; adenocarcinoma; IMAB362; oxaliplatin; HER2; claudiximab; capecitabine; gastric cancer; HER2 Negative; zolbetuximab
MeSH Terms: conditions — Adenocarcinoma; Neoplasms; Stomach Neoplasms | interventions — zolbetuximab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zolbetuximab plus CAPOX (Experimental): Participants received an IV infusion (as a minimum of 2-hour infusion) of zolbetuximab at a loading dose of 800 mg/m^2 on C1D1 followed by subsequent doses of 600 mg/m^2 every 3 weeks starting from C1D22 until participant meets study treatment discontinuation criteria. Participants also received up to 8 treatments of CAPOX. Oxaliplatin was administered 130 mg/m^2 IV on day 1 of each cycle over 2 hours for a maximum of 8 treatments; Capecitabine was administered orally at 1000 mg/m^2 twice daily (bid) on days 1 through 14 of each cycle until the participant met study treatment discontinuation criteria. After a maximum of 8 treatments of oxaliplatin, participants may have continued to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the participant met study treatment discontinuation criteria. Each cycle was approximately 21 days.
  Interventions: Drug: zolbetuximab; Drug: oxaliplatin; Drug: capecitabine
- Placebo plus CAPOX (Placebo Comparator): Participants received an IV infusion (as a minimum of 2-hour infusion) of placebo matched to zolbetuximab on C1D1 followed by subsequent doses every 3 weeks starting from C1D22 until participant meets study treatment discontinuation criteria. Participants also received up to 8 treatments of CAPOX. Oxaliplatin was administered 130 mg/m^2 IV on day 1 of each cycle over 2 hours for a maximum of 8 treatments; Capecitabine was administered orally at 1000 mg/m^2 bid on days 1 through 14 of each cycle until the participant met study treatment discontinuation criteria. After a maximum of 8 treatments of oxaliplatin, participants may have continued to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the participant met study treatment discontinuation criteria. Each cycle was approximately 21 days.
  Interventions: Drug: oxaliplatin; Drug: capecitabine; Drug: placebo

INTERVENTIONS:
Drug: zolbetuximab — Zolbetuximab were administered as a minimum 2-hour IV infusion.
  Other Names: IMAB362
  Arms: Zolbetuximab plus CAPOX
Drug: oxaliplatin — Oxaliplatin were administered as a 2-hour IV infusion.
Drug: capecitabine — Capecitabine were administered orally twice daily (bid).
Drug: placebo — Placebo were administered as a minimum 2-hour IV infusion.
  Arms: Placebo plus CAPOX

SUMMARY:
Zolbetuximab is being studied in people with cancer in and around the stomach or where the food pipe (esophagus) joins the stomach, called GEJ cancer. Most people with this type of cancer have a protein called Claudin 18.2 in their tumor. Zolbetuximab is thought to work by attaching to the Claudin 18.2 protein in their tumor, which switches on the body's immune system to attack the tumor.

There is an unmet medical need to treat people with advanced stomach cancer or GEJ cancer. This study will give more information about how well zolbetuximab works when given with chemotherapy in adults with advanced stomach cancer or GEJ cancer. In this study, adults with advanced stomach cancer or GEJ cancer will either be given zolbetuximab with chemotherapy or a placebo with chemotherapy. A placebo looks like zolbetuximab but doesn't have any medicine in it. Zolbetuximab with chemotherapy has already been approved to treat stomach cancer and GEJ cancer in some countries. This study is being done in countries where zolbetuximab has not yet been approved for use. If zolbetuximab becomes approved for use in those countries taking part in this study, the people taking part in those countries will leave this study and receive licensed zolbetuximab.

The main aim(s) of the study is(are) to determine the efficacy of zolbetuximab combined with chemotherapy compared to a placebo combined with chemotherapy in treating adults with Claudin 18.2-positive, HER2-negative, locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma.

Adults with locally advanced unresectable or metastatic stomach cancer or GEJ cancer can take part. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body. A tumor sample of their cancer will also have the Claudin 18.2 protein. They may have been previously treated with certain standard therapies but have not been treated with chemotherapy for their cancer. People cannot take part if they need to take medicines to suppress their immune system, have blockages or bleeding in their gut, have specific uncontrollable cancers such as symptomatic or untreated cancers in the nervous system, or have a specific heart condition, or infections.

The study treatments are either zolbetuximab with chemotherapy or placebo with chemotherapy. People who take part will receive just one of the treatments by chance. Study treatment will be double-blinded. That means that the people in the study and the study doctors will not know who takes which of the study treatments. Study treatment will be given in cycles. The study treatment is given to people slowly through a tube into a vein. This is called an infusion. The chemotherapy is called CAPOX (capecitabine and oxaliplatin) and will be given as an infusion and also as tablets. People will have 1 infusion of either zolbetuximab or placebo together with oxaliplatin chemotherapy in 3-week (21-day) cycles. People will also take 1 tablet of capecitabine (chemotherapy) twice a day for the first 2 weeks (14 days) of each cycle. People may receive zolbetuximab or placebo until their cancer worsens, they cannot tolerate the treatment, or they need to start another cancer treatment. People will receive CAPOX for up to about 6 months (8 treatment cycles). After the 6 months, people may receive capecitabine chemotherapy only, until their cancer worsens, they cannot tolerate the study treatment, or they need to start another cancer treatment. People will visit the clinic on certain days during their treatment. The study doctors will check if people had any medical problems from zolbetuximab or the other study treatments. Also, people in the study will have health checks. On some visits, they will have scans to check for any changes in their cancer. People will have the option of giving a tumor sample after their study treatment has finished. People will visit the clinic within 7 days after they stop their study treatment. People will be asked about any medical problems and will have a health check. People who start treatment with licensed zolbetuximab will not need to attend the clinic for further visits and will receive standard of care health checks. People who continue study treatment will visit the clinic at 1 and 3 months after they stop their study treatment. They will continue to have scans every 9 or 12 weeks to check for any changes in their cancer. They will have telephone health checks every 3 months. The number of visits and checks done at each visit will depend on the health of each person and whether they completed their treatment or not.

DETAILED DESCRIPTION:
After the marketing approval in Japan on 26 Mar 2024, this study continued as "post marketing clinical study" in Japan. In the rest of the countries which participated in this study, this study continued as clinical study.

ELIGIBILITY:
Inclusion Criteria:

* A female subject is eligible to participate if she is not pregnant (negative serum pregnancy test at screening; female subjects with elevated serum beta human chorionic gonadotropin (βhCG) and a demonstrated non-pregnant status through additional testing are eligible) and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study treatment administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs.
* A male subject with female partner(s) of childbearing potential:

  * must agree to use contraception during the treatment period and for 6 months after the final study treatment administration.
* A male subject must not donate sperm during the treatment period and for 6 months after the final study treatment administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study treatment administration.
* Subject has histologically confirmed diagnosis of Gastric or GEJ adenocarcinoma.
* Subject has radiologically confirmed locally advanced unresectable or metastatic disease within 28 days prior to randomization.
* Subject has radiologically evaluable disease (measurable and/or non-measurable disease according to RECIST 1.1), per local assessment, ≤ 28 days prior to randomization. For subjects with only 1 evaluable lesion and prior radiotherapy ≤ 3 months before randomization, the lesion must either be outside the field of prior radiotherapy or have documented progression following radiation therapy.
* Subject's tumor expresses CLDN18.2 in ≥ 75% of tumor cells demonstrating moderate to strong membranous staining as determined by central IHC testing.
* Subject has a HER2-negative tumor as determined by local or central testing on a gastric or GEJ tumor specimen. (Unique to China: Subject has a known HER2-negative gastric or GEJ tumor.)
* Subject has ECOG performance status 0 or 1.
* Subject has predicted life expectancy ≥ 12 weeks.
* Subject must meet all of the following criteria based on the centrally or locally analyzed laboratory tests collected within 14 days prior to randomization. In the case of multiple sample collections within this period, the most recent sample collection with available results should be used to determine eligibility.

  * Hemoglobin (Hb) ≥ 9 g/dl. Subjects requiring transfusions are eligible if they have a post-transfusion Hgb ≥ 9 g/dL.
  * Absolute Neutrophil Count (ANC) ≥ 1.5x10^9/L
  * Platelets ≥ 100x10^9/L
  * Albumin ≥ 2.5 g/dL
  * Total Bilirubin ≤ 1.5 x upper limit of normal (ULN) without liver metastases (or < 3.0 x ULN if liver metastases are present)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN without liver metastases (or ≤ 5 x ULN if liver metastases are present)
  * Estimated creatinine clearance ≥ 30 mL/min
  * Prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time (PTT) ≤ 1.5 x ULN (except for subjects receiving anticoagulation therapy)

Exclusion Criteria:

* Subject has received prior systemic chemotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma. However, subject may have received either neo-adjuvant or adjuvant chemotherapy, immunotherapy or other systemic anticancer therapies as long as it was completed at least 6 months prior to randomization.
* Subject has received radiotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma ≤ 14 days prior to randomization and has not recovered from any related toxicity.
* Subject has received treatment with herbal medications or other treatments that have known antitumor activity within 28 days prior to randomization.
* Subject has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to randomization. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone), receiving a single dose of systemic corticosteroids or receiving systemic corticosteroids as premedication for radiologic imaging contrast use are allowed.
* Subject has received other investigational agents or devices within 28 days prior to randomization.
* Subject has prior severe allergic reaction or intolerance to known ingredients of zolbetuximab or other monoclonal antibodies, including humanized or chimeric antibodies.
* Subject has known immediate or delayed hypersensitivity, intolerance or contraindication to any component of study treatment.
* Subject has prior severe allergic reaction or intolerance to any component of CAPOX.
* Subject has known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Subject has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting.
* Subject has significant gastric bleeding and/or untreated gastric ulcers that exclude the subject from participation.
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection or known active hepatitis B (positive hepatitis B surface antigen (HBs Ag)) or C infection. NOTE: Screening for these infections should be conducted per local requirements.

  * For subjects who are negative for HBs Ag, but hepatitis B core antibody (HBc Ab) positive, an HB deoxyribonucleic acid (DNA) test will be performed and if positive, the subject will be excluded.
  * Subjects with positive hepatitis C virus (HCV) serology, but negative HCV ribonucleic acid (RNA) test are eligible.
  * Subjects treated for HCV with undetectable viral load results are eligible.
* Subject has an active autoimmune disease that has required systemic treatment within the past 3 months prior to randomization.
* Subject has active infection requiring systemic therapy that has not completely resolved within 7 days prior to randomization.
* Subject has significant cardiovascular disease, including any of the following:

  * Congestive heart failure (defined as New York Heart Association Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, stenting, coronary artery bypass graft, cerebrovascular accident (CVA) or hypertensive crisis within 6 months prior to randomization.
  * History of clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation or Torsades de Pointes
  * QTc interval > 450 msec for male subjects; QTc interval > 470 msec for female subjects
  * History or family history of congenital long QT syndrome
  * Cardiac arrhythmias requiring anti-arrhythmic medications (Subject with rate controlled atrial fibrillation for > 1 month prior to randomization are eligible).
* Subject has a history of central nervous system (CNS) metastases and/or carcinomatous meningitis from gastric/GEJ cancer..
* Subject has known peripheral sensory neuropathy > grade 1 unless the absence of deep tendon reflexes is the sole neurological abnormality.
* Subject has had a major surgical procedure ≤ 28 days prior to randomization.

  * Subject is without complete recovery from a major surgical procedure ≤ 14 days prior to randomization.
* Subject has psychiatric illness or social situations that would preclude study compliance.
* Subject has another malignancy for which treatment is required.
* Subject has any concurrent disease, infection, or co-morbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (165):
- United States (11):
  - Pacific Cancer Care, Monterey, California
  - University of Kansas Cancer Center and Medical Pavilion, Fairway, Kansas
  - Ochsner Clinic CCOP, New Orleans, Louisiana
  - New Mexico Oncology Hematology, Albuquerque, New Mexico
  - Weill Cornell Medical College (WCMC), New York, New York
  - Montefiore Medical Center (MMC), The Bronx, New York
  - Prisma Health Cancer Institute, Boiling Springs, South Carolina
  - Parkland Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Cancer Center and Institute of Academic Medicine - Oncology, Houston, Texas
  - Utah Cancer Specialist, Salt Lake City, Utah
- Argentina (6):
  - Site AR54009, Buenos Aires
  - Site GB44005, Northwood
  - Site AR54006, Pergamino
  - Site AR54001, San Miguel de Tucumán
  - Site AR54004, San Miguel de Tucumán
  - Site AR54003, Viedma
- Canada (3):
  - Site CA15003, Chicoutimi, Quebec
  - Site CA15002, Rimouski, Quebec
  - Site CA15004, Calgary
- China (41):
  - Site CN86034, Fuzhou, Fujian
  - Site CN86037, Fuzhou, Fujian
  - Site CN86032, Haikou, Hainan
  - Site CN86012, Zhengzhou, Henan
  - Site CN86029, Changsha, Hunan
  - Site CN86043, Hengyang, Hunan
  - Site CN86027, Suzhou, Jiangsu
  - Site CN86046, Wuxi, Jiangsu
  - Site CN86007, Hangzhou, Zhejiang
  - Site CN86044, Baoding
  - Site CN86035, Beijing
  - Site CN86050, Beijing
  - Site CN86025, Bengbu
  - Site CN86002, Changchun
  - Site CN86049, Changchun
  - Site CN86053, Changchun
  - Site CN86021, Changzhou
  - Site CN86039, Chengdu
  - Site CN86052, Dalian
  - Site CN86054, Dalian
  - Site CN86015, Fuzhou
  - Site CN86001, Guangzhou
  - Site CN86042, Guangzhou
  - Site CN86051, Haebrin
  - Site CN86036, Hangzhou
  - Site CN86038, Linyi
  - Site CN86016, Nanjing
  - Site CN86045, Nanning
  - Site CN86014, Shanghai
  - Site CN86026, Shantou
  - Site CN86047, Shenyang
  - Site CN86017, Shijiazhuang
  - Site CN86009, Tianjin
  - Site CN86040, Tianjin
  - Site CN86031, Ürümqi
  - Site CN86004, Wuhan
  - Site CN86005, Wuhan
  - Site CN86013, Xi'an
  - Site CN86030, Xiamen
  - Site CN86011, Xuzhou
  - Site CN86024, Zhengzhou
- Croatia (3):
  - Site HR38501, Varaždin
  - Site HR38502, Zagreb
  - Site HR38503, Zagreb
- Greece (7):
  - Site GR30001, Athens
  - Site GR30004, Heraklion
  - Site GR30003, Larissa
  - Site GR30005, Neo Faliro, Piraeus
  - Site GR30007, Rio Patras
  - Site GR30002, Thessaloniki
  - Site GR3006, Thessaloniki
- Ireland (2):
  - Site IE35301, Dublin
  - Site IE35302, Dublin
- Japan (12):
  - Site JP81007, Fukuoka, Fukuoka
  - Site JP81008, Akashi, Hyōgo
  - Site JP81003, Kawasaki, Kanagawa
  - Site JP81001, Yokohama, Kanagawa
  - Site JP81010, Suita, Osaka
  - Site JP81005, Utsunomiya, Tochigi
  - Site JP81002, Chiba
  - Site JP81006, Kashiwa
  - Site JP81004, Kita-gun
  - Site JP81012, Kōtoku
  - Site JP81009, Matsuyama
  - Site JP81011, Tsukiji
- Malaysia (5):
  - Site MY60001, George Town
  - Site MY60004, Kota Kinabalu
  - Site MY60002, Kuala Lumpur
  - Site MY60003, Kuala Lumpur
  - Site MY60005, Kuala Lumpur
- Netherlands (2):
  - Site NL31004, Groningen
  - Site NL31003, Tilburg
- Portugal (10):
  - Site PT35109, Braga
  - Site PT35110, Coimbra
  - Site PT35111, Guimarães
  - Site PT35102, Lisbon
  - Site PT35106, Lisbon
  - Site PT35105, Porto
  - Site PT35108, Porto
  - Site PT35104, Santa Maria da Feira
  - Site PT35101, Setúbal
  - Site PT35107, Vila Real
- Romania (8):
  - Site RO40002, Bucharest
  - Site RO40005, Cluj-Napoca
  - Site RO40007, Cluj-Napoca
  - Site RO40003, Craiova
  - Site RO40004, Floreşti
  - Site RO40001, Iași
  - Site RO40006, Iași
  - Site RO40008, Timișoara
- South Korea (13):
  - Site KR82002, Daegu
  - Site KR82006, Goyang-si
  - Site KR82007, Gyeonggi-do
  - Site KR82014, Incheon
  - Site KR82008, Jeollanam-do
  - Site KR82010, Jeonju
  - Site KR82011, Seongnam-si
  - Site KR82001, Seoul
  - Site KR82003, Seoul
  - Site KR82012, Seoul
  - Site KR82013, Seoul
  - Site KR82015, Seoul
  - Site KR82009, Suwon
- Spain (13):
  - Site ES34005, A Coruña
  - Site ES34006, Barcelona
  - Site ES34009, Barcelona
  - Site ES34010, Barcelona
  - Site ES34001, Elche
  - Site ES34002, Madrid
  - Site ES34003, Madrid
  - Site ES34008, Madrid
  - Site ES34013, Madrid
  - Site ES34011, Málaga
  - Site ES34004, Pamplona
  - Site ES34007, Valencia
  - Site ES34012, Valencia
- Taiwan (4):
  - Site TW88602, Kaohsiung City
  - Site TW88603, Taichung
  - Site TW88604, Taipei
  - Site TW88605, Tianan
- Thailand (11):
  - Site TH66002, Bangkok
  - Site TH66005, Bangkok
  - Site TH66007, Bangkok
  - Site TH66009, Bangkok
  - Site TH66011, Laksi
  - Site TH66001, Muang
  - Site TH66003, Muang
  - Site TH66006, Pathum Thani
  - Site TH66010, Pathumwan
  - Site TH66004, Songkhla
  - Site TH66008, Vadhana
- Turkey (Türkiye) (11):
  - Site TR90008, Pendik, Istanbul
  - Site TR90003, Atakum
  - Site TR90004, Balcalı
  - Site TR90012, Bornova
  - Site TR90001, Bursa
  - Site TR90002, Istanbul
  - Site TR90010, Istanbul
  - Site TR90015, Istanbul
  - Site TR90007, Konya
  - Site TR90013, Konyaalti
  - Site TR90011, Malatya
- United Kingdom (3):
  - Site GB44002, Bristol
  - Site GB44004, Cardiff
  - Site GB44001, London

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Shitara K, Shah MA, Lordick F, Bang YJ, Ilson D, Van Cutsem E, Enzinger P, Kim SS, Klempner SJ, Moran D, Park JW, Bhattacharya P, Ajani JA, Xu RH. Zolbetuximab plus chemotherapy for locally advanced unresectable or metastatic stomach or gastroesophageal junction cancers: a plain language summary. Future Oncol. 2024;20(26):1861-1877. doi: 10.1080/14796694.2024.2342107. Epub 2024 May 24. PMID 38861294
- [Derived] Shah MA, Shitara K, Ajani JA, Bang YJ, Enzinger P, Ilson D, Lordick F, Van Cutsem E, Gallego Plazas J, Huang J, Shen L, Oh SC, Sunpaweravong P, Soo Hoo HF, Turk HM, Oh M, Park JW, Moran D, Bhattacharya P, Arozullah A, Xu RH. Zolbetuximab plus CAPOX in CLDN18.2-positive gastric or gastroesophageal junction adenocarcinoma: the randomized, phase 3 GLOW trial. Nat Med. 2023 Aug;29(8):2133-2141. doi: 10.1038/s41591-023-02465-7. Epub 2023 Jul 31. PMID 37524953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with claudin (CLDN)18.2-positive, human epidermal growth factor receptor 2 (HER2) -negative locally advanced unresectable or metastatic gastric and gastroesophageal junction (GEJ) adenocarcinoma
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study. Randomization was stratified by region (Asia vs Non-Asia), number of organs with metastatic sites (0 to 2 vs ≥ 3) and prior gastrectomy (Yes or No)
Groups:
- CAPOX+ Zolbetuximab: Participants received an intravenous (IV) infusion (as a minimum of 2-hour infusion) of zolbetuximab at a loading dose of 800 milligrams per square meter (mg/m^2) on cycle 1 day 1 (C1D1) followed by subsequent doses of 600 mg/m^2 every 3 weeks starting from C2D1 until participant met study treatment discontinuation criteria. Participants also received up to 8 treatments of capecitabine and oxaliplatin (CAPOX) treatment. Oxaliplatin was administered 130 mg/m^2 IV on day 1 of each cycle over 2 hours for a maximum of 8 treatments; Capecitabine was administered orally at 1000 mg/m^2 twice daily (bid) on days 1 through 14 of each cycle until the participant met study treatment discontinuation criteria. After a maximum of 8 treatments of oxaliplatin, participants may have continued to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the participant met study treatment discontinuation criteria. Each cycle was approximately 21 days.
- CAPOX+ Placebo: Participants received an IV infusion (as a minimum of 2-hour infusion) of placebo matched to zolbetuximab on C1D1 followed by subsequent doses every 3 weeks starting from C2D1 until participant met study treatment discontinuation criteria. Participants also received up to 8 treatments of CAPOX. Oxaliplatin was administered 130 mg/m^2 IV on day 1 of each cycle over 2 hours for a maximum of 8 treatments; Capecitabine was administered orally at 1000 mg/m^2 bid on days 1 through 14 of each cycle until the participant met study treatment discontinuation criteria. After a maximum of 8 treatments of oxaliplatin, participants may have continued to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the participant met study treatment discontinuation criteria. Each cycle was approximately 21 days.
Period: Overall Study
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Started | 254 | 249
Completed | 9 | 2
Not Completed | 245 | 247
Not completed — Miscellaneous | 28 | 19
Not completed — Withdrawal by Subject | 37 | 22
Not completed — Protocol Deviation | 2 | 1
Not completed — Progressive disease | 117 | 168
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 25 | 22
Not completed — Adverse Event | 35 | 14

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized to 1 of the treatment arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo | Total
Number analyzed (Participants) | 254 | 253 | 507
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (12.1) | 56.7 (13) | 57.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 97 | 192
  Male | 159 | 156 | 315
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 242 | 241 | 483
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 158 | 158 | 316
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 94 | 90 | 184
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region (Asia vs Non-Asia) [Number; unit: Participants]
  Asia | 157 | 158 | 315
  Non-Asia | 97 | 95 | 192
Number of organs with metastatic sites [Number; unit: Participants]
  0-2 metastatic sites | 189 | 188 | 377
  >=3 metastatic sites | 65 | 65 | 130
Prior Gastrectomy [Number; unit: Participants]
  Yes | 75 | 75 | 150
  No | 179 | 178 | 357

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the date of radiological progressive disease (PD) (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 by independent review committee [IRC]) or death from any cause, whichever was earliest. PD was defined as development of new, or progression of existing metastases to the primary cancer under the study. Kaplan-Meier estimates was used.
Time Frame: From the date of randomization until 61 months and 12 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- CAPOX+ Zolbetuximab: Participants received an intravenous (IV) infusion (as a minimum of 2-hour infusion) of zolbetuximab at a loading dose of 800 milligrams per square meter (mg/m^2) on cycle 1 day 1 (C1D1) followed by subsequent doses of 600 mg/m^2 every 3 weeks starting from C2D1 until participant met study treatment discontinuation criteria. Participants also received up to 8 treatments of capecitabine and oxaliplatin (CAPOX) treatment. Oxaliplatin was administered 130 mg/m^2 IV on day 1 of each cycle over 2 hours for a maximum of 8 treatments; Capecitabine was administered orally at 1000 mg/m^2 twice daily (bid) on days 1 through 14 of each cycle until the participant met study treatment discontinuation criteria. After a maximum of 8 treatments of oxaliplatin, participants may have continued to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the participant met study treatment discontinuation criteria. Each cycle was approximately 21
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 254 | 253
Months | 8.21 [7.26 to 8.84] | 6.80 [6.14 to 8.08]
Statistical Analysis 1: Comparison: CAPOX+ Zolbetuximab; Test type: Superiority; p = 0.0005, Log Rank; Hazard Ratio (HR) = 0.689, 95% CI 2-sided [0.552 to 0.860] — Log-rank test stratified by:* Region (Asia vs Non-Asia), * Number of organs with metastatic sites (0 to 2 vs >= 3), * Prior gastrectomy (Yes or No)

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause. Kaplan-Meier estimates was used.
Time Frame: From the date of randomization until 61 months and 12 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 254 | 253
Months | 14.32 [12.09 to 16.39] | 12.16 [10.28 to 13.67]
Statistical Analysis 1: Comparison: CAPOX+ Zolbetuximab; Test type: Superiority; p = 0.0047, Log Rank; Hazard Ratio (HR) = 0.763, 95% CI 2-sided [0.622 to 0.936] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Confirmed Deterioration (TTCD) Using Physical Functioning as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core Questionnaire (EORTC QLQ-C30)
Description: TTCD: time from randomization to first clinically meaning full deterioration (CMFD) that was confirmed at the next scheduled visit. The EORTC-QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Most items are scored 1 ('not at all') to 4 ('very much') except for the items contributing to the global health status which are scored 1 ('very poor') to 7 ('excellent'). All raw domain scores are linearly transformed to a 0-100 scale with higher scores on symptoms indicate a worse health state. Clinically meaningful deterioration was defined if a participant's change from baseline (CFB) exceeded a pre-specified threshold (as per investigator's discretion) denoting a clinically meaningful change. Kaplan-Meier estimates was used.
Time Frame: From the date of randomization until 61 months and 12 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 254 | 253
Months | 7.95 [5.88 to 19.78] | 7.92 [6.47 to 11.30]
Statistical Analysis 1: Comparison: CAPOX+ Zolbetuximab; Test type: Superiority; p = 0.4654, Log Rank; Hazard Ratio (HR) = 1.012, 95% CI 2-sided [0.772 to 1.328] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Confirmed Deterioration (TTCD) Using Oesophago-gastric Questionnaire (OG25) on Abdominal Pain and Discomfort as Measured by EORTC QLQ-OG25 Plus STO22 Belching Subscale
Description: TTCD:time from randomization to first CMFD confirmed at next scheduled visit.OG25 evaluated gastric & gastroesophageal junction cancer-specific symptoms,had 25 items with 6 scales:dysphagia,eating restrictions,reflux,odynophagia,pain, discomfort,anxiety,and 10 single items:trouble with(taste, swallowing saliva, coughing, talking),eating in front of others,dry mouth,body image,choked when swallowing,weight loss and hair loss. STO22: gastric cancer quality of life questionnaire with 22 questions.For OG25 and STO22,items scored on(1:not at all; 2:a little, 3:quite a bit, 4:very much) and 1 question was "yes or no" for STO22.Linear transformation was used; score ranged from 0 to 100; higher score=better level of functioning or greater degree of symptoms. An item from STO22 instrument related to belching was used with OG25. CMFD: if participant's CFB exceeded pre-specified threshold (per investigator's discretion) denoting a clinically meaningful change. Kaplan-Meier estimates was used
Time Frame: From the date of randomization until 61 months and 12 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 254 | 253
Months | NA [28.16 to NA] — Data was not estimable because less than 50% of participants had event (data was estimated using KM and it requires at least 50% of event to be able to calculate time using KM. | 25.82 [18.46 to NA] — The lower bound of the confidence interval for the median survival time may not be estimable, even if the median itself can be calculated, in scenarios with significant early censoring and a limited number of events
Statistical Analysis 1: Comparison: CAPOX+ Zolbetuximab; Test type: Superiority; p = 0.4478, Log Rank; Hazard Ratio (HR) = 1.030, 95% CI 2-sided [0.673 to 1.577] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Confirmed Deterioration (TTCD) Using Global Health Status as Measured by EORTC QLQ-C30
Description: TTCD: time from randomization to first CMFD that was confirmed at the next scheduled visit.The EORTC-QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Most items are scored 1 ('not at all') to 4 ('very much') except for the items contributing to the global health status/QoL, which are scored 1 (very poor) to 7 (excellent). All raw domain scores are linearly transformed to a 0-100 scale with higher scores on symptoms indicate a worse health state. Clinically meaningful deterioration was defined if a participant's CFB exceeded a pre-specified threshold (as per investigator's discretion) denoting a clinically meaningful change. Kaplan-Meier estimates was used.
Time Frame: From the date of randomization until 61 months and 12 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 254 | 253
Months | 9.40 [7.36 to 24.80] | 7.49 [6.11 to 9.86]
Statistical Analysis 1: Comparison: CAPOX+ Zolbetuximab; Test type: Superiority; p = 0.1670, Log Rank; Hazard Ratio (HR) = 0.869, 95% CI 2-sided [0.655 to 1.153] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) as was assessed by IRC per RECIST 1.1. CR was defined as complete resolution of all attributable clinical symptoms and physical findings. PR was defined as partial resolution of at Least some of the clinical symptoms and physical findings.
Time Frame: From the date of randomization until 61 months and 12 days
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 254 | 253
Percentage of Participants | 42.5 [36.36 to 48.85] | 39.1 [33.08 to 45.44]
Statistical Analysis 1: Comparison: CAPOX+ Zolbetuximab; Test type: Superiority; p = 0.2219, Cochran-Mantel-Haenszel — Based on 1-sided Cochran-Mantel-Haenszel (CMH) test. Stratification factors were Region, Number of Metastatic Sites and Prior Gastrectomy

7. Secondary Outcome: Duration Of Response (DOR)
Description: DOR was defined as the time from the date of the first response (CR/PR) until the date of PD as assessed by IRC per RECIST 1.1 or date of death from any cause, whichever is earliest.CR was defined as complete resolution of all attributable clinical symptoms and physical findings. PR was defined as partial resolution of at Least some of the clinical symptoms and physical findings. PD was defined as development of new, or progression of existing metastases to the primary cancer under the study. Kaplan-Meier estimates was used.
Time Frame: From first response (CR/PR) until 61 months and 12 days
Population: FAS- All Objective Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 108 | 102
Months | 6.28 [5.39 to 8.28] | 6.08 [4.44 to 6.34]
Statistical Analysis 1: Comparison: CAPOX+ Zolbetuximab; Test type: Superiority; p = 0.0826, Log Rank; Hazard Ratio (HR) = 0.781, 95% CI 2-sided [0.552 to 1.105] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) is any untoward medical occurrence in a participant administered a study drug, and which does not have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.TEAE defined as an AE observed after starting administration of the study drug through 30 days after the last dose.
Time Frame: From first dose until 61 months and 12 days
Population: FAS
Measure: Number; unit: Participants
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 254 | 249
Participants | 251 [NA to NA] | 244 [NA to NA]

9. Secondary Outcome: Number of Participant With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG grades 0-5, where 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair and 5 = Dead.
Time Frame: Baseline, cycle (C) 1 day (D)1 through C60 D1
Population: FAS
Measure: Number; unit: Participants
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 253 | 250
Participants
  Baseline Score 0 | 108 | 108
  Baseline Score 1 | 145 | 142
  Baseline Score 2 | 0 | 0
  Baseline Score 3 | 0 | 0
  Baseline Score 4 | 0 | 0
  Baseline Score 5 | 0 | 0
  C2D1 Score 0: number analyzed (Participants) | 219 | 225
  C2D1 Score 0 | 85 | 97
  C2D1 Score 1: number analyzed (Participants) | 219 | 225
  C2D1 Score 1 | 129 | 126
  C2D1 Score 2: number analyzed (Participants) | 219 | 225
  C2D1 Score 2 | 5 | 2
  C2D1 Score 3: number analyzed (Participants) | 219 | 225
  C2D1 Score 3 | 0 | 0
  C2D1 Score 4: number analyzed (Participants) | 219 | 225
  C2D1 Score 4 | 0 | 0
  C2D1 Score 5: number analyzed (Participants) | 219 | 225
  C2D1 Score 5 | 0 | 0
  C3D1 Score 0: number analyzed (Participants) | 196 | 210
  C3D1 Score 0 | 80 | 91
  C3D1 Score 1: number analyzed (Participants) | 196 | 210
  C3D1 Score 1 | 116 | 117
  C3D1 Score 2: number analyzed (Participants) | 196 | 210
  C3D1 Score 2 | 0 | 2
  C3D1 Score 3: number analyzed (Participants) | 196 | 210
  C3D1 Score 3 | 0 | 0
  C3D1 Score 4: number analyzed (Participants) | 196 | 210
  C3D1 Score 4 | 0 | 0
  C3D1 Score 5: number analyzed (Participants) | 196 | 210
  C3D1 Score 5 | 0 | 0
  C4D1 Score 0: number analyzed (Participants) | 180 | 179
  C4D1 Score 0 | 74 | 79
  C4D1 Score 1: number analyzed (Participants) | 180 | 179
  C4D1 Score 1 | 106 | 98
  C4D1 Score 2: number analyzed (Participants) | 180 | 179
  C4D1 Score 2 | 0 | 2
  C4D1 Score 3: number analyzed (Participants) | 180 | 179
  C4D1 Score 3 | 0 | 0
  C4D1 Score 4: number analyzed (Participants) | 180 | 179
  C4D1 Score 4 | 0 | 0
  C4D1 Score 5: number analyzed (Participants) | 180 | 179
  C4D1 Score 5 | 0 | 0
  C5D1 Score 0: number analyzed (Participants) | 168 | 175
  C5D1 Score 0 | 68 | 75
  C5D1 Score 1: number analyzed (Participants) | 168 | 175
  C5D1 Score 1 | 98 | 98
  C5D1 Score 2: number analyzed (Participants) | 168 | 175
  C5D1 Score 2 | 2 | 2
  C5D1 Score 3: number analyzed (Participants) | 168 | 175
  C5D1 Score 3 | 0 | 0
  C5D1 Score 4: number analyzed (Participants) | 168 | 175
  C5D1 Score 4 | 0 | 0
  C5D1 Score 5: number analyzed (Participants) | 168 | 175
  C5D1 Score 5 | 0 | 0
  C6D1 Score 0: number analyzed (Participants) | 159 | 156
  C6D1 Score 0 | 71 | 72
  C6D1 Score 1: number analyzed (Participants) | 159 | 156
  C6D1 Score 1 | 86 | 80
  C6D1 Score 2: number analyzed (Participants) | 159 | 156
  C6D1 Score 2 | 2 | 3
  C6D1 Score 3: number analyzed (Participants) | 159 | 156
  C6D1 Score 3 | 0 | 1
  C6D1 Score 4: number analyzed (Participants) | 159 | 156
  C6D1 Score 4 | 0 | 0
  C6D1 Score 5: number analyzed (Participants) | 159 | 156
  C6D1 Score 5 | 0 | 0
  C7D1 Score 0: number analyzed (Participants) | 122 | 136
  C7D1 Score 0 | 52 | 60
  C7D1 Score 1: number analyzed (Participants) | 122 | 136
  C7D1 Score 1 | 67 | 76
  C7D1 Score 2: number analyzed (Participants) | 122 | 136
  C7D1 Score 2 | 2 | 0
  C7D1 Score 3: number analyzed (Participants) | 122 | 136
  C7D1 Score 3 | 1 | 0
  C7D1 Score 4: number analyzed (Participants) | 122 | 136
  C7D1 Score 4 | 0 | 0
  C7D1 Score 5: number analyzed (Participants) | 122 | 136
  C7D1 Score 5 | 0 | 0
  C8D1 Score 0: number analyzed (Participants) | 113 | 114
  C8D1 Score 0 | 49 | 44
  C8D1 Score 1: number analyzed (Participants) | 113 | 114
  C8D1 Score 1 | 63 | 70
  C8D1 Score 2: number analyzed (Participants) | 113 | 114
  C8D1 Score 2 | 1 | 0
  C8D1 Score 3: number analyzed (Participants) | 113 | 114
  C8D1 Score 3 | 0 | 0
  C8D1 Score 4: number analyzed (Participants) | 113 | 114
  C8D1 Score 4 | 0 | 0
  C8D1 Score 5: number analyzed (Participants) | 113 | 114
  C8D1 Score 5 | 0 | 0
  C9D1 Score 0: number analyzed (Participants) | 106 | 106
  C9D1 Score 0 | 47 | 47
  C9D1 Score 1: number analyzed (Participants) | 106 | 106
  C9D1 Score 1 | 57 | 59
  C9D1 Score 2: number analyzed (Participants) | 106 | 106
  C9D1 Score 2 | 2 | 0
  C9D1 Score 3: number analyzed (Participants) | 106 | 106
  C9D1 Score 3 | 0 | 0
  C9D1 Score 4: number analyzed (Participants) | 106 | 106
  C9D1 Score 4 | 0 | 0
  C9D1 Score 5: number analyzed (Participants) | 106 | 106
  C9D1 Score 5 | 0 | 0
  C10D1 Score 0: number analyzed (Participants) | 88 | 84
  C10D1 Score 0 | 39 | 40
  C10D1 Score 1: number analyzed (Participants) | 88 | 84
  C10D1 Score 1 | 47 | 44
  C10D1 Score 2: number analyzed (Participants) | 88 | 84
  C10D1 Score 2 | 2 | 0
  C10D1 Score 3: number analyzed (Participants) | 88 | 84
  C10D1 Score 3 | 0 | 0
  C10D1 Score 4: number analyzed (Participants) | 88 | 84
  C10D1 Score 4 | 0 | 0
  C10D1 Score 5: number analyzed (Participants) | 88 | 84
  C10D1 Score 5 | 0 | 0
  C11D1 Score 0: number analyzed (Participants) | 86 | 77
  C11D1 Score 0 | 41 | 34
  C11D1 Score 1: number analyzed (Participants) | 86 | 77
  C11D1 Score 1 | 45 | 43
  C11D1 Score 2: number analyzed (Participants) | 86 | 77
  C11D1 Score 2 | 0 | 0
  C11D1 Score 3: number analyzed (Participants) | 86 | 77
  C11D1 Score 3 | 0 | 0
  C11D1 Score 4: number analyzed (Participants) | 86 | 77
  C11D1 Score 4 | 0 | 0
  C11D1 Score 5: number analyzed (Participants) | 86 | 77
  C11D1 Score 5 | 0 | 0
  C12D1 Score 0: number analyzed (Participants) | 77 | 65
  C12D1 Score 0 | 39 | 29
  C12D1 Score 1: number analyzed (Participants) | 77 | 65
  C12D1 Score 1 | 38 | 36
  C12D1 Score 2: number analyzed (Participants) | 77 | 65
  C12D1 Score 2 | 0 | 0
  C12D1 Score 3: number analyzed (Participants) | 77 | 65
  C12D1 Score 3 | 0 | 0
  C12D1 Score 4: number analyzed (Participants) | 77 | 65
  C12D1 Score 4 | 0 | 0
  C12D1 Score 5: number analyzed (Participants) | 77 | 65
  C12D1 Score 5 | 0 | 0
  C13D1 Score 0: number analyzed (Participants) | 67 | 54
  C13D1 Score 0 | 33 | 24
  C13D1 Score 1: number analyzed (Participants) | 67 | 54
  C13D1 Score 1 | 34 | 30
  C13D1 Score 2: number analyzed (Participants) | 67 | 54
  C13D1 Score 2 | 0 | 0
  C13D1 Score 3: number analyzed (Participants) | 67 | 54
  C13D1 Score 3 | 0 | 0
  C13D1 Score 4: number analyzed (Participants) | 67 | 54
  C13D1 Score 4 | 0 | 0
  C13D1 Score 5: number analyzed (Participants) | 67 | 54
  C13D1 Score 5 | 0 | 0
  C14D1 Score 0: number analyzed (Participants) | 64 | 48
  C14D1 Score 0 | 32 | 20
  C14D1 Score 1: number analyzed (Participants) | 64 | 48
  C14D1 Score 1 | 32 | 28
  C14D1 Score 2: number analyzed (Participants) | 64 | 48
  C14D1 Score 2 | 0 | 0
  C14D1 Score 3: number analyzed (Participants) | 64 | 48
  C14D1 Score 3 | 0 | 0
  C14D1 Score 4: number analyzed (Participants) | 64 | 48
  C14D1 Score 4 | 0 | 0
  C14D1 Score 5: number analyzed (Participants) | 64 | 48
  C14D1 Score 5 | 0 | 0
  C15D1 Score 0: number analyzed (Participants) | 54 | 41
  C15D1 Score 0 | 24 | 16
  C15D1 Score 1: number analyzed (Participants) | 54 | 41
  C15D1 Score 1 | 30 | 25
  C15D1 Score 2: number analyzed (Participants) | 54 | 41
  C15D1 Score 2 | 0 | 0
  C15D1 Score 3: number analyzed (Participants) | 54 | 41
  C15D1 Score 3 | 0 | 0
  C15D1 Score 4: number analyzed (Participants) | 54 | 41
  C15D1 Score 4 | 0 | 0
  C15D1 Score 5: number analyzed (Participants) | 54 | 41
  C15D1 Score 5 | 0 | 0
  C16D1 Score 0: number analyzed (Participants) | 51 | 35
  C16D1 Score 0 | 23 | 18
  C16D1 Score 1: number analyzed (Participants) | 51 | 35
  C16D1 Score 1 | 27 | 17
  C16D1 Score 2: number analyzed (Participants) | 51 | 35
  C16D1 Score 2 | 1 | 0
  C16D1 Score 3: number analyzed (Participants) | 51 | 35
  C16D1 Score 3 | 0 | 0
  C16D1 Score 4: number analyzed (Participants) | 51 | 35
  C16D1 Score 4 | 0 | 0
  C16D1 Score 5: number analyzed (Participants) | 51 | 35
  C16D1 Score 5 | 0 | 0
  C17D1 Score 0: number analyzed (Participants) | 47 | 29
  C17D1 Score 0 | 22 | 17
  C17D1 Score 1: number analyzed (Participants) | 47 | 29
  C17D1 Score 1 | 24 | 12
  C17D1 Score 2: number analyzed (Participants) | 47 | 29
  C17D1 Score 2 | 1 | 0
  C17D1 Score 3: number analyzed (Participants) | 47 | 29
  C17D1 Score 3 | 0 | 0
  C17D1 Score 4: number analyzed (Participants) | 47 | 29
  C17D1 Score 4 | 0 | 0
  C17D1 Score 5: number analyzed (Participants) | 47 | 29
  C17D1 Score 5 | 0 | 0
  C18D1 Score 0: number analyzed (Participants) | 47 | 24
  C18D1 Score 0 | 26 | 16
  C18D1 Score 1: number analyzed (Participants) | 47 | 24
  C18D1 Score 1 | 21 | 8
  C18D1 Score 2: number analyzed (Participants) | 47 | 24
  C18D1 Score 2 | 0 | 0
  C18D1 Score 3: number analyzed (Participants) | 47 | 24
  C18D1 Score 3 | 0 | 0
  C18D1 Score 4: number analyzed (Participants) | 47 | 24
  C18D1 Score 4 | 0 | 0
  C18D1 Score 5: number analyzed (Participants) | 47 | 24
  C18D1 Score 5 | 0 | 0
  C19D1 Score 0: number analyzed (Participants) | 43 | 22
  C19D1 Score 0 | 22 | 14
  C19D1 Score 1: number analyzed (Participants) | 43 | 22
  C19D1 Score 1 | 21 | 8
  C19D1 Score 2: number analyzed (Participants) | 43 | 22
  C19D1 Score 2 | 0 | 0
  C19D1 Score 3: number analyzed (Participants) | 43 | 22
  C19D1 Score 3 | 0 | 0
  C19D1 Score 4: number analyzed (Participants) | 43 | 22
  C19D1 Score 4 | 0 | 0
  C19D1 Score 5: number analyzed (Participants) | 43 | 22
  C19D1 Score 5 | 0 | 0
  C20D1 Score 0: number analyzed (Participants) | 43 | 21
  C20D1 Score 0 | 24 | 15
  C20D1 Score 1: number analyzed (Participants) | 43 | 21
  C20D1 Score 1 | 19 | 6
  C20D1 Score 2: number analyzed (Participants) | 43 | 21
  C20D1 Score 2 | 0 | 0
  C20D1 Score 3: number analyzed (Participants) | 43 | 21
  C20D1 Score 3 | 0 | 0
  C20D1 Score 4: number analyzed (Participants) | 43 | 21
  C20D1 Score 4 | 0 | 0
  C20D1 Score 5: number analyzed (Participants) | 43 | 21
  C20D1 Score 5 | 0 | 0
  C21D1 Score 0: number analyzed (Participants) | 40 | 22
  C21D1 Score 0 | 23 | 15
  C21D1 Score 1: number analyzed (Participants) | 40 | 22
  C21D1 Score 1 | 17 | 7
  C21D1 Score 2: number analyzed (Participants) | 40 | 22
  C21D1 Score 2 | 0 | 0
  C21D1 Score 3: number analyzed (Participants) | 40 | 22
  C21D1 Score 3 | 0 | 0
  C21D1 Score 4: number analyzed (Participants) | 40 | 22
  C21D1 Score 4 | 0 | 0
  C21D1 Score 5: number analyzed (Participants) | 40 | 22
  C21D1 Score 5 | 0 | 0
  C22D1 Score 0: number analyzed (Participants) | 33 | 17
  C22D1 Score 0 | 17 | 12
  C22D1 Score 1: number analyzed (Participants) | 33 | 17
  C22D1 Score 1 | 15 | 5
  C22D1 Score 2: number analyzed (Participants) | 33 | 17
  C22D1 Score 2 | 1 | 0
  C22D1 Score 3: number analyzed (Participants) | 33 | 17
  C22D1 Score 3 | 0 | 0
  C22D1 Score 4: number analyzed (Participants) | 33 | 17
  C22D1 Score 4 | 0 | 0
  C22D1 Score 5: number analyzed (Participants) | 33 | 17
  C22D1 Score 5 | 0 | 0
  C23D1 Score 0: number analyzed (Participants) | 34 | 18
  C23D1 Score 0 | 20 | 14
  C23D1 Score 1: number analyzed (Participants) | 34 | 18
  C23D1 Score 1 | 14 | 4
  C23D1 Score 2: number analyzed (Participants) | 34 | 18
  C23D1 Score 2 | 0 | 0
  C23D1 Score 3: number analyzed (Participants) | 34 | 18
  C23D1 Score 3 | 0 | 0
  C23D1 Score 4: number analyzed (Participants) | 34 | 18
  C23D1 Score 4 | 0 | 0
  C23D1 Score 5: number analyzed (Participants) | 34 | 18
  C23D1 Score 5 | 0 | 0
  C24D1 Score 0: number analyzed (Participants) | 32 | 16
  C24D1 Score 0 | 19 | 11
  C24D1 Score 1: number analyzed (Participants) | 32 | 16
  C24D1 Score 1 | 13 | 5
  C24D1 Score 2: number analyzed (Participants) | 32 | 16
  C24D1 Score 2 | 0 | 0
  C24D1 Score 3: number analyzed (Participants) | 32 | 16
  C24D1 Score 3 | 0 | 0
  C24D1 Score 4: number analyzed (Participants) | 32 | 16
  C24D1 Score 4 | 0 | 0
  C24D1 Score 5: number analyzed (Participants) | 32 | 16
  C24D1 Score 5 | 0 | 0
  C25D1 Score 0: number analyzed (Participants) | 31 | 16
  C25D1 Score 0 | 17 | 11
  C25D1 Score 1: number analyzed (Participants) | 31 | 16
  C25D1 Score 1 | 14 | 5
  C25D1 Score 2: number analyzed (Participants) | 31 | 16
  C25D1 Score 2 | 0 | 0
  C25D1 Score 3: number analyzed (Participants) | 31 | 16
  C25D1 Score 3 | 0 | 0
  C25D1 Score 4: number analyzed (Participants) | 31 | 16
  C25D1 Score 4 | 0 | 0
  C25D1 Score 5: number analyzed (Participants) | 31 | 16
  C25D1 Score 5 | 0 | 0
  C26D1 Score 0: number analyzed (Participants) | 30 | 12
  C26D1 Score 0 | 19 | 8
  C26D1 Score 1: number analyzed (Participants) | 30 | 12
  C26D1 Score 1 | 11 | 4
  C26D1 Score 2: number analyzed (Participants) | 30 | 12
  C26D1 Score 2 | 0 | 0
  C26D1 Score 3: number analyzed (Participants) | 30 | 12
  C26D1 Score 3 | 0 | 0
  C26D1 Score 4: number analyzed (Participants) | 30 | 12
  C26D1 Score 4 | 0 | 0
  C26D1 Score 5: number analyzed (Participants) | 30 | 12
  C26D1 Score 5 | 0 | 0
  C27D1 Score 0: number analyzed (Participants) | 28 | 12
  C27D1 Score 0 | 17 | 8
  C27D1 Score 1: number analyzed (Participants) | 28 | 12
  C27D1 Score 1 | 11 | 4
  C27D1 Score 2: number analyzed (Participants) | 28 | 12
  C27D1 Score 2 | 0 | 0
  C27D1 Score 3: number analyzed (Participants) | 28 | 12
  C27D1 Score 3 | 0 | 0
  C27D1 Score 4: number analyzed (Participants) | 28 | 12
  C27D1 Score 4 | 0 | 0
  C27D1 Score 5: number analyzed (Participants) | 28 | 12
  C27D1 Score 5 | 0 | 0
  C28D1 Score 0: number analyzed (Participants) | 24 | 12
  C28D1 Score 0 | 17 | 8
  C28D1 Score 1: number analyzed (Participants) | 24 | 12
  C28D1 Score 1 | 7 | 4
  C28D1 Score 2: number analyzed (Participants) | 24 | 12
  C28D1 Score 2 | 0 | 0
  C28D1 Score 3: number analyzed (Participants) | 24 | 12
  C28D1 Score 3 | 0 | 0
  C28D1 Score 4: number analyzed (Participants) | 24 | 12
  C28D1 Score 4 | 0 | 0
  C28D1 Score 5: number analyzed (Participants) | 24 | 12
  C28D1 Score 5 | 0 | 0
  C29D1 Score 0: number analyzed (Participants) | 24 | 12
  C29D1 Score 0 | 17 | 8
  C29D1 Score 1: number analyzed (Participants) | 24 | 12
  C29D1 Score 1 | 7 | 4
  C29D1 Score 2: number analyzed (Participants) | 24 | 12
  C29D1 Score 2 | 0 | 0
  C29D1 Score 3: number analyzed (Participants) | 24 | 12
  C29D1 Score 3 | 0 | 0
  C29D1 Score 4: number analyzed (Participants) | 24 | 12
  C29D1 Score 4 | 0 | 0
  C29D1 Score 5: number analyzed (Participants) | 24 | 12
  C29D1 Score 5 | 0 | 0
  C30D1 Score 0: number analyzed (Participants) | 22 | 8
  C30D1 Score 0 | 15 | 4
  C30D1 Score 1: number analyzed (Participants) | 22 | 8
  C30D1 Score 1 | 7 | 4
  C30D1 Score 2: number analyzed (Participants) | 22 | 8
  C30D1 Score 2 | 0 | 0
  C30D1 Score 3: number analyzed (Participants) | 22 | 8
  C30D1 Score 3 | 0 | 0
  C30D1 Score 4: number analyzed (Participants) | 22 | 8
  C30D1 Score 4 | 0 | 0
  C30D1 Score 5: number analyzed (Participants) | 22 | 8
  C30D1 Score 5 | 0 | 0
  C31D1 Score 0: number analyzed (Participants) | 22 | 7
  C31D1 Score 0 | 15 | 3
  C31D1 Score 1: number analyzed (Participants) | 22 | 7
  C31D1 Score 1 | 7 | 4
  C31D1 Score 2: number analyzed (Participants) | 22 | 7
  C31D1 Score 2 | 0 | 0
  C31D1 Score 3: number analyzed (Participants) | 22 | 7
  C31D1 Score 3 | 0 | 0
  C31D1 Score 4: number analyzed (Participants) | 22 | 7
  C31D1 Score 4 | 0 | 0
  C31D1 Score 5: number analyzed (Participants) | 22 | 7
  C31D1 Score 5 | 0 | 0
  C32D1 Score 0: number analyzed (Participants) | 19 | 8
  C32D1 Score 0 | 13 | 4
  C32D1 Score 1: number analyzed (Participants) | 19 | 8
  C32D1 Score 1 | 6 | 4
  C32D1 Score 2: number analyzed (Participants) | 19 | 8
  C32D1 Score 2 | 0 | 0
  C32D1 Score 3: number analyzed (Participants) | 19 | 8
  C32D1 Score 3 | 0 | 0
  C32D1 Score 4: number analyzed (Participants) | 19 | 8
  C32D1 Score 4 | 0 | 0
  C32D1 Score 5: number analyzed (Participants) | 19 | 8
  C32D1 Score 5 | 0 | 0
  C33D1 Score 0: number analyzed (Participants) | 16 | 7
  C33D1 Score 0 | 11 | 4
  C33D1 Score 1: number analyzed (Participants) | 16 | 7
  C33D1 Score 1 | 5 | 3
  C33D1 Score 2: number analyzed (Participants) | 16 | 7
  C33D1 Score 2 | 0 | 0
  C33D1 Score 3: number analyzed (Participants) | 16 | 7
  C33D1 Score 3 | 0 | 0
  C33D1 Score 4: number analyzed (Participants) | 16 | 7
  C33D1 Score 4 | 0 | 0
  C33D1 Score 5: number analyzed (Participants) | 16 | 7
  C33D1 Score 5 | 0 | 0
  C34D1 Score 0: number analyzed (Participants) | 14 | 7
  C34D1 Score 0 | 11 | 4
  C34D1 Score 1: number analyzed (Participants) | 14 | 7
  C34D1 Score 1 | 3 | 3
  C34D1 Score 2: number analyzed (Participants) | 14 | 7
  C34D1 Score 2 | 0 | 0
  C34D1 Score 3: number analyzed (Participants) | 14 | 7
  C34D1 Score 3 | 0 | 0
  C34D1 Score 4: number analyzed (Participants) | 14 | 7
  C34D1 Score 4 | 0 | 0
  C34D1 Score 5: number analyzed (Participants) | 14 | 7
  C34D1 Score 5 | 0 | 0
  C35D1 Score 0: number analyzed (Participants) | 15 | 6
  C35D1 Score 0 | 10 | 3
  C35D1 Score 1: number analyzed (Participants) | 15 | 6
  C35D1 Score 1 | 5 | 3
  C35D1 Score 2: number analyzed (Participants) | 15 | 6
  C35D1 Score 2 | 0 | 0
  C35D1 Score 3: number analyzed (Participants) | 15 | 6
  C35D1 Score 3 | 0 | 0
  C35D1 Score 4: number analyzed (Participants) | 15 | 6
  C35D1 Score 4 | 0 | 0
  C35D1 Score 5: number analyzed (Participants) | 15 | 6
  C35D1 Score 5 | 0 | 0
  C36D1 Score 0: number analyzed (Participants) | 16 | 4
  C36D1 Score 0 | 10 | 1
  C36D1 Score 1: number analyzed (Participants) | 16 | 4
  C36D1 Score 1 | 6 | 3
  C36D1 Score 2: number analyzed (Participants) | 16 | 4
  C36D1 Score 2 | 0 | 0
  C36D1 Score 3: number analyzed (Participants) | 16 | 4
  C36D1 Score 3 | 0 | 0
  C36D1 Score 4: number analyzed (Participants) | 16 | 4
  C36D1 Score 4 | 0 | 0
  C36D1 Score 5: number analyzed (Participants) | 16 | 4
  C36D1 Score 5 | 0 | 0
  C37D1 Score 0: number analyzed (Participants) | 14 | 4
  C37D1 Score 0 | 9 | 3
  C37D1 Score 1: number analyzed (Participants) | 14 | 4
  C37D1 Score 1 | 5 | 1
  C37D1 Score 2: number analyzed (Participants) | 14 | 4
  C37D1 Score 2 | 0 | 0
  C37D1 Score 3: number analyzed (Participants) | 14 | 4
  C37D1 Score 3 | 0 | 0
  C37D1 Score 4: number analyzed (Participants) | 14 | 4
  C37D1 Score 4 | 0 | 0
  C37D1 Score 5: number analyzed (Participants) | 14 | 4
  C37D1 Score 5 | 0 | 0
  C38D1 Score 0: number analyzed (Participants) | 13 | 3
  C38D1 Score 0 | 8 | 2
  C38D1 Score 1: number analyzed (Participants) | 13 | 3
  C38D1 Score 1 | 5 | 1
  C38D1 Score 2: number analyzed (Participants) | 13 | 3
  C38D1 Score 2 | 0 | 0
  C38D1 Score 3: number analyzed (Participants) | 13 | 3
  C38D1 Score 3 | 0 | 0
  C38D1 Score 4: number analyzed (Participants) | 13 | 3
  C38D1 Score 4 | 0 | 0
  C38D1 Score 5: number analyzed (Participants) | 13 | 3
  C38D1 Score 5 | 0 | 0
  C39D1 Score 0: number analyzed (Participants) | 11 | 1
  C39D1 Score 0 | 8 | 1
  C39D1 Score 1: number analyzed (Participants) | 11 | 1
  C39D1 Score 1 | 3 | 0
  C39D1 Score 2: number analyzed (Participants) | 11 | 1
  C39D1 Score 2 | 0 | 0
  C39D1 Score 3: number analyzed (Participants) | 11 | 1
  C39D1 Score 3 | 0 | 0
  C39D1 Score 4: number analyzed (Participants) | 11 | 1
  C39D1 Score 4 | 0 | 0
  C39D1 Score 5: number analyzed (Participants) | 11 | 1
  C39D1 Score 5 | 0 | 0
  C40D1 Score 0: number analyzed (Participants) | 11 | 1
  C40D1 Score 0 | 8 | 1
  C40D1 Score 1: number analyzed (Participants) | 11 | 1
  C40D1 Score 1 | 3 | 0
  C40D1 Score 2: number analyzed (Participants) | 11 | 1
  C40D1 Score 2 | 0 | 0
  C40D1 Score 3: number analyzed (Participants) | 11 | 1
  C40D1 Score 3 | 0 | 0
  C40D1 Score 4: number analyzed (Participants) | 11 | 1
  C40D1 Score 4 | 0 | 0
  C40D1 Score 5: number analyzed (Participants) | 11 | 1
  C40D1 Score 5 | 0 | 0
  C41D1 Score 0: number analyzed (Participants) | 11 | 1
  C41D1 Score 0 | 8 | 1
  C41D1 Score 1: number analyzed (Participants) | 11 | 1
  C41D1 Score 1 | 3 | 0
  C41D1 Score 2: number analyzed (Participants) | 11 | 1
  C41D1 Score 2 | 0 | 0
  C41D1 Score 3: number analyzed (Participants) | 11 | 1
  C41D1 Score 3 | 0 | 0
  C41D1 Score 4: number analyzed (Participants) | 11 | 1
  C41D1 Score 4 | 0 | 0
  C41D1 Score 5: number analyzed (Participants) | 11 | 1
  C41D1 Score 5 | 0 | 0
  C42D1 Score 0: number analyzed (Participants) | 10 | 1
  C42D1 Score 0 | 7 | 1
  C42D1 Score 1: number analyzed (Participants) | 10 | 1
  C42D1 Score 1 | 3 | 0
  C42D1 Score 2: number analyzed (Participants) | 10 | 1
  C42D1 Score 2 | 0 | 0
  C42D1 Score 3: number analyzed (Participants) | 10 | 1
  C42D1 Score 3 | 0 | 0
  C42D1 Score 4: number analyzed (Participants) | 10 | 1
  C42D1 Score 4 | 0 | 0
  C42D1 Score 5: number analyzed (Participants) | 10 | 1
  C42D1 Score 5 | 0 | 0
  C43D1 Score 0: number analyzed (Participants) | 7 | 1
  C43D1 Score 0 | 5 | 1
  C43D1 Score 1: number analyzed (Participants) | 7 | 1
  C43D1 Score 1 | 2 | 0
  C43D1 Score 2: number analyzed (Participants) | 7 | 1
  C43D1 Score 2 | 0 | 0
  C43D1 Score 3: number analyzed (Participants) | 7 | 1
  C43D1 Score 3 | 0 | 0
  C43D1 Score 4: number analyzed (Participants) | 7 | 1
  C43D1 Score 4 | 0 | 0
  C43D1 Score 5: number analyzed (Participants) | 7 | 1
  C43D1 Score 5 | 0 | 0
  C44D1 Score 0: number analyzed (Participants) | 9 | 1
  C44D1 Score 0 | 7 | 1
  C44D1 Score 1: number analyzed (Participants) | 9 | 1
  C44D1 Score 1 | 2 | 0
  C44D1 Score 2: number analyzed (Participants) | 9 | 1
  C44D1 Score 2 | 0 | 0
  C44D1 Score 3: number analyzed (Participants) | 9 | 1
  C44D1 Score 3 | 0 | 0
  C44D1 Score 4: number analyzed (Participants) | 9 | 1
  C44D1 Score 4 | 0 | 0
  C44D1 Score 5: number analyzed (Participants) | 9 | 1
  C44D1 Score 5 | 0 | 0
  C45D1 Score 0: number analyzed (Participants) | 9 | 1
  C45D1 Score 0 | 7 | 1
  C45D1 Score 1: number analyzed (Participants) | 9 | 1
  C45D1 Score 1 | 2 | 0
  C45D1 Score 2: number analyzed (Participants) | 9 | 1
  C45D1 Score 2 | 0 | 0
  C45D1 Score 3: number analyzed (Participants) | 9 | 1
  C45D1 Score 3 | 0 | 0
  C45D1 Score 4: number analyzed (Participants) | 9 | 1
  C45D1 Score 4 | 0 | 0
  C45D1 Score 5: number analyzed (Participants) | 9 | 1
  C45D1 Score 5 | 0 | 0
  C46D1 Score 0: number analyzed (Participants) | 9 | 0
  C46D1 Score 0 | 7 |
  C46D1 Score 1: number analyzed (Participants) | 9 | 0
  C46D1 Score 1 | 2 |
  C46D1 Score 2: number analyzed (Participants) | 9 | 0
  C46D1 Score 2 | 0 |
  C46D1 Score 3: number analyzed (Participants) | 9 | 0
  C46D1 Score 3 | 0 |
  C46D1 Score 4: number analyzed (Participants) | 9 | 0
  C46D1 Score 4 | 0 |
  C46D1 Score 5: number analyzed (Participants) | 9 | 0
  C46D1 Score 5 | 0 |
  C47D1 Score 0: number analyzed (Participants) | 8 | 0
  C47D1 Score 0 | 6 |
  C47D1 Score 1: number analyzed (Participants) | 8 | 0
  C47D1 Score 1 | 2 |
  C47D1 Score 2: number analyzed (Participants) | 8 | 0
  C47D1 Score 2 | 0 |
  C47D1 Score 3: number analyzed (Participants) | 8 | 0
  C47D1 Score 3 | 0 |
  C47D1 Score 4: number analyzed (Participants) | 8 | 0
  C47D1 Score 4 | 0 |
  C47D1 Score 5: number analyzed (Participants) | 8 | 0
  C47D1 Score 5 | 0 |
  C48D1 Score 0: number analyzed (Participants) | 7 | 0
  C48D1 Score 0 | 5 |
  C48D1 Score 1: number analyzed (Participants) | 7 | 0
  C48D1 Score 1 | 2 |
  C48D1 Score 2: number analyzed (Participants) | 7 | 0
  C48D1 Score 2 | 0 |
  C48D1 Score 3: number analyzed (Participants) | 7 | 0
  C48D1 Score 3 | 0 |
  C48D1 Score 4: number analyzed (Participants) | 7 | 0
  C48D1 Score 4 | 0 |
  C48D1 Score 5: number analyzed (Participants) | 7 | 0
  C48D1 Score 5 | 0 |
  C49D1 Score 0: number analyzed (Participants) | 5 | 0
  C49D1 Score 0 | 3 |
  C49D1 Score 1: number analyzed (Participants) | 5 | 0
  C49D1 Score 1 | 2 |
  C49D1 Score 2: number analyzed (Participants) | 5 | 0
  C49D1 Score 2 | 0 |
  C49D1 Score 3: number analyzed (Participants) | 5 | 0
  C49D1 Score 3 | 0 |
  C49D1 Score 4: number analyzed (Participants) | 5 | 0
  C49D1 Score 4 | 0 |
  C49D1 Score 5: number analyzed (Participants) | 5 | 0
  C49D1 Score 5 | 0 |
  C50D1 Score 0: number analyzed (Participants) | 4 | 0
  C50D1 Score 0 | 2 |
  C50D1 Score 1: number analyzed (Participants) | 4 | 0
  C50D1 Score 1 | 2 |
  C50D1 Score 2: number analyzed (Participants) | 4 | 0
  C50D1 Score 2 | 0 |
  C50D1 Score 3: number analyzed (Participants) | 4 | 0
  C50D1 Score 3 | 0 |
  C50D1 Score 4: number analyzed (Participants) | 4 | 0
  C50D1 Score 4 | 0 |
  C50D1 Score 5: number analyzed (Participants) | 4 | 0
  C50D1 Score 5 | 0 |
  C51D1 Score 0: number analyzed (Participants) | 4 | 0
  C51D1 Score 0 | 2 |
  C51D1 Score 1: number analyzed (Participants) | 4 | 0
  C51D1 Score 1 | 2 |
  C51D1 Score 2: number analyzed (Participants) | 4 | 0
  C51D1 Score 2 | 0 |
  C51D1 Score 3: number analyzed (Participants) | 4 | 0
  C51D1 Score 3 | 0 |
  C51D1 Score 4: number analyzed (Participants) | 4 | 0
  C51D1 Score 4 | 0 |
  C51D1 Score 5: number analyzed (Participants) | 4 | 0
  C51D1 Score 5 | 0 |
  C52D1 Score 0: number analyzed (Participants) | 4 | 0
  C52D1 Score 0 | 2 |
  C52D1 Score 1: number analyzed (Participants) | 4 | 0
  C52D1 Score 1 | 2 |
  C52D1 Score 2: number analyzed (Participants) | 4 | 0
  C52D1 Score 2 | 0 |
  C52D1 Score 3: number analyzed (Participants) | 4 | 0
  C52D1 Score 3 | 0 |
  C52D1 Score 4: number analyzed (Participants) | 4 | 0
  C52D1 Score 4 | 0 |
  C52D1 Score 5: number analyzed (Participants) | 4 | 0
  C52D1 Score 5 | 0 |
  C53D1 Score 0: number analyzed (Participants) | 3 | 0
  C53D1 Score 0 | 2 |
  C53D1 Score 1: number analyzed (Participants) | 3 | 0
  C53D1 Score 1 | 1 |
  C53D1 Score 2: number analyzed (Participants) | 3 | 0
  C53D1 Score 2 | 0 |
  C53D1 Score 3: number analyzed (Participants) | 3 | 0
  C53D1 Score 3 | 0 |
  C53D1 Score 4: number analyzed (Participants) | 3 | 0
  C53D1 Score 4 | 0 |
  C53D1 Score 5: number analyzed (Participants) | 3 | 0
  C53D1 Score 5 | 0 |
  C54D1 Score 0: number analyzed (Participants) | 3 | 0
  C54D1 Score 0 | 2 |
  C54D1 Score 1: number analyzed (Participants) | 3 | 0
  C54D1 Score 1 | 1 |
  C54D1 Score 2: number analyzed (Participants) | 3 | 0
  C54D1 Score 2 | 0 |
  C54D1 Score 3: number analyzed (Participants) | 3 | 0
  C54D1 Score 3 | 0 |
  C54D1 Score 4: number analyzed (Participants) | 3 | 0
  C54D1 Score 4 | 0 |
  C54D1 Score 5: number analyzed (Participants) | 3 | 0
  C54D1 Score 5 | 0 |
  C55D1 Score 0: number analyzed (Participants) | 2 | 0
  C55D1 Score 0 | 1 |
  C55D1 Score 1: number analyzed (Participants) | 2 | 0
  C55D1 Score 1 | 1 |
  C55D1 Score 2: number analyzed (Participants) | 2 | 0
  C55D1 Score 2 | 0 |
  C55D1 Score 3: number analyzed (Participants) | 2 | 0
  C55D1 Score 3 | 0 |
  C55D1 Score 4: number analyzed (Participants) | 2 | 0
  C55D1 Score 4 | 0 |
  C55D1 Score 5: number analyzed (Participants) | 2 | 0
  C55D1 Score 5 | 0 |
  C56D1 Score 0: number analyzed (Participants) | 2 | 0
  C56D1 Score 0 | 1 |
  C56D1 Score 1: number analyzed (Participants) | 2 | 0
  C56D1 Score 1 | 1 |
  C56D1 Score 2: number analyzed (Participants) | 2 | 0
  C56D1 Score 2 | 0 |
  C56D1 Score 3: number analyzed (Participants) | 2 | 0
  C56D1 Score 3 | 0 |
  C56D1 Score 4: number analyzed (Participants) | 2 | 0
  C56D1 Score 4 | 0 |
  C56D1 Score 5: number analyzed (Participants) | 2 | 0
  C56D1 Score 5 | 0 |
  C57D1 Score 0: number analyzed (Participants) | 1 | 0
  C57D1 Score 0 | 1 |
  C57D1 Score 1: number analyzed (Participants) | 1 | 0
  C57D1 Score 1 | 0 |
  C57D1 Score 2: number analyzed (Participants) | 1 | 0
  C57D1 Score 2 | 0 |
  C57D1 Score 3: number analyzed (Participants) | 1 | 0
  C57D1 Score 3 | 0 |
  C57D1 Score 4: number analyzed (Participants) | 1 | 0
  C57D1 Score 4 | 0 |
  C57D1 Score 5: number analyzed (Participants) | 1 | 0
  C57D1 Score 5 | 0 |
  C58D1 Score 0: number analyzed (Participants) | 1 | 0
  C58D1 Score 0 | 1 |
  C58D1 Score 1: number analyzed (Participants) | 1 | 0
  C58D1 Score 1 | 0 |
  C58D1 Score 2: number analyzed (Participants) | 1 | 0
  C58D1 Score 2 | 0 |
  C58D1 Score 3: number analyzed (Participants) | 1 | 0
  C58D1 Score 3 | 0 |
  C58D1 Score 4: number analyzed (Participants) | 1 | 0
  C58D1 Score 4 | 0 |
  C58D1 Score 5: number analyzed (Participants) | 1 | 0
  C58D1 Score 5 | 0 |
  C59D1 Score 0: number analyzed (Participants) | 1 | 0
  C59D1 Score 0 | 1 |
  C59D1 Score 1: number analyzed (Participants) | 1 | 0
  C59D1 Score 1 | 0 |
  C59D1 Score 2: number analyzed (Participants) | 1 | 0
  C59D1 Score 2 | 0 |
  C59D1 Score 3: number analyzed (Participants) | 1 | 0
  C59D1 Score 3 | 0 |
  C59D1 Score 4: number analyzed (Participants) | 1 | 0
  C59D1 Score 4 | 0 |
  C59D1 Score 5: number analyzed (Participants) | 1 | 0
  C59D1 Score 5 | 0 |
  C60D1 Score 0: number analyzed (Participants) | 1 | 0
  C60D1 Score 0 | 1 |
  C60D1 Score 1: number analyzed (Participants) | 1 | 0
  C60D1 Score 1 | 0 |
  C60D1 Score 2: number analyzed (Participants) | 1 | 0
  C60D1 Score 2 | 0 |
  C60D1 Score 3: number analyzed (Participants) | 1 | 0
  C60D1 Score 3 | 0 |
  C60D1 Score 4: number analyzed (Participants) | 1 | 0
  C60D1 Score 4 | 0 |
  C60D1 Score 5: number analyzed (Participants) | 1 | 0
  C60D1 Score 5 | 0 |

10. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) Measured by the EORTC-QLQ-C30 Questionnaire
Description: The EORTC-QLQ-C30 is a cancer-specific instrument consisting of 5 functional domain scales: physical, role, emotional, social and cognitive.It is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Most items are scored 1 ('not at all') to 4 ('very much') except for the items contributing to the global health status/QoL, which are scored 1 ('very poor') to 7 ('excellent'). All raw domain scores are linearly transformed to a 0-100 scale with higher scores on symptoms indicate a worse health state.
Time Frame: Baseline, on D1 from C2 through C39, 30-day follow up, 90-day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 243 | 242
Unit on a scale
  Global Health Status Baseline | 68.83 (18.94) | 66.15 (19.40)
  Global Health Status C2D1: number analyzed (Participants) | 208 | 217
  Global Health Status C2D1 | 0.04 (17.35) | 2.96 (18.89)
  Global Health Status C3D1: number analyzed (Participants) | 182 | 197
  Global Health Status C3D1 | 1.47 (17.15) | 3.68 (20.69)
  Global Health Status C4D1: number analyzed (Participants) | 169 | 169
  Global Health Status C4D1 | 2.61 (18.79) | 4.54 (20.59)
  Global Health Status C5D1: number analyzed (Participants) | 159 | 165
  Global Health Status C5D1 | 0.89 (20.96) | 3.48 (19.57)
  Global Health Status C6D1: number analyzed (Participants) | 149 | 146
  Global Health Status C6D1 | 0.84 (19.32) | 3.94 (20.51)
  Global Health Status C7D1: number analyzed (Participants) | 120 | 126
  Global Health Status C7D1 | 1.94 (18.29) | 2.12 (19.69)
  Global Health Status C8D1: number analyzed (Participants) | 108 | 110
  Global Health Status C8D1 | 0.77 (16.96) | 4.32 (20.31)
  Global Health Status C9D1: number analyzed (Participants) | 102 | 103
  Global Health Status C9D1 | 1.88 (20.91) | 3.32 (20.89)
  Global Health Status C10D1: number analyzed (Participants) | 85 | 79
  Global Health Status C10D1 | 2.65 (20.38) | 3.48 (22.23)
  Global Health Status C11D1: number analyzed (Participants) | 81 | 71
  Global Health Status C11D1 | 1.23 (21.89) | 3.99 (23.18)
  Global Health Status C12D1: number analyzed (Participants) | 75 | 57
  Global Health Status C12D1 | 2.44 (23.44) | 2.63 (22.06)
  Global Health Status C13D1: number analyzed (Participants) | 60 | 48
  Global Health Status C13D1 | 3.47 (24.22) | 3.30 (20.82)
  Global Health Status C14D1: number analyzed (Participants) | 55 | 44
  Global Health Status C14D1 | 1.52 (18.08) | 3.79 (21.15)
  Global Health Status C15D1: number analyzed (Participants) | 51 | 36
  Global Health Status C15D1 | 2.94 (22.78) | 2.08 (21.02)
  Global Health Status C16D1: number analyzed (Participants) | 48 | 31
  Global Health Status C16D1 | 3.65 (22.67) | 5.65 (17.40)
  Global Health Status C17D1: number analyzed (Participants) | 43 | 25
  Global Health Status C17D1 | 6.01 (19.36) | 3.33 (20.41)
  Global Health Status C18D1: number analyzed (Participants) | 41 | 21
  Global Health Status C18D1 | 3.66 (21.33) | 3.97 (31.36)
  Global Health Status C19D1: number analyzed (Participants) | 40 | 20
  Global Health Status C19D1 | 4.17 (17.50) | 10.42 (15.97)
  Global Health Status C20D1: number analyzed (Participants) | 39 | 19
  Global Health Status C20D1 | 1.50 (17.72) | 3.95 (19.71)
  Global Health Status C21D1: number analyzed (Participants) | 36 | 20
  Global Health Status C21D1 | 4.17 (18.53) | 2.92 (18.98)
  Global Health Status C22D1: number analyzed (Participants) | 31 | 17
  Global Health Status C22D1 | 4.03 (19.71) | 9.31 (22.99)
  Global Health Status C23D1: number analyzed (Participants) | 31 | 16
  Global Health Status C23D1 | 4.03 (16.92) | 9.38 (19.69)
  Global Health Status C24D1: number analyzed (Participants) | 29 | 12
  Global Health Status C24D1 | 2.87 (19.32) | 9.72 (21.86)
  Global Health Status C25D1: number analyzed (Participants) | 28 | 12
  Global Health Status C25D1 | 1.79 (18.75) | 10.42 (24.39)
  Global Health Status C26D1: number analyzed (Participants) | 26 | 9
  Global Health Status C26D1 | 4.81 (16.36) | 3.70 (19.59)
  Global Health Status C27D1: number analyzed (Participants) | 25 | 10
  Global Health Status C27D1 | 4.00 (18.18) | 6.67 (11.65)
  Global Health Status C28D1: number analyzed (Participants) | 21 | 11
  Global Health Status C28D1 | 1.98 (18.62) | 5.30 (14.08)
  Global Health Status C29D1: number analyzed (Participants) | 22 | 12
  Global Health Status C29D1 | 3.03 (14.21) | 4.86 (14.42)
  Global Health Status C30D1: number analyzed (Participants) | 20 | 0
  Global Health Status C30D1 | 2.92 (14.12) |
  Global Health Status C31D1: number analyzed (Participants) | 20 | 0
  Global Health Status C31D1 | 2.08 (19.28) |
  Global Health Status C32D1: number analyzed (Participants) | 18 | 0
  Global Health Status C32D1 | 2.78 (16.17) |
  Global Health Status C33D1: number analyzed (Participants) | 15 | 0
  Global Health Status C33D1 | 5.56 (17.72) |
  Global Health Status C34D1: number analyzed (Participants) | 12 | 0
  Global Health Status C34D1 | 8.33 (20.72) |
  Global Health Status C35D1: number analyzed (Participants) | 13 | 0
  Global Health Status C35D1 | 4.49 (17.88) |
  Global Health Status C36D1: number analyzed (Participants) | 12 | 0
  Global Health Status C36D1 | 2.78 (17.16) |
  Global Health Status C37D1: number analyzed (Participants) | 11 | 0
  Global Health Status C37D1 | 10.61 (15.85) |
  Global Health Status C38D1: number analyzed (Participants) | 10 | 0
  Global Health Status C38D1 | 8.33 (21.15) |
  Global Health Status C39D1: number analyzed (Participants) | 9 | 0
  Global Health Status C39D1 | 3.70 (13.89) |
  Global Health Status 30 day follow up: number analyzed (Participants) | 57 | 78
  Global Health Status 30 day follow up | -8.63 (25.10) | -10.68 (24.65)
  Global Health Status 90 day follow up: number analyzed (Participants) | 61 | 79
  Global Health Status 90 day follow up | -5.46 (21.19) | -4.96 (22.86)
  Physical Functioning Baseline | 83.79 (16.85) | 83.55 (17.22)
  Physical Functioning C2D1: number analyzed (Participants) | 208 | 217
  Physical Functioning C2D1 | -0.93 (14.62) | -0.77 (13.70)
  Physical Functioning C3D1: number analyzed (Participants) | 182 | 197
  Physical Functioning C3D1 | -1.76 (14.13) | -0.07 (14.94)
  Physical Functioning C4D1: number analyzed (Participants) | 169 | 169
  Physical Functioning C4D1 | -0.16 (14.25) | 1.07 (15.38)
  Physical Functioning C5D1: number analyzed (Participants) | 159 | 165
  Physical Functioning C5D1 | -0.67 (15.32) | 0.24 (16.29)
  Physical Functioning C6D1: number analyzed (Participants) | 149 | 146
  Physical Functioning C6D1 | -0.89 (15.47) | -0.96 (17.94)
  Physical Functioning C7D1: number analyzed (Participants) | 120 | 126
  Physical Functioning C7D1 | -1.78 (16.05) | 0.21 (17.69)
  Physical Functioning C8D1: number analyzed (Participants) | 108 | 110
  Physical Functioning C8D1 | -3.27 (15.51) | -1.33 (17.08)
  Physical Functioning C9D1: number analyzed (Participants) | 102 | 103
  Physical Functioning C9D1 | -3.20 (17.84) | -0.84 (18.26)
  Physical Functioning C10D1: number analyzed (Participants) | 85 | 79
  Physical Functioning C10D1 | -2.75 (17.13) | -2.28 (18.76)
  Physical Functioning C11D1: number analyzed (Participants) | 81 | 71
  Physical Functioning C11D1 | -0.82 (15.00) | -0.09 (17.11)
  Physical Functioning C12D1: number analyzed (Participants) | 75 | 57
  Physical Functioning C12D1 | -0.89 (17.31) | -0.70 (19.18)
  Physical Functioning C13D1: number analyzed (Participants) | 60 | 48
  Physical Functioning C13D1 | -0.56 (18.59) | 0.97 (13.89)
  Physical Functioning C14D1: number analyzed (Participants) | 55 | 44
  Physical Functioning C14D1 | 0.12 (15.95) | 1.21 (13.04)
  Physical Functioning C15D1: number analyzed (Participants) | 51 | 36
  Physical Functioning C15D1 | 0.39 (14.20) | 0.00 (13.62)
  Physical Functioning C16D1: number analyzed (Participants) | 48 | 31
  Physical Functioning C16D1 | -0.42 (14.77) | 0.86 (12.14)
  Physical Functioning C17D1: number analyzed (Participants) | 43 | 25
  Physical Functioning C17D1 | 2.33 (14.61) | 2.13 (16.75)
  Physical Functioning C18D1: number analyzed (Participants) | 41 | 21
  Physical Functioning C18D1 | -2.93 (17.32) | 3.49 (15.44)
  Physical Functioning C19D1: number analyzed (Participants) | 40 | 20
  Physical Functioning C19D1 | 1.33 (10.48) | 4.00 (13.40)
  Physical Functioning C20D1: number analyzed (Participants) | 39 | 19
  Physical Functioning C20D1 | -0.85 (11.96) | 2.81 (16.68)
  Physical Functioning C21D1: number analyzed (Participants) | 36 | 20
  Physical Functioning C21D1 | -0.74 (13.31) | 3.33 (12.89)
  Physical Functioning C22D1: number analyzed (Participants) | 31 | 17
  Physical Functioning C22D1 | -0.22 (12.11) | 5.49 (17.52)
  Physical Functioning C23D1: number analyzed (Participants) | 31 | 16
  Physical Functioning C23D1 | -0.22 (14.35) | 5.83 (19.30)
  Physical Functioning C24D1: number analyzed (Participants) | 29 | 12
  Physical Functioning C24D1 | 2.30 (14.61) | 5.56 (17.71)
  Physical Functioning C25D1: number analyzed (Participants) | 28 | 12
  Physical Functioning C25D1 | 0.48 (17.40) | 3.89 (23.35)
  Physical Functioning C26D1: number analyzed (Participants) | 26 | 9
  Physical Functioning C26D1 | 1.28 (17.28) | 2.96 (17.36)
  Physical Functioning C27D1: number analyzed (Participants) | 25 | 10
  Physical Functioning C27D1 | 1.07 (16.52) | 2.00 (13.72)
  Physical Functioning C28D1: number analyzed (Participants) | 21 | 11
  Physical Functioning C28D1 | -1.27 (16.55) | -1.82 (19.80)
  Physical Functioning C29D1: number analyzed (Participants) | 22 | 12
  Physical Functioning C29D1 | -3.33 (23.25) | 1.11 (18.16)
  Physical Functioning C30D1: number analyzed (Participants) | 20 | 0
  Physical Functioning C30D1 | 1.67 (16.17) |
  Physical Functioning C31D1: number analyzed (Participants) | 20 | 0
  Physical Functioning C31D1 | 2.00 (16.91) |
  Physical Functioning C32D1: number analyzed (Participants) | 18 | 0
  Physical Functioning C32D1 | -1.11 (19.97) |
  Physical Functioning C33D1: number analyzed (Participants) | 15 | 0
  Physical Functioning C33D1 | 2.22 (18.11) |
  Physical Functioning C34D1: number analyzed (Participants) | 12 | 0
  Physical Functioning C34D1 | 6.67 (17.98) |
  Physical Functioning C35D1: number analyzed (Participants) | 13 | 0
  Physical Functioning C35D1 | 7.18 (18.55) |
  Physical Functioning C36D1: number analyzed (Participants) | 12 | 0
  Physical Functioning C36D1 | 6.67 (17.98) |
  Physical Functioning C37D1: number analyzed (Participants) | 11 | 0
  Physical Functioning C37D1 | 7.27 (17.24) |
  Physical Functioning C38D1: number analyzed (Participants) | 10 | 0
  Physical Functioning C38D1 | 6.67 (21.55) |
  Physical Functioning C39D1: number analyzed (Participants) | 9 | 0
  Physical Functioning C39D1 | 2.96 (10.06) |
  Physical Functioning 30 day follow up: number analyzed (Participants) | 57 | 78
  Physical Functioning 30 day follow up | -8.65 (22.36) | -9.91 (20.29)
  Physical Functioning 90 day follow up: number analyzed (Participants) | 61 | 79
  Physical Functioning 90 day follow up | -10.16 (20.28) | -10.63 (22.28)
  Role Functioning Baseline | 83.20 (22.52) | 82.23 (23.59)
  Role Functioning C2D1: number analyzed (Participants) | 208 | 217
  Role Functioning C2D1 | -2.64 (20.52) | -1.92 (19.97)
  Role Functioning C3D1: number analyzed (Participants) | 182 | 197
  Role Functioning C3D1 | -2.38 (21.82) | -2.28 (24.38)
  Role Functioning C4D1: number analyzed (Participants) | 169 | 169
  Role Functioning C4D1 | -2.37 (20.36) | -0.79 (24.65)
  Role Functioning C5D1: number analyzed (Participants) | 159 | 165
  Role Functioning C5D1 | -0.94 (20.73) | -0.40 (25.03)
  Role Functioning C6D1: number analyzed (Participants) | 149 | 146
  Role Functioning C6D1 | -3.69 (22.91) | -3.08 (24.68)
  Role Functioning C7D1: number analyzed (Participants) | 120 | 126
  Role Functioning C7D1 | -2.08 (20.68) | -0.79 (23.74)
  Role Functioning C8D1: number analyzed (Participants) | 108 | 110
  Role Functioning C8D1 | -5.25 (21.57) | -5.61 (26.16)
  Role Functioning C9D1: number analyzed (Participants) | 102 | 103
  Role Functioning C9D1 | -5.39 (23.71) | -2.59 (23.89)
  Role Functioning C10D1: number analyzed (Participants) | 85 | 79
  Role Functioning C10D1 | -3.92 (24.89) | -3.59 (26.91)
  Role Functioning C11D1: number analyzed (Participants) | 81 | 71
  Role Functioning C11D1 | -3.50 (19.31) | -3.29 (28.40)
  Role Functioning C12D1: number analyzed (Participants) | 75 | 57
  Role Functioning C12D1 | -3.33 (23.89) | -2.63 (26.69)
  Role Functioning C13D1: number analyzed (Participants) | 60 | 48
  Role Functioning C13D1 | -0.83 (24.44) | -0.35 (27.39)
  Role Functioning C14D1: number analyzed (Participants) | 55 | 44
  Role Functioning C14D1 | -1.21 (21.48) | 0.76 (21.25)
  Role Functioning C15D1: number analyzed (Participants) | 51 | 36
  Role Functioning C15D1 | -0.65 (21.07) | -0.46 (24.72)
  Role Functioning C16D1: number analyzed (Participants) | 48 | 31
  Role Functioning C16D1 | 1.74 (23.12) | 0.00 (21.08)
  Role Functioning C17D1: number analyzed (Participants) | 43 | 25
  Role Functioning C17D1 | 3.10 (22.50) | 2.67 (28.74)
  Role Functioning C18D1: number analyzed (Participants) | 41 | 21
  Role Functioning C18D1 | -3.25 (20.49) | 6.35 (21.39)
  Role Functioning C19D1: number analyzed (Participants) | 40 | 20
  Role Functioning C19D1 | -0.42 (20.50) | 6.67 (17.44)
  Role Functioning C20D1: number analyzed (Participants) | 39 | 19
  Role Functioning C20D1 | 1.28 (20.37) | 10.53 (22.37)
  Role Functioning C21D1: number analyzed (Participants) | 36 | 20
  Role Functioning C21D1 | -0.93 (20.29) | 6.67 (23.82)
  Role Functioning C22D1: number analyzed (Participants) | 31 | 17
  Role Functioning C22D1 | 0.54 (19.48) | 8.82 (24.38)
  Role Functioning C23D1: number analyzed (Participants) | 31 | 16
  Role Functioning C23D1 | 0.00 (18.76) | 9.37 (30.41)
  Role Functioning C24D1: number analyzed (Participants) | 29 | 12
  Role Functioning C24D1 | 0.00 (18.37) | 6.94 (27.02)
  Role Functioning C25D1: number analyzed (Participants) | 28 | 12
  Role Functioning C25D1 | 1.79 (20.95) | 8.33 (28.87)
  Role Functioning C26D1: number analyzed (Participants) | 26 | 9
  Role Functioning C26D1 | -0.64 (20.81) | -3.70 (27.36)
  Role Functioning C27D1: number analyzed (Participants) | 25 | 10
  Role Functioning C27D1 | 0.00 (17.35) | -3.33 (23.31)
  Role Functioning C28D1: number analyzed (Participants) | 21 | 11
  Role Functioning C28D1 | 1.59 (18.18) | -4.55 (21.20)
  Role Functioning C29D1: number analyzed (Participants) | 22 | 12
  Role Functioning C29D1 | -1.52 (24.62) | 2.78 (19.89)
  Role Functioning C30D1: number analyzed (Participants) | 20 | 0
  Role Functioning C30D1 | 3.33 (19.19) |
  Role Functioning C31D1: number analyzed (Participants) | 20 | 0
  Role Functioning C31D1 | 7.50 (21.27) |
  Role Functioning C32D1: number analyzed (Participants) | 18 | 0
  Role Functioning C32D1 | 5.56 (23.57) |
  Role Functioning C33D1: number analyzed (Participants) | 15 | 0
  Role Functioning C33D1 | 6.67 (20.70) |
  Role Functioning C34D1: number analyzed (Participants) | 12 | 0
  Role Functioning C34D1 | 9.72 (24.06) |
  Role Functioning C35D1: number analyzed (Participants) | 13 | 0
  Role Functioning C35D1 | 7.69 (21.10) |
  Role Functioning C36D1: number analyzed (Participants) | 12 | 0
  Role Functioning C36D1 | 9.72 (21.86) |
  Role Functioning C37D1: number analyzed (Participants) | 11 | 0
  Role Functioning C37D1 | 12.12 (23.68) |
  Role Functioning C38D1: number analyzed (Participants) | 10 | 0
  Role Functioning C38D1 | 13.33 (21.94) |
  Role Functioning C39D1: number analyzed (Participants) | 9 | 0
  Role Functioning C39D1 | 7.41 (22.22) |
  Role Functioning 30 day follow up: number analyzed (Participants) | 57 | 78
  Role Functioning 30 day follow up | -13.16 (27.95) | -16.88 (31.38)
  Role Functioning 90 day follow up: number analyzed (Participants) | 61 | 79
  Role Functioning 90 day follow up | -10.93 (27.03) | -9.49 (30.39)
  Emotional Functioning Baseline | 80.42 (19.13) | 78.79 (19.41)
  Emotional Functioning C2D1: number analyzed (Participants) | 208 | 217
  Emotional Functioning C2D1 | 1.32 (15.92) | 4.42 (16.49)
  Emotional Functioning C3D1: number analyzed (Participants) | 182 | 197
  Emotional Functioning C3D1 | 0.05 (16.21) | 3.00 (18.84)
  Emotional Functioning C4D1: number analyzed (Participants) | 169 | 169
  Emotional Functioning C4D1 | 2.42 (15.52) | 2.51 (19.52)
  Emotional Functioning C5D1: number analyzed (Participants) | 159 | 165
  Emotional Functioning C5D1 | 2.46 (17.35) | 3.69 (17.81)
  Emotional Functioning C6D1: number analyzed (Participants) | 149 | 146
  Emotional Functioning C6D1 | 1.79 (15.96) | 3.77 (19.18)
  Emotional Functioning C7D1: number analyzed (Participants) | 120 | 126
  Emotional Functioning C7D1 | 3.54 (17.90) | 2.12 (21.24)
  Emotional Functioning C8D1: number analyzed (Participants) | 108 | 110
  Emotional Functioning C8D1 | 0.77 (19.15) | 2.20 (18.08)
  Emotional Functioning C9D1: number analyzed (Participants) | 102 | 103
  Emotional Functioning C9D1 | 2.53 (19.19) | 2.59 (19.07)
  Emotional Functioning C10D1: number analyzed (Participants) | 85 | 79
  Emotional Functioning C10D1 | 5.20 (21.13) | 1.79 (20.62)
  Emotional Functioning C11D1: number analyzed (Participants) | 81 | 71
  Emotional Functioning C11D1 | 5.35 (20.47) | 2.58 (20.97)
  Emotional Functioning C12D1: number analyzed (Participants) | 75 | 57
  Emotional Functioning C12D1 | 6.44 (19.93) | 2.05 (21.49)
  Emotional Functioning C13D1: number analyzed (Participants) | 60 | 48
  Emotional Functioning C13D1 | 6.11 (20.40) | 1.91 (21.42)
  Emotional Functioning C14D1: number analyzed (Participants) | 55 | 44
  Emotional Functioning C14D1 | 3.94 (19.96) | -1.33 (18.76)
  Emotional Functioning C15D1: number analyzed (Participants) | 51 | 36
  Emotional Functioning C15D1 | 4.25 (16.61) | -1.85 (21.19)
  Emotional Functioning C16D1: number analyzed (Participants) | 48 | 31
  Emotional Functioning C16D1 | 3.99 (15.75) | -0.27 (23.22)
  Emotional Functioning C17D1: number analyzed (Participants) | 43 | 25
  Emotional Functioning C17D1 | 5.81 (15.16) | 5.33 (16.12)
  Emotional Functioning C18D1: number analyzed (Participants) | 41 | 21
  Emotional Functioning C18D1 | 2.24 (15.59) | 3.97 (19.65)
  Emotional Functioning C19D1: number analyzed (Participants) | 40 | 20
  Emotional Functioning C19D1 | 5.00 (15.07) | 4.58 (13.10)
  Emotional Functioning C20D1: number analyzed (Participants) | 39 | 19
  Emotional Functioning C20D1 | 3.85 (15.40) | 1.75 (19.95)
  Emotional Functioning C21D1: number analyzed (Participants) | 36 | 20
  Emotional Functioning C21D1 | 3.94 (18.31) | 5.00 (18.22)
  Emotional Functioning C22D1: number analyzed (Participants) | 31 | 17
  Emotional Functioning C22D1 | 4.30 (14.25) | 2.45 (18.58)
  Emotional Functioning C23D1: number analyzed (Participants) | 31 | 16
  Emotional Functioning C23D1 | 2.42 (11.42) | 3.65 (23.56)
  Emotional Functioning C24D1: number analyzed (Participants) | 29 | 12
  Emotional Functioning C24D1 | 2.59 (14.79) | -0.69 (23.96)
  Emotional Functioning C25D1: number analyzed (Participants) | 28 | 12
  Emotional Functioning C25D1 | 2.68 (16.36) | -0.69 (20.24)
  Emotional Functioning C26D1: number analyzed (Participants) | 26 | 9
  Emotional Functioning C26D1 | 4.17 (16.37) | -3.70 (18.69)
  Emotional Functioning C27D1: number analyzed (Participants) | 25 | 10
  Emotional Functioning C27D1 | 3.00 (18.30) | -5.83 (19.66)
  Emotional Functioning C28D1: number analyzed (Participants) | 21 | 11
  Emotional Functioning C28D1 | 0.79 (19.53) | -3.79 (19.85)
  Emotional Functioning C29D1: number analyzed (Participants) | 22 | 12
  Emotional Functioning C29D1 | 2.65 (17.33) | -3.47 (27.17)
  Emotional Functioning C30D1: number analyzed (Participants) | 20 | 0
  Emotional Functioning C30D1 | -0.42 (17.41) |
  Emotional Functioning C31D1: number analyzed (Participants) | 20 | 0
  Emotional Functioning C31D1 | 1.25 (17.16) |
  Emotional Functioning C32D1: number analyzed (Participants) | 18 | 0
  Emotional Functioning C32D1 | 3.70 (16.96) |
  Emotional Functioning C33D1: number analyzed (Participants) | 15 | 0
  Emotional Functioning C33D1 | 5.56 (18.81) |
  Emotional Functioning C34D1: number analyzed (Participants) | 12 | 0
  Emotional Functioning C34D1 | 11.81 (12.03) |
  Emotional Functioning C35D1: number analyzed (Participants) | 13 | 0
  Emotional Functioning C35D1 | 5.13 (15.79) |
  Emotional Functioning C36D1: number analyzed (Participants) | 12 | 0
  Emotional Functioning C36D1 | 9.03 (15.27) |
  Emotional Functioning C37D1: number analyzed (Participants) | 11 | 0
  Emotional Functioning C37D1 | 11.36 (15.93) |
  Emotional Functioning C38D1: number analyzed (Participants) | 10 | 0
  Emotional Functioning C38D1 | 10.83 (14.72) |
  Emotional Functioning C39D1: number analyzed (Participants) | 9 | 0
  Emotional Functioning C39D1 | -1.85 (21.15) |
  Emotional Functioning 30 day follow up: number analyzed (Participants) | 57 | 78
  Emotional Functioning 30 day follow up | -5.99 (26.01) | -5.02 (24.15)
  Emotional Functioning 90 day follow up: number analyzed (Participants) | 61 | 79
  Emotional Functioning 90 day follow up | -4.37 (15.34) | 0.21 (21.88)
  Cognitive Functioning Baseline | 90.95 (14.86) | 87.81 (18.01)
  Cognitive Functioning C2D1: number analyzed (Participants) | 208 | 217
  Cognitive Functioning C2D1 | -0.24 (13.36) | 0.54 (15.50)
  Cognitive Functioning C3D1: number analyzed (Participants) | 182 | 197
  Cognitive Functioning C3D1 | -1.47 (14.90) | 0.51 (15.51)
  Cognitive Functioning C4D1: number analyzed (Participants) | 169 | 169
  Cognitive Functioning C4D1 | -0.59 (13.47) | 1.87 (15.58)
  Cognitive Functioning C5D1: number analyzed (Participants) | 159 | 165
  Cognitive Functioning C5D1 | -1.89 (15.80) | 2.22 (15.13)
  Cognitive Functioning C6D1: number analyzed (Participants) | 149 | 146
  Cognitive Functioning C6D1 | -1.45 (14.87) | 0.91 (16.81)
  Cognitive Functioning C7D1: number analyzed (Participants) | 120 | 126
  Cognitive Functioning C7D1 | 0.00 (16.31) | -1.19 (17.02)
  Cognitive Functioning C8D1: number analyzed (Participants) | 108 | 110
  Cognitive Functioning C8D1 | -2.16 (15.13) | 0.15 (18.27)
  Cognitive Functioning C9D1: number analyzed (Participants) | 102 | 103
  Cognitive Functioning C9D1 | -1.96 (14.70) | 0.97 (18.05)
  Cognitive Functioning C10D1: number analyzed (Participants) | 85 | 79
  Cognitive Functioning C10D1 | -0.59 (17.15) | -0.42 (19.61)
  Cognitive Functioning C11D1: number analyzed (Participants) | 81 | 71
  Cognitive Functioning C11D1 | -1.23 (14.86) | -1.41 (18.42)
  Cognitive Functioning C12D1: number analyzed (Participants) | 75 | 57
  Cognitive Functioning C12D1 | -0.22 (13.83) | 1.17 (16.62)
  Cognitive Functioning C13D1: number analyzed (Participants) | 60 | 48
  Cognitive Functioning C13D1 | -0.28 (15.19) | 0.69 (22.00)
  Cognitive Functioning C14D1: number analyzed (Participants) | 55 | 44
  Cognitive Functioning C14D1 | 0.61 (15.70) | 0.00 (19.02)
  Cognitive Functioning C15D1: number analyzed (Participants) | 51 | 36
  Cognitive Functioning C15D1 | -0.98 (15.06) | -1.39 (19.67)
  Cognitive Functioning C16D1: number analyzed (Participants) | 48 | 31
  Cognitive Functioning C16D1 | 1.39 (16.43) | -2.69 (20.68)
  Cognitive Functioning C17D1: number analyzed (Participants) | 43 | 25
  Cognitive Functioning C17D1 | 0.78 (12.57) | 2.67 (14.97)
  Cognitive Functioning C18D1: number analyzed (Participants) | 41 | 21
  Cognitive Functioning C18D1 | 1.63 (13.85) | 2.38 (16.06)
  Cognitive Functioning C19D1: number analyzed (Participants) | 40 | 20
  Cognitive Functioning C19D1 | 0.42 (16.66) | 3.33 (11.60)
  Cognitive Functioning C20D1: number analyzed (Participants) | 39 | 19
  Cognitive Functioning C20D1 | 0.85 (17.91) | 1.75 (21.44)
  Cognitive Functioning C21D1: number analyzed (Participants) | 36 | 20
  Cognitive Functioning C21D1 | 0.93 (19.08) | 6.67 (18.26)
  Cognitive Functioning C22D1: number analyzed (Participants) | 31 | 17
  Cognitive Functioning C22D1 | 2.69 (18.31) | 4.90 (20.21)
  Cognitive Functioning C23D1: number analyzed (Participants) | 31 | 16
  Cognitive Functioning C23D1 | 1.61 (17.93) | 6.25 (17.08)
  Cognitive Functioning C24D1: number analyzed (Participants) | 29 | 12
  Cognitive Functioning C24D1 | 2.30 (18.75) | 0.00 (15.89)
  Cognitive Functioning C25D1: number analyzed (Participants) | 28 | 12
  Cognitive Functioning C25D1 | 1.79 (18.89) | 1.39 (19.41)
  Cognitive Functioning C26D1: number analyzed (Participants) | 26 | 9
  Cognitive Functioning C26D1 | 1.92 (19.05) | 0.00 (16.67)
  Cognitive Functioning C27D1: number analyzed (Participants) | 25 | 10
  Cognitive Functioning C27D1 | 2.67 (17.13) | -1.67 (14.59)
  Cognitive Functioning C28D1: number analyzed (Participants) | 21 | 11
  Cognitive Functioning C28D1 | 3.17 (18.72) | -3.03 (14.56)
  Cognitive Functioning C29D1: number analyzed (Participants) | 22 | 12
  Cognitive Functioning C29D1 | 0.76 (21.50) | 0.00 (14.21)
  Cognitive Functioning C30D1: number analyzed (Participants) | 20 | 0
  Cognitive Functioning C30D1 | 0.00 (18.73) |
  Cognitive Functioning C31D1: number analyzed (Participants) | 20 | 0
  Cognitive Functioning C31D1 | 0.00 (18.73) |
  Cognitive Functioning C32D1: number analyzed (Participants) | 18 | 0
  Cognitive Functioning C32D1 | 2.78 (21.58) |
  Cognitive Functioning C33D1: number analyzed (Participants) | 15 | 0
  Cognitive Functioning C33D1 | 5.56 (20.57) |
  Cognitive Functioning C34D1: number analyzed (Participants) | 12 | 0
  Cognitive Functioning C34D1 | 6.94 (21.86) |
  Cognitive Functioning C35D1: number analyzed (Participants) | 13 | 0
  Cognitive Functioning C35D1 | 6.41 (24.09) |
  Cognitive Functioning C36D1: number analyzed (Participants) | 12 | 0
  Cognitive Functioning C36D1 | 8.33 (19.46) |
  Cognitive Functioning C37D1: number analyzed (Participants) | 11 | 0
  Cognitive Functioning C37D1 | 9.09 (21.56) |
  Cognitive Functioning C38D1: number analyzed (Participants) | 10 | 0
  Cognitive Functioning C38D1 | 8.33 (23.90) |
  Cognitive Functioning C39D1: number analyzed (Participants) | 9 | 0
  Cognitive Functioning C39D1 | 1.85 (13.03) |
  Cognitive Functioning 30 day follow up: number analyzed (Participants) | 57 | 78
  Cognitive Functioning 30 day follow up | -2.63 (18.84) | -4.27 (20.18)
  Cognitive Functioning 90 day follow up: number analyzed (Participants) | 61 | 79
  Cognitive Functioning 90 day follow up | -7.65 (17.37) | -2.32 (20.28)
  Social Functioning Baseline | 79.42 (22.16) | 79.55 (23.48)
  Social Functioning C2D1: number analyzed (Participants) | 208 | 217
  Social Functioning C2D1 | 0.88 (21.31) | -1.61 (20.88)
  Social Functioning C3D1: number analyzed (Participants) | 182 | 197
  Social Functioning C3D1 | -1.47 (23.65) | -1.44 (22.70)
  Social Functioning C4D1: number analyzed (Participants) | 169 | 169
  Social Functioning C4D1 | 0.79 (23.77) | 1.97 (21.73)
  Social Functioning C5D1: number analyzed (Participants) | 159 | 165
  Social Functioning C5D1 | 2.20 (25.58) | 0.20 (22.31)
  Social Functioning C6D1: number analyzed (Participants) | 149 | 146
  Social Functioning C6D1 | -0.78 (25.29) | -1.37 (22.53)
  Social Functioning C7D1: number analyzed (Participants) | 120 | 126
  Social Functioning C7D1 | -0.97 (26.22) | -0.66 (24.71)
  Social Functioning C8D1: number analyzed (Participants) | 108 | 110
  Social Functioning C8D1 | -0.93 (27.33) | -2.12 (23.58)
  Social Functioning C9D1: number analyzed (Participants) | 102 | 103
  Social Functioning C9D1 | -0.98 (24.01) | -0.32 (24.47)
  Social Functioning C10D1: number analyzed (Participants) | 85 | 79
  Social Functioning C10D1 | 2.55 (25.39) | -0.84 (27.20)
  Social Functioning C11D1: number analyzed (Participants) | 81 | 71
  Social Functioning C11D1 | 3.29 (23.19) | -2.58 (25.14)
  Social Functioning C12D1: number analyzed (Participants) | 75 | 57
  Social Functioning C12D1 | 3.33 (23.09) | -1.75 (28.12)
  Social Functioning C13D1: number analyzed (Participants) | 60 | 48
  Social Functioning C13D1 | 3.89 (24.43) | -0.35 (23.19)
  Social Functioning C14D1: number analyzed (Participants) | 55 | 44
  Social Functioning C14D1 | 2.12 (20.80) | 1.52 (24.86)
  Social Functioning C15D1: number analyzed (Participants) | 51 | 36
  Social Functioning C15D1 | 1.63 (22.42) | -2.78 (23.06)
  Social Functioning C16D1: number analyzed (Participants) | 48 | 31
  Social Functioning C16D1 | 4.86 (20.03) | 1.08 (19.21)
  Social Functioning C17D1: number analyzed (Participants) | 43 | 25
  Social Functioning C17D1 | 5.43 (18.45) | 3.33 (15.96)
  Social Functioning C18D1: number analyzed (Participants) | 41 | 21
  Social Functioning C18D1 | 0.81 (22.96) | 2.38 (16.90)
  Social Functioning C19D1: number analyzed (Participants) | 40 | 20
  Social Functioning C19D1 | 5.42 (19.02) | 8.33 (20.59)
  Social Functioning C20D1: number analyzed (Participants) | 39 | 19
  Social Functioning C20D1 | 2.56 (21.81) | 7.02 (20.27)
  Social Functioning C21D1: number analyzed (Participants) | 36 | 20
  Social Functioning C21D1 | 2.31 (21.88) | 4.17 (17.83)
  Social Functioning C22D1: number analyzed (Participants) | 31 | 17
  Social Functioning C22D1 | 5.91 (21.32) | 4.90 (15.33)
  Social Functioning C23D1: number analyzed (Participants) | 31 | 16
  Social Functioning C23D1 | 4.30 (24.33) | 8.33 (18.26)
  Social Functioning C24D1: number analyzed (Participants) | 29 | 12
  Social Functioning C24D1 | 4.02 (23.84) | -1.39 (15.01)
  Social Functioning C25D1: number analyzed (Participants) | 28 | 12
  Social Functioning C25D1 | 4.76 (21.21) | -2.78 (15.62)
  Social Functioning C26D1: number analyzed (Participants) | 26 | 9
  Social Functioning C26D1 | 5.77 (23.54) | 3.70 (24.69)
  Social Functioning C27D1: number analyzed (Participants) | 25 | 10
  Social Functioning C27D1 | 4.00 (25.59) | 5.00 (15.81)
  Social Functioning C28D1: number analyzed (Participants) | 21 | 11
  Social Functioning C28D1 | 4.76 (29.88) | 3.03 (16.36)
  Social Functioning C29D1: number analyzed (Participants) | 22 | 12
  Social Functioning C29D1 | 3.03 (26.55) | 0.00 (21.32)
  Social Functioning C30D1: number analyzed (Participants) | 20 | 0
  Social Functioning C30D1 | 3.33 (28.41) |
  Social Functioning C31D1: number analyzed (Participants) | 20 | 0
  Social Functioning C31D1 | 3.33 (27.36) |
  Social Functioning C32D1: number analyzed (Participants) | 18 | 0
  Social Functioning C32D1 | 0.93 (29.41) |
  Social Functioning C33D1: number analyzed (Participants) | 15 | 0
  Social Functioning C33D1 | 3.33 (34.04) |
  Social Functioning C34D1: number analyzed (Participants) | 12 | 0
  Social Functioning C34D1 | 5.56 (35.06) |
  Social Functioning C35D1: number analyzed (Participants) | 13 | 0
  Social Functioning C35D1 | 2.56 (32.52) |
  Social Functioning C36D1: number analyzed (Participants) | 12 | 0
  Social Functioning C36D1 | 5.56 (33.58) |
  Social Functioning C37D1: number analyzed (Participants) | 11 | 0
  Social Functioning C37D1 | 6.06 (36.72) |
  Social Functioning C38D1: number analyzed (Participants) | 10 | 0
  Social Functioning C38D1 | 13.33 (31.23) |
  Social Functioning C39D1: number analyzed (Participants) | 9 | 0
  Social Functioning C39D1 | 0.00 (33.33) |
  Social Functioning 30 day follow up: number analyzed (Participants) | 57 | 78
  Social Functioning 30 day follow up | -4.09 (28.22) | -12.82 (26.03)
  Social Functioning 90 day follow up: number analyzed (Participants) | 61 | 79
  Social Functioning 90 day follow up | 0.27 (24.05) | -8.23 (26.40)
  Fatigue Baseline | 26.29 (22.00) | 27.55 (22.43)
  Fatigue C2D1: number analyzed (Participants) | 208 | 217
  Fatigue C2D1 | 1.66 (19.69) | 0.15 (19.11)
  Fatigue C3D1: number analyzed (Participants) | 182 | 197
  Fatigue C3D1 | 3.17 (21.71) | 0.96 (21.26)
  Fatigue C4D1: number analyzed (Participants) | 169 | 169
  Fatigue C4D1 | 1.05 (21.93) | -0.46 (22.03)
  Fatigue C5D1: number analyzed (Participants) | 159 | 165
  Fatigue C5D1 | 1.40 (23.21) | -0.81 (23.52)
  Fatigue C6D1: number analyzed (Participants) | 149 | 146
  Fatigue C6D1 | 2.83 (21.07) | 0.91 (25.25)
  Fatigue C7D1: number analyzed (Participants) | 120 | 126
  Fatigue C7D1 | 1.11 (20.99) | -1.06 (23.11)
  Fatigue C8D1: number analyzed (Participants) | 108 | 110
  Fatigue C8D1 | 4.94 (20.34) | 0.10 (23.05)
  Fatigue C9D1: number analyzed (Participants) | 102 | 103
  Fatigue C9D1 | 1.96 (24.94) | -0.86 (23.06)
  Fatigue C10D1: number analyzed (Participants) | 85 | 79
  Fatigue C10D1 | 1.57 (25.67) | -0.42 (24.81)
  Fatigue C11D1: number analyzed (Participants) | 81 | 71
  Fatigue C11D1 | -0.14 (22.53) | -0.31 (24.34)
  Fatigue C12D1: number analyzed (Participants) | 75 | 57
  Fatigue C12D1 | -0.89 (24.08) | 0.00 (23.19)
  Fatigue C13D1: number analyzed (Participants) | 60 | 48
  Fatigue C13D1 | -3.70 (25.03) | 0.00 (20.76)
  Fatigue C14D1: number analyzed (Participants) | 55 | 44
  Fatigue C14D1 | -2.22 (19.99) | -0.76 (19.82)
  Fatigue C15D1: number analyzed (Participants) | 51 | 36
  Fatigue C15D1 | -3.27 (21.12) | -0.62 (17.20)
  Fatigue C16D1: number analyzed (Participants) | 48 | 31
  Fatigue C16D1 | -4.63 (21.60) | -2.15 (17.55)
  Fatigue C17D1: number analyzed (Participants) | 43 | 25
  Fatigue C17D1 | -2.07 (18.98) | -1.78 (18.61)
  Fatigue C18D1: number analyzed (Participants) | 41 | 21
  Fatigue C18D1 | -0.81 (17.10) | -7.94 (17.26)
  Fatigue C19D1: number analyzed (Participants) | 40 | 20
  Fatigue C19D1 | -1.11 (17.93) | -4.44 (15.46)
  Fatigue C20D1: number analyzed (Participants) | 39 | 19
  Fatigue C20D1 | 0.57 (16.51) | -4.68 (18.64)
  Fatigue C21D1: number analyzed (Participants) | 36 | 20
  Fatigue C21D1 | 1.23 (16.75) | -3.33 (18.77)
  Fatigue C22D1: number analyzed (Participants) | 31 | 17
  Fatigue C22D1 | -2.87 (19.02) | -3.27 (18.33)
  Fatigue C23D1: number analyzed (Participants) | 31 | 16
  Fatigue C23D1 | -1.43 (17.62) | -4.17 (22.18)
  Fatigue C24D1: number analyzed (Participants) | 29 | 12
  Fatigue C24D1 | -1.15 (17.65) | -3.70 (19.73)
  Fatigue C25D1: number analyzed (Participants) | 28 | 12
  Fatigue C25D1 | -3.17 (18.36) | -0.93 (17.38)
  Fatigue C26D1: number analyzed (Participants) | 26 | 9
  Fatigue C26D1 | -1.71 (21.70) | 0.00 (11.11)
  Fatigue C27D1: number analyzed (Participants) | 25 | 10
  Fatigue C27D1 | -3.11 (14.17) | 2.22 (15.54)
  Fatigue C28D1: number analyzed (Participants) | 21 | 11
  Fatigue C28D1 | -2.65 (16.06) | 8.08 (13.23)
  Fatigue C29D1: number analyzed (Participants) | 22 | 12
  Fatigue C29D1 | -3.54 (14.70) | 5.56 (18.65)
  Fatigue C30D1: number analyzed (Participants) | 20 | 0
  Fatigue C30D1 | -2.78 (13.90) |
  Fatigue C31D1: number analyzed (Participants) | 20 | 0
  Fatigue C31D1 | -2.22 (17.14) |
  Fatigue C32D1: number analyzed (Participants) | 18 | 0
  Fatigue C32D1 | -5.56 (18.77) |
  Fatigue C33D1: number analyzed (Participants) | 15 | 0
  Fatigue C33D1 | -8.15 (19.91) |
  Fatigue C34D1: number analyzed (Participants) | 12 | 0
  Fatigue C34D1 | -12.04 (18.63) |
  Fatigue C35D1: number analyzed (Participants) | 13 | 0
  Fatigue C35D1 | -10.26 (12.39) |
  Fatigue C36D1: number analyzed (Participants) | 12 | 0
  Fatigue C36D1 | -12.04 (10.00) |
  Fatigue C37D1: number analyzed (Participants) | 11 | 0
  Fatigue C37D1 | -12.12 (14.45) |
  Fatigue C38D1: number analyzed (Participants) | 10 | 0
  Fatigue C38D1 | -12.22 (21.24) |
  Fatigue C39D1: number analyzed (Participants) | 9 | 0
  Fatigue C39D1 | -7.41 (19.25) |
  Fatigue 30 day follow up: number analyzed (Participants) | 57 | 78
  Fatigue 30 day follow up | 11.50 (23.09) | 13.68 (27.15)
  Fatigue 90 day follow up: number analyzed (Participants) | 61 | 79
  Fatigue 90 day follow up | 11.84 (21.55) | 7.31 (22.00)
  Nausea and Vomiting Baseline | 10.49 (18.08) | 15.08 (23.20)
  Nausea and Vomiting C2D1: number analyzed (Participants) | 208 | 217
  Nausea and Vomiting C2D1 | 6.41 (19.77) | -0.92 (20.77)
  Nausea and Vomiting C3D1: number analyzed (Participants) | 182 | 197
  Nausea and Vomiting C3D1 | 5.86 (19.88) | 0.17 (22.21)
  Nausea and Vomiting C4D1: number analyzed (Participants) | 169 | 169
  Nausea and Vomiting C4D1 | 4.73 (20.67) | -2.76 (22.98)
  Nausea and Vomiting C5D1: number analyzed (Participants) | 159 | 165
  Nausea and Vomiting C5D1 | 4.93 (21.01) | -3.74 (25.06)
  Nausea and Vomiting C6D1: number analyzed (Participants) | 149 | 146
  Nausea and Vomiting C6D1 | 6.04 (20.25) | -1.60 (24.71)
  Nausea and Vomiting C7D1: number analyzed (Participants) | 120 | 126
  Nausea and Vomiting C7D1 | 1.25 (19.94) | -2.91 (24.59)
  Nausea and Vomiting C8D1: number analyzed (Participants) | 108 | 110
  Nausea and Vomiting C8D1 | 3.09 (20.14) | -6.97 (23.83)
  Nausea and Vomiting C9D1: number analyzed (Participants) | 102 | 103
  Nausea and Vomiting C9D1 | 1.80 (20.83) | -6.15 (20.74)
  Nausea and Vomiting C10D1: number analyzed (Participants) | 85 | 79
  Nausea and Vomiting C10D1 | 0.39 (20.25) | -7.17 (24.99)
  Nausea and Vomiting C11D1: number analyzed (Participants) | 81 | 71
  Nausea and Vomiting C11D1 | -1.65 (19.65) | -6.81 (24.17)
  Nausea and Vomiting C12D1: number analyzed (Participants) | 75 | 57
  Nausea and Vomiting C12D1 | -1.11 (19.82) | -2.34 (25.48)
  Nausea and Vomiting C13D1: number analyzed (Participants) | 60 | 48
  Nausea and Vomiting C13D1 | -3.33 (20.54) | -7.99 (23.82)
  Nausea and Vomiting C14D1: number analyzed (Participants) | 55 | 44
  Nausea and Vomiting C14D1 | -1.21 (19.73) | -4.17 (21.00)
  Nausea and Vomiting C15D1: number analyzed (Participants) | 51 | 36
  Nausea and Vomiting C15D1 | -2.94 (18.17) | -5.56 (20.31)
  Nausea and Vomiting C16D1: number analyzed (Participants) | 48 | 31
  Nausea and Vomiting C16D1 | -1.04 (20.17) | -5.91 (20.43)
  Nausea and Vomiting C17D1: number analyzed (Participants) | 43 | 25
  Nausea and Vomiting C17D1 | -1.94 (18.62) | 2.67 (13.33)
  Nausea and Vomiting C18D1: number analyzed (Participants) | 41 | 21
  Nausea and Vomiting C18D1 | 0.81 (20.40) | -4.76 (11.95)
  Nausea and Vomiting C19D1: number analyzed (Participants) | 40 | 20
  Nausea and Vomiting C19D1 | 0.00 (20.32) | -4.17 (11.94)
  Nausea and Vomiting C20D1: number analyzed (Participants) | 39 | 19
  Nausea and Vomiting C20D1 | -0.85 (19.10) | -4.39 (12.22)
  Nausea and Vomiting C21D1: number analyzed (Participants) | 36 | 20
  Nausea and Vomiting C21D1 | 0.00 (19.92) | -3.33 (11.60)
  Nausea and Vomiting C22D1: number analyzed (Participants) | 31 | 17
  Nausea and Vomiting C22D1 | -2.69 (20.23) | -5.88 (13.10)
  Nausea and Vomiting C23D1: number analyzed (Participants) | 31 | 16
  Nausea and Vomiting C23D1 | -3.76 (21.39) | -7.29 (12.12)
  Nausea and Vomiting C24D1: number analyzed (Participants) | 29 | 12
  Nausea and Vomiting C24D1 | -3.45 (20.11) | -1.39 (11.14)
  Nausea and Vomiting C25D1: number analyzed (Participants) | 28 | 12
  Nausea and Vomiting C25D1 | -4.17 (20.60) | -6.94 (13.22)
  Nausea and Vomiting C26D1: number analyzed (Participants) | 26 | 9
  Nausea and Vomiting C26D1 | -4.49 (20.85) | -1.85 (24.22)
  Nausea and Vomiting C27D1: number analyzed (Participants) | 25 | 10
  Nausea and Vomiting C27D1 | -4.67 (20.14) | -5.00 (15.81)
  Nausea and Vomiting C28D1: number analyzed (Participants) | 21 | 11
  Nausea and Vomiting C28D1 | -0.79 (23.85) | -3.03 (14.56)
  Nausea and Vomiting C29D1: number analyzed (Participants) | 22 | 12
  Nausea and Vomiting C29D1 | -3.79 (21.78) | -9.72 (13.22)
  Nausea and Vomiting C30D1: number analyzed (Participants) | 20 | 0
  Nausea and Vomiting C30D1 | -3.33 (21.36) |
  Nausea and Vomiting C31D1: number analyzed (Participants) | 20 | 0
  Nausea and Vomiting C31D1 | -4.17 (23.49) |
  Nausea and Vomiting C32D1: number analyzed (Participants) | 18 | 0
  Nausea and Vomiting C32D1 | -2.78 (25.72) |
  Nausea and Vomiting C33D1: number analyzed (Participants) | 15 | 0
  Nausea and Vomiting C33D1 | -8.89 (21.70) |
  Nausea and Vomiting C34D1: number analyzed (Participants) | 12 | 0
  Nausea and Vomiting C34D1 | -8.33 (25.13) |
  Nausea and Vomiting C35D1: number analyzed (Participants) | 13 | 0
  Nausea and Vomiting C35D1 | -6.41 (25.04) |
  Nausea and Vomiting C36D1: number analyzed (Participants) | 12 | 0
  Nausea and Vomiting C36D1 | -6.94 (25.08) |
  Nausea and Vomiting C37D1: number analyzed (Participants) | 11 | 0
  Nausea and Vomiting C37D1 | -9.09 (20.23) |
  Nausea and Vomiting C38D1: number analyzed (Participants) | 10 | 0
  Nausea and Vomiting C38D1 | -6.67 (14.05) |
  Nausea and Vomiting C39D1: number analyzed (Participants) | 9 | 0
  Nausea and Vomiting C39D1 | -5.56 (8.33) |
  Nausea and Vomiting 30 day follow up: number analyzed (Participants) | 57 | 78
  Nausea and Vomiting 30 day follow up | 4.39 (19.80) | 0.21 (24.25)
  Nausea and Vomiting 90 day follow up: number analyzed (Participants) | 61 | 79
  Nausea and Vomiting 90 day follow up | 7.38 (21.20) | -1.05 (26.06)
  Pain Baseline | 21.67 (22.14) | 24.10 (23.71)
  Pain C2D1: number analyzed (Participants) | 208 | 217
  Pain C2D1 | -4.17 (22.43) | -4.61 (20.08)
  Pain C3D1: number analyzed (Participants) | 182 | 197
  Pain C3D1 | -5.40 (21.16) | -3.38 (22.77)
  Pain C4D1: number analyzed (Participants) | 169 | 169
  Pain C4D1 | -7.10 (21.18) | -7.40 (22.41)
  Pain C5D1: number analyzed (Participants) | 159 | 165
  Pain C5D1 | -4.82 (22.06) | -6.26 (26.05)
  Pain C6D1: number analyzed (Participants) | 149 | 146
  Pain C6D1 | -3.13 (19.79) | -6.85 (26.09)
  Pain C7D1: number analyzed (Participants) | 120 | 126
  Pain C7D1 | -6.39 (22.16) | -7.67 (22.57)
  Pain C8D1: number analyzed (Participants) | 108 | 110
  Pain C8D1 | -4.17 (22.22) | -5.61 (24.96)
  Pain C9D1: number analyzed (Participants) | 102 | 103
  Pain C9D1 | -5.07 (21.72) | -8.09 (24.46)
  Pain C10D1: number analyzed (Participants) | 85 | 79
  Pain C10D1 | -4.12 (22.11) | -6.33 (25.50)
  Pain C11D1: number analyzed (Participants) | 81 | 71
  Pain C11D1 | -6.38 (21.01) | -6.34 (26.78)
  Pain C12D1: number analyzed (Participants) | 75 | 57
  Pain C12D1 | -4.44 (22.48) | -7.02 (24.99)
  Pain C13D1: number analyzed (Participants) | 60 | 48
  Pain C13D1 | -6.39 (23.98) | -7.64 (24.54)
  Pain C14D1: number analyzed (Participants) | 55 | 44
  Pain C14D1 | -5.76 (22.27) | -6.06 (24.14)
  Pain C15D1: number analyzed (Participants) | 51 | 36
  Pain C15D1 | -6.54 (19.17) | -7.41 (21.25)
  Pain C16D1: number analyzed (Participants) | 48 | 31
  Pain C16D1 | -6.25 (19.64) | -6.45 (23.04)
  Pain C17D1: number analyzed (Participants) | 43 | 25
  Pain C17D1 | -5.04 (19.43) | -7.33 (25.95)
  Pain C18D1: number analyzed (Participants) | 41 | 21
  Pain C18D1 | -1.63 (18.18) | -11.90 (27.96)
  Pain C19D1: number analyzed (Participants) | 40 | 20
  Pain C19D1 | -2.50 (18.32) | -7.50 (26.20)
  Pain C20D1: number analyzed (Participants) | 39 | 19
  Pain C20D1 | -0.85 (16.64) | -8.77 (30.11)
  Pain C21D1: number analyzed (Participants) | 36 | 20
  Pain C21D1 | -2.31 (19.58) | -11.67 (29.17)
  Pain C22D1: number analyzed (Participants) | 31 | 17
  Pain C22D1 | -2.69 (18.31) | -12.75 (30.35)
  Pain C23D1: number analyzed (Participants) | 31 | 16
  Pain C23D1 | -3.76 (18.11) | -15.63 (30.10)
  Pain C24D1: number analyzed (Participants) | 29 | 12
  Pain C24D1 | -4.02 (18.18) | -8.33 (29.73)
  Pain C25D1: number analyzed (Participants) | 28 | 12
  Pain C25D1 | -1.19 (21.24) | -11.11 (29.59)
  Pain C26D1: number analyzed (Participants) | 26 | 9
  Pain C26D1 | -3.85 (19.61) | -9.26 (18.84)
  Pain C27D1: number analyzed (Participants) | 25 | 10
  Pain C27D1 | -4.00 (20.57) | -6.67 (23.83)
  Pain C28D1: number analyzed (Participants) | 21 | 11
  Pain C28D1 | -4.76 (21.18) | -3.03 (19.46)
  Pain C29D1: number analyzed (Participants) | 22 | 12
  Pain C29D1 | -3.79 (21.16) | -11.11 (23.92)
  Pain C30D1: number analyzed (Participants) | 20 | 0
  Pain C30D1 | -6.67 (19.79) |
  Pain C31D1: number analyzed (Participants) | 20 | 0
  Pain C31D1 | -6.67 (21.90) |
  Pain C32D1: number analyzed (Participants) | 18 | 0
  Pain C32D1 | -6.48 (22.97) |
  Pain C33D1: number analyzed (Participants) | 15 | 0
  Pain C33D1 | -10.00 (22.54) |
  Pain C34D1: number analyzed (Participants) | 12 | 0
  Pain C34D1 | -13.89 (21.12) |
  Pain C35D1: number analyzed (Participants) | 13 | 0
  Pain C35D1 | -10.26 (22.09) |
  Pain C36D1: number analyzed (Participants) | 12 | 0
  Pain C36D1 | -12.50 (21.47) |
  Pain C37D1: number analyzed (Participants) | 11 | 0
  Pain C37D1 | -12.12 (23.68) |
  Pain C38D1: number analyzed (Participants) | 10 | 0
  Pain C38D1 | -5.00 (24.91) |
  Pain C39D1: number analyzed (Participants) | 9 | 0
  Pain C39D1 | -9.26 (16.90) |
  Pain 30 day follow up: number analyzed (Participants) | 57 | 78
  Pain 30 day follow up | 4.97 (27.45) | 8.76 (26.42)
  Pain 90 day follow up: number analyzed (Participants) | 61 | 79
  Pain 90 day follow up | 4.37 (22.55) | 2.11 (22.70)
  Dyspnoea Baseline | 9.74 (17.96) | 10.88 (19.35)
  Dyspnoea C2D1: number analyzed (Participants) | 208 | 217
  Dyspnoea C2D1 | 2.24 (15.89) | -0.77 (17.99)
  Dyspnoea C3D1: number analyzed (Participants) | 182 | 197
  Dyspnoea C3D1 | -0.37 (16.80) | 0.51 (22.20)
  Dyspnoea C4D1: number analyzed (Participants) | 169 | 169
  Dyspnoea C4D1 | 0.00 (16.67) | -0.39 (23.28)
  Dyspnoea C5D1: number analyzed (Participants) | 159 | 165
  Dyspnoea C5D1 | -0.42 (19.48) | -2.22 (23.03)
  Dyspnoea C6D1: number analyzed (Participants) | 149 | 146
  Dyspnoea C6D1 | 1.12 (19.54) | 0.00 (21.80)
  Dyspnoea C7D1: number analyzed (Participants) | 120 | 126
  Dyspnoea C7D1 | 1.67 (20.20) | -0.53 (22.70)
  Dyspnoea C8D1: number analyzed (Participants) | 108 | 110
  Dyspnoea C8D1 | 1.85 (19.25) | 2.12 (23.58)
  Dyspnoea C9D1: number analyzed (Participants) | 102 | 103
  Dyspnoea C9D1 | 0.65 (18.15) | -2.27 (20.49)
  Dyspnoea C10D1: number analyzed (Participants) | 85 | 79
  Dyspnoea C10D1 | 1.18 (20.86) | -0.42 (24.16)
  Dyspnoea C11D1: number analyzed (Participants) | 81 | 71
  Dyspnoea C11D1 | 0.41 (20.07) | -3.29 (21.20)
  Dyspnoea C12D1: number analyzed (Participants) | 75 | 57
  Dyspnoea C12D1 | -1.33 (20.09) | -2.92 (19.19)
  Dyspnoea C13D1: number analyzed (Participants) | 60 | 48
  Dyspnoea C13D1 | -0.56 (23.36) | -2.78 (21.56)
  Dyspnoea C14D1: number analyzed (Participants) | 55 | 44
  Dyspnoea C14D1 | -0.61 (20.78) | -4.55 (19.81)
  Dyspnoea C15D1: number analyzed (Participants) | 51 | 36
  Dyspnoea C15D1 | 0.00 (17.64) | -4.63 (16.24)
  Dyspnoea C16D1: number analyzed (Participants) | 48 | 31
  Dyspnoea C16D1 | -0.69 (16.11) | -3.23 (21.70)
  Dyspnoea C17D1: number analyzed (Participants) | 43 | 25
  Dyspnoea C17D1 | 0.00 (16.27) | -6.67 (21.52)
  Dyspnoea C18D1: number analyzed (Participants) | 41 | 21
  Dyspnoea C18D1 | 1.63 (16.59) | -9.52 (18.69)
  Dyspnoea C19D1: number analyzed (Participants) | 40 | 20
  Dyspnoea C19D1 | 0.00 (16.88) | -11.67 (19.57)
  Dyspnoea C20D1: number analyzed (Participants) | 39 | 19
  Dyspnoea C20D1 | 2.56 (19.32) | -10.53 (22.37)
  Dyspnoea C21D1: number analyzed (Participants) | 36 | 20
  Dyspnoea C21D1 | 0.93 (16.88) | -10.00 (19.04)
  Dyspnoea C22D1: number analyzed (Participants) | 31 | 17
  Dyspnoea C22D1 | 1.08 (20.15) | -9.80 (22.87)
  Dyspnoea C23D1: number analyzed (Participants) | 31 | 16
  Dyspnoea C23D1 | 0.00 (14.91) | -8.33 (22.77)
  Dyspnoea C24D1: number analyzed (Participants) | 29 | 12
  Dyspnoea C24D1 | 0.00 (17.82) | -5.56 (19.25)
  Dyspnoea C25D1: number analyzed (Participants) | 28 | 12
  Dyspnoea C25D1 | 0.00 (20.29) | -5.56 (19.25)
  Dyspnoea C26D1: number analyzed (Participants) | 26 | 9
  Dyspnoea C26D1 | -3.85 (14.38) | -7.41 (14.70)
  Dyspnoea C27D1: number analyzed (Participants) | 25 | 10
  Dyspnoea C27D1 | 2.67 (16.44) | -6.67 (14.05)
  Dyspnoea C28D1: number analyzed (Participants) | 21 | 11
  Dyspnoea C28D1 | -1.59 (16.59) | -9.09 (21.56)
  Dyspnoea C29D1: number analyzed (Participants) | 22 | 12
  Dyspnoea C29D1 | 7.58 (27.08) | -11.11 (21.71)
  Dyspnoea C30D1: number analyzed (Participants) | 20 | 0
  Dyspnoea C30D1 | 0.00 (18.73) |
  Dyspnoea C31D1: number analyzed (Participants) | 20 | 0
  Dyspnoea C31D1 | -1.67 (22.88) |
  Dyspnoea C32D1: number analyzed (Participants) | 18 | 0
  Dyspnoea C32D1 | 0.00 (22.87) |
  Dyspnoea C33D1: number analyzed (Participants) | 15 | 0
  Dyspnoea C33D1 | 2.22 (23.46) |
  Dyspnoea C34D1: number analyzed (Participants) | 12 | 0
  Dyspnoea C34D1 | -8.33 (20.72) |
  Dyspnoea C35D1: number analyzed (Participants) | 13 | 0
  Dyspnoea C35D1 | -2.56 (21.35) |
  Dyspnoea C36D1: number analyzed (Participants) | 12 | 0
  Dyspnoea C36D1 | -5.56 (19.25) |
  Dyspnoea C37D1: number analyzed (Participants) | 11 | 0
  Dyspnoea C37D1 | -9.09 (21.56) |
  Dyspnoea C38D1: number analyzed (Participants) | 10 | 0
  Dyspnoea C38D1 | -3.33 (18.92) |
  Dyspnoea C39D1: number analyzed (Participants) | 9 | 0
  Dyspnoea C39D1 | -3.70 (20.03) |
  Dyspnoea 30 day follow up: number analyzed (Participants) | 57 | 78
  Dyspnoea 30 day follow up | 3.51 (16.29) | 4.27 (23.02)
  Dyspnoea 90 day follow up: number analyzed (Participants) | 61 | 79
  Dyspnoea 90 day follow up | 2.73 (15.27) | 2.53 (24.33)
  Insomnia Baseline | 20.99 (27.16) | 24.79 (26.66)
  Insomnia C2D1: number analyzed (Participants) | 208 | 217
  Insomnia C2D1 | -1.44 (27.47) | -1.54 (27.55)
  Insomnia C3D1: number analyzed (Participants) | 182 | 197
  Insomnia C3D1 | -0.55 (28.14) | -2.54 (28.56)
  Insomnia C4D1: number analyzed (Participants) | 169 | 169
  Insomnia C4D1 | -4.73 (28.47) | -5.13 (27.94)
  Insomnia C5D1: number analyzed (Participants) | 159 | 165
  Insomnia C5D1 | -2.73 (28.06) | -4.44 (28.16)
  Insomnia C6D1: number analyzed (Participants) | 149 | 146
  Insomnia C6D1 | -5.15 (28.40) | -2.51 (30.35)
  Insomnia C7D1: number analyzed (Participants) | 120 | 126
  Insomnia C7D1 | -5.28 (28.34) | -2.91 (31.28)
  Insomnia C8D1: number analyzed (Participants) | 108 | 110
  Insomnia C8D1 | 0.31 (29.00) | -4.85 (25.48)
  Insomnia C9D1: number analyzed (Participants) | 102 | 103
  Insomnia C9D1 | -4.90 (29.44) | -4.21 (27.88)
  Insomnia C10D1: number analyzed (Participants) | 85 | 79
  Insomnia C10D1 | -5.49 (29.48) | -0.42 (28.49)
  Insomnia C11D1: number analyzed (Participants) | 81 | 71
  Insomnia C11D1 | -2.47 (29.71) | 0.94 (30.33)
  Insomnia C12D1: number analyzed (Participants) | 75 | 57
  Insomnia C12D1 | -0.89 (27.39) | -0.58 (29.87)
  Insomnia C13D1: number analyzed (Participants) | 60 | 48
  Insomnia C13D1 | -3.33 (24.32) | 1.39 (33.66)
  Insomnia C14D1: number analyzed (Participants) | 55 | 44
  Insomnia C14D1 | 0.61 (27.59) | -0.76 (33.32)
  Insomnia C15D1: number analyzed (Participants) | 51 | 36
  Insomnia C15D1 | 5.23 (23.45) | 1.85 (30.80)
  Insomnia C16D1: number analyzed (Participants) | 48 | 31
  Insomnia C16D1 | 0.00 (25.73) | 6.45 (24.97)
  Insomnia C17D1: number analyzed (Participants) | 43 | 25
  Insomnia C17D1 | 1.55 (25.15) | 12.00 (31.74)
  Insomnia C18D1: number analyzed (Participants) | 41 | 21
  Insomnia C18D1 | 0.00 (24.72) | 4.76 (24.23)
  Insomnia C19D1: number analyzed (Participants) | 40 | 20
  Insomnia C19D1 | 0.00 (21.35) | 6.67 (38.39)
  Insomnia C20D1: number analyzed (Participants) | 39 | 19
  Insomnia C20D1 | -0.85 (17.91) | 7.02 (23.78)
  Insomnia C21D1: number analyzed (Participants) | 36 | 20
  Insomnia C21D1 | 0.00 (19.52) | 8.33 (30.35)
  Insomnia C22D1: number analyzed (Participants) | 31 | 17
  Insomnia C22D1 | -5.38 (17.42) | 9.80 (34.89)
  Insomnia C23D1: number analyzed (Participants) | 31 | 16
  Insomnia C23D1 | -3.23 (15.76) | 4.17 (34.16)
  Insomnia C24D1: number analyzed (Participants) | 29 | 12
  Insomnia C24D1 | 0.00 (17.82) | 0.00 (24.62)
  Insomnia C25D1: number analyzed (Participants) | 28 | 12
  Insomnia C25D1 | -2.38 (20.14) | 2.78 (22.29)
  Insomnia C26D1: number analyzed (Participants) | 26 | 9
  Insomnia C26D1 | -2.56 (18.67) | 3.70 (20.03)
  Insomnia C27D1: number analyzed (Participants) | 25 | 10
  Insomnia C27D1 | -4.00 (17.53) | 6.67 (21.08)
  Insomnia C28D1: number analyzed (Participants) | 21 | 11
  Insomnia C28D1 | -1.59 (19.65) | 15.15 (27.34)
  Insomnia C29D1: number analyzed (Participants) | 22 | 12
  Insomnia C29D1 | 1.52 (21.77) | 8.33 (25.13)
  Insomnia C30D1: number analyzed (Participants) | 20 | 0
  Insomnia C30D1 | -1.67 (17.01) |
  Insomnia C31D1: number analyzed (Participants) | 20 | 0
  Insomnia C31D1 | 1.67 (17.01) |
  Insomnia C32D1: number analyzed (Participants) | 18 | 0
  Insomnia C32D1 | 0.00 (22.87) |
  Insomnia C33D1: number analyzed (Participants) | 15 | 0
  Insomnia C33D1 | -2.22 (19.79) |
  Insomnia C34D1: number analyzed (Participants) | 12 | 0
  Insomnia C34D1 | -2.78 (22.29) |
  Insomnia C35D1: number analyzed (Participants) | 13 | 0
  Insomnia C35D1 | 0.00 (23.57) |
  Insomnia C36D1: number analyzed (Participants) | 12 | 0
  Insomnia C36D1 | -2.78 (17.16) |
  Insomnia C37D1: number analyzed (Participants) | 11 | 0
  Insomnia C37D1 | 3.03 (23.35) |
  Insomnia C38D1: number analyzed (Participants) | 10 | 0
  Insomnia C38D1 | 6.67 (34.43) |
  Insomnia C39D1: number analyzed (Participants) | 9 | 0
  Insomnia C39D1 | 7.41 (22.22) |
  Insomnia 30 day follow up: number analyzed (Participants) | 57 | 78
  Insomnia 30 day follow up | 6.43 (30.50) | 8.55 (36.21)
  Insomnia 90 day follow up: number analyzed (Participants) | 61 | 79
  Insomnia 90 day follow up | 6.56 (22.62) | 0.42 (28.99)
  Appetite Loss Baseline | 26.20 (29.91) | 24.66 (29.17)
  Appetite Loss C2D1: number analyzed (Participants) | 208 | 217
  Appetite Loss C2D1 | 3.69 (31.97) | -2.61 (27.37)
  Appetite Loss C3D1: number analyzed (Participants) | 182 | 197
  Appetite Loss C3D1 | 0.73 (34.86) | -2.71 (27.43)
  Appetite Loss C4D1: number analyzed (Participants) | 169 | 169
  Appetite Loss C4D1 | -3.55 (34.32) | -5.13 (33.13)
  Appetite Loss C5D1: number analyzed (Participants) | 159 | 165
  Appetite Loss C5D1 | -2.94 (36.24) | -4.44 (33.03)
  Appetite Loss C6D1: number analyzed (Participants) | 149 | 146
  Appetite Loss C6D1 | -0.22 (34.55) | -2.51 (33.47)
  Appetite Loss C7D1: number analyzed (Participants) | 120 | 126
  Appetite Loss C7D1 | -4.44 (37.41) | -6.88 (31.36)
  Appetite Loss C8D1: number analyzed (Participants) | 108 | 110
  Appetite Loss C8D1 | -1.23 (31.55) | -6.36 (32.71)
  Appetite Loss C9D1: number analyzed (Participants) | 102 | 103
  Appetite Loss C9D1 | -3.92 (36.72) | -7.12 (34.51)
  Appetite Loss C10D1: number analyzed (Participants) | 85 | 79
  Appetite Loss C10D1 | -3.92 (31.04) | -10.13 (32.62)
  Appetite Loss C11D1: number analyzed (Participants) | 81 | 71
  Appetite Loss C11D1 | -7.82 (31.30) | -12.21 (33.92)
  Appetite Loss C12D1: number analyzed (Participants) | 75 | 57
  Appetite Loss C12D1 | -8.00 (31.40) | -11.11 (30.43)
  Appetite Loss C13D1: number analyzed (Participants) | 60 | 48
  Appetite Loss C13D1 | -9.44 (36.36) | -12.50 (31.23)
  Appetite Loss C14D1: number analyzed (Participants) | 55 | 44
  Appetite Loss C14D1 | -12.12 (31.01) | -11.36 (30.45)
  Appetite Loss C15D1: number analyzed (Participants) | 51 | 36
  Appetite Loss C15D1 | -9.80 (30.03) | -11.11 (29.81)
  Appetite Loss C16D1: number analyzed (Participants) | 48 | 31
  Appetite Loss C16D1 | -9.72 (32.22) | -8.60 (32.17)
  Appetite Loss C17D1: number analyzed (Participants) | 43 | 25
  Appetite Loss C17D1 | -8.53 (32.61) | -6.67 (36.00)
  Appetite Loss C18D1: number analyzed (Participants) | 41 | 21
  Appetite Loss C18D1 | -12.20 (32.28) | -9.52 (35.19)
  Appetite Loss C19D1: number analyzed (Participants) | 40 | 20
  Appetite Loss C19D1 | -14.17 (30.09) | -15.00 (20.16)
  Appetite Loss C20D1: number analyzed (Participants) | 39 | 19
  Appetite Loss C20D1 | -7.69 (33.74) | -15.79 (30.16)
  Appetite Loss C21D1: number analyzed (Participants) | 36 | 20
  Appetite Loss C21D1 | -4.63 (33.00) | -10.00 (34.37)
  Appetite Loss C22D1: number analyzed (Participants) | 31 | 17
  Appetite Loss C22D1 | -10.75 (32.65) | -17.65 (31.44)
  Appetite Loss C23D1: number analyzed (Participants) | 31 | 16
  Appetite Loss C23D1 | -10.75 (30.29) | -14.58 (40.31)
  Appetite Loss C24D1: number analyzed (Participants) | 29 | 12
  Appetite Loss C24D1 | -13.79 (28.89) | -16.67 (33.33)
  Appetite Loss C25D1: number analyzed (Participants) | 28 | 12
  Appetite Loss C25D1 | -10.71 (30.16) | -16.67 (33.33)
  Appetite Loss C26D1: number analyzed (Participants) | 26 | 9
  Appetite Loss C26D1 | -12.82 (35.37) | -14.81 (17.57)
  Appetite Loss C27D1: number analyzed (Participants) | 25 | 10
  Appetite Loss C27D1 | -8.00 (30.85) | -10.00 (31.62)
  Appetite Loss C28D1: number analyzed (Participants) | 21 | 11
  Appetite Loss C28D1 | -14.29 (32.61) | 0.00 (29.81)
  Appetite Loss C29D1: number analyzed (Participants) | 22 | 12
  Appetite Loss C29D1 | -16.67 (28.64) | -11.11 (29.59)
  Appetite Loss C30D1: number analyzed (Participants) | 20 | 0
  Appetite Loss C30D1 | -10.00 (32.62) |
  Appetite Loss C31D1: number analyzed (Participants) | 20 | 0
  Appetite Loss C31D1 | -16.67 (31.53) |
  Appetite Loss C32D1: number analyzed (Participants) | 18 | 0
  Appetite Loss C32D1 | -14.81 (36.55) |
  Appetite Loss C33D1: number analyzed (Participants) | 15 | 0
  Appetite Loss C33D1 | -17.78 (37.52) |
  Appetite Loss C34D1: number analyzed (Participants) | 12 | 0
  Appetite Loss C34D1 | -27.78 (34.33) |
  Appetite Loss C35D1: number analyzed (Participants) | 13 | 0
  Appetite Loss C35D1 | -17.95 (35.00) |
  Appetite Loss C36D1: number analyzed (Participants) | 12 | 0
  Appetite Loss C36D1 | -19.44 (36.12) |
  Appetite Loss C37D1: number analyzed (Participants) | 11 | 0
  Appetite Loss C37D1 | -18.18 (37.61) |
  Appetite Loss C38D1: number analyzed (Participants) | 10 | 0
  Appetite Loss C38D1 | -23.33 (41.72) |
  Appetite Loss C39D1: number analyzed (Participants) | 9 | 0
  Appetite Loss C39D1 | -18.52 (37.68) |
  Appetite Loss 30 day follow up: number analyzed (Participants) | 57 | 78
  Appetite Loss 30 day follow up | 4.68 (38.03) | 6.41 (29.94)
  Appetite Loss 90 day follow up: number analyzed (Participants) | 61 | 79
  Appetite Loss 90 day follow up | 3.28 (38.83) | 0.84 (32.46)
  Constipation Baseline | 18.11 (26.09) | 17.63 (27.02)
  Constipation C2D1: number analyzed (Participants) | 208 | 217
  Constipation C2D1 | -0.64 (24.94) | -2.76 (25.10)
  Constipation C3D1: number analyzed (Participants) | 182 | 197
  Constipation C3D1 | -2.38 (26.23) | -5.25 (23.58)
  Constipation C4D1: number analyzed (Participants) | 169 | 169
  Constipation C4D1 | -4.73 (26.30) | -6.90 (29.07)
  Constipation C5D1: number analyzed (Participants) | 159 | 165
  Constipation C5D1 | -2.73 (25.97) | -4.65 (26.77)
  Constipation C6D1: number analyzed (Participants) | 149 | 146
  Constipation C6D1 | -5.82 (26.77) | -4.34 (29.36)
  Constipation C7D1: number analyzed (Participants) | 120 | 126
  Constipation C7D1 | -7.78 (26.19) | -2.12 (32.32)
  Constipation C8D1: number analyzed (Participants) | 108 | 110
  Constipation C8D1 | -4.63 (27.14) | -3.03 (31.13)
  Constipation C9D1: number analyzed (Participants) | 102 | 103
  Constipation C9D1 | -4.25 (22.82) | -5.50 (29.19)
  Constipation C10D1: number analyzed (Participants) | 85 | 79
  Constipation C10D1 | -6.27 (26.97) | -7.17 (30.97)
  Constipation C11D1: number analyzed (Participants) | 81 | 71
  Constipation C11D1 | -4.94 (28.44) | -3.29 (33.88)
  Constipation C12D1: number analyzed (Participants) | 75 | 57
  Constipation C12D1 | -6.22 (25.52) | -1.17 (26.70)
  Constipation C13D1: number analyzed (Participants) | 60 | 48
  Constipation C13D1 | -7.78 (25.58) | -3.47 (33.85)
  Constipation C14D1: number analyzed (Participants) | 55 | 44
  Constipation C14D1 | -6.06 (25.73) | -2.27 (28.21)
  Constipation C15D1: number analyzed (Participants) | 51 | 36
  Constipation C15D1 | -4.58 (27.50) | -3.70 (32.64)
  Constipation C16D1: number analyzed (Participants) | 48 | 31
  Constipation C16D1 | -2.78 (26.48) | -2.15 (33.26)
  Constipation C17D1: number analyzed (Participants) | 43 | 25
  Constipation C17D1 | -3.88 (27.42) | -1.33 (26.32)
  Constipation C18D1: number analyzed (Participants) | 41 | 21
  Constipation C18D1 | -5.69 (25.71) | -6.35 (29.10)
  Constipation C19D1: number analyzed (Participants) | 40 | 20
  Constipation C19D1 | -5.83 (23.74) | -6.67 (17.44)
  Constipation C20D1: number analyzed (Participants) | 39 | 19
  Constipation C20D1 | 0.00 (31.53) | -7.02 (26.24)
  Constipation C21D1: number analyzed (Participants) | 36 | 20
  Constipation C21D1 | 0.00 (26.43) | -5.00 (31.11)
  Constipation C22D1: number analyzed (Participants) | 31 | 17
  Constipation C22D1 | -2.15 (32.13) | 1.96 (24.92)
  Constipation C23D1: number analyzed (Participants) | 31 | 16
  Constipation C23D1 | -3.23 (27.70) | 0.00 (34.43)
  Constipation C24D1: number analyzed (Participants) | 29 | 12
  Constipation C24D1 | -3.45 (22.44) | 5.56 (31.25)
  Constipation C25D1: number analyzed (Participants) | 28 | 12
  Constipation C25D1 | -3.57 (24.58) | 0.00 (24.62)
  Constipation C26D1: number analyzed (Participants) | 26 | 9
  Constipation C26D1 | -5.13 (26.15) | 7.41 (14.70)
  Constipation C27D1: number analyzed (Participants) | 25 | 10
  Constipation C27D1 | -6.67 (25.46) | 10.00 (22.50)
  Constipation C28D1: number analyzed (Participants) | 21 | 11
  Constipation C28D1 | -4.76 (19.11) | 12.12 (22.47)
  Constipation C29D1: number analyzed (Participants) | 22 | 12
  Constipation C29D1 | 0.00 (20.57) | 5.56 (19.25)
  Constipation C30D1: number analyzed (Participants) | 20 | 0
  Constipation C30D1 | -3.33 (21.36) |
  Constipation C31D1: number analyzed (Participants) | 20 | 0
  Constipation C31D1 | 0.00 (18.73) |
  Constipation C32D1: number analyzed (Participants) | 18 | 0
  Constipation C32D1 | 1.85 (17.98) |
  Constipation C33D1: number analyzed (Participants) | 15 | 0
  Constipation C33D1 | -6.67 (18.69) |
  Constipation C34D1: number analyzed (Participants) | 12 | 0
  Constipation C34D1 | -8.33 (15.08) |
  Constipation C35D1: number analyzed (Participants) | 13 | 0
  Constipation C35D1 | -7.69 (14.62) |
  Constipation C36D1: number analyzed (Participants) | 12 | 0
  Constipation C36D1 | -8.33 (15.08) |
  Constipation C37D1: number analyzed (Participants) | 11 | 0
  Constipation C37D1 | -12.12 (16.82) |
  Constipation C38D1: number analyzed (Participants) | 10 | 0
  Constipation C38D1 | -6.67 (14.05) |
  Constipation C39D1: number analyzed (Participants) | 9 | 0
  Constipation C39D1 | -3.70 (11.11) |
  Constipation 30 day follow up: number analyzed (Participants) | 57 | 78
  Constipation 30 day follow up | -2.34 (30.12) | 4.70 (28.29)
  Constipation 90 day follow up: number analyzed (Participants) | 61 | 79
  Constipation 90 day follow up | 1.09 (27.19) | 5.91 (31.01)
  Diarrhoea Baseline | 8.09 (16.41) | 7.71 (15.34)
  Diarrhoea C2D1: number analyzed (Participants) | 208 | 217
  Diarrhoea C2D1 | 2.56 (20.56) | 5.68 (22.98)
  Diarrhoea C3D1: number analyzed (Participants) | 182 | 197
  Diarrhoea C3D1 | 2.93 (21.40) | 4.06 (20.63)
  Diarrhoea C4D1: number analyzed (Participants) | 169 | 169
  Diarrhoea C4D1 | 1.38 (21.00) | 3.94 (22.07)
  Diarrhoea C5D1: number analyzed (Participants) | 159 | 165
  Diarrhoea C5D1 | 1.47 (20.66) | 4.44 (20.34)
  Diarrhoea C6D1: number analyzed (Participants) | 149 | 146
  Diarrhoea C6D1 | 2.91 (24.79) | 3.65 (21.49)
  Diarrhoea C7D1: number analyzed (Participants) | 120 | 126
  Diarrhoea C7D1 | 1.94 (24.17) | 5.29 (19.51)
  Diarrhoea C8D1: number analyzed (Participants) | 108 | 110
  Diarrhoea C8D1 | 1.23 (21.82) | 2.12 (18.77)
  Diarrhoea C9D1: number analyzed (Participants) | 102 | 103
  Diarrhoea C9D1 | 1.31 (23.42) | 0.65 (19.79)
  Diarrhoea C10D1: number analyzed (Participants) | 85 | 79
  Diarrhoea C10D1 | 1.18 (19.55) | -2.53 (17.52)
  Diarrhoea C11D1: number analyzed (Participants) | 81 | 71
  Diarrhoea C11D1 | -3.29 (21.48) | -0.94 (18.66)
  Diarrhoea C12D1: number analyzed (Participants) | 75 | 57
  Diarrhoea C12D1 | -1.33 (17.71) | -2.92 (20.20)
  Diarrhoea C13D1: number analyzed (Participants) | 60 | 48
  Diarrhoea C13D1 | -3.89 (16.34) | -4.17 (17.70)
  Diarrhoea C14D1: number analyzed (Participants) | 55 | 44
  Diarrhoea C14D1 | -3.03 (17.30) | -2.27 (20.83)
  Diarrhoea C15D1: number analyzed (Participants) | 51 | 36
  Diarrhoea C15D1 | -1.31 (19.96) | -2.78 (20.12)
  Diarrhoea C16D1: number analyzed (Participants) | 48 | 31
  Diarrhoea C16D1 | -1.39 (16.78) | -3.23 (13.21)
  Diarrhoea C17D1: number analyzed (Participants) | 43 | 25
  Diarrhoea C17D1 | -0.78 (19.91) | -4.00 (11.06)
  Diarrhoea C18D1: number analyzed (Participants) | 41 | 21
  Diarrhoea C18D1 | -1.63 (16.59) | -4.76 (19.11)
  Diarrhoea C19D1: number analyzed (Participants) | 40 | 20
  Diarrhoea C19D1 | -2.50 (15.81) | -3.33 (14.91)
  Diarrhoea C20D1: number analyzed (Participants) | 39 | 19
  Diarrhoea C20D1 | -1.71 (17.01) | -3.51 (15.29)
  Diarrhoea C21D1: number analyzed (Participants) | 36 | 20
  Diarrhoea C21D1 | -0.93 (18.66) | -3.33 (14.91)
  Diarrhoea C22D1: number analyzed (Participants) | 31 | 17
  Diarrhoea C22D1 | 0.00 (14.91) | -5.88 (21.20)
  Diarrhoea C23D1: number analyzed (Participants) | 31 | 16
  Diarrhoea C23D1 | 1.08 (16.06) | -8.33 (14.91)
  Diarrhoea C24D1: number analyzed (Participants) | 29 | 12
  Diarrhoea C24D1 | 2.30 (12.38) | -2.78 (9.62)
  Diarrhoea C25D1: number analyzed (Participants) | 28 | 12
  Diarrhoea C25D1 | 0.00 (15.71) | -2.78 (17.16)
  Diarrhoea C26D1: number analyzed (Participants) | 26 | 9
  Diarrhoea C26D1 | 0.00 (13.33) | 0.00 (16.67)
  Diarrhoea C27D1: number analyzed (Participants) | 25 | 10
  Diarrhoea C27D1 | 1.33 (15.15) | -3.33 (18.92)
  Diarrhoea C28D1: number analyzed (Participants) | 21 | 11
  Diarrhoea C28D1 | 0.00 (14.91) | -6.06 (20.10)
  Diarrhoea C29D1: number analyzed (Participants) | 22 | 12
  Diarrhoea C29D1 | 3.03 (17.55) | -8.33 (25.13)
  Diarrhoea C30D1: number analyzed (Participants) | 20 | 0
  Diarrhoea C30D1 | 1.67 (17.01) |
  Diarrhoea C31D1: number analyzed (Participants) | 20 | 0
  Diarrhoea C31D1 | -1.67 (13.13) |
  Diarrhoea C32D1: number analyzed (Participants) | 18 | 0
  Diarrhoea C32D1 | 5.56 (17.15) |
  Diarrhoea C33D1: number analyzed (Participants) | 15 | 0
  Diarrhoea C33D1 | 0.00 (17.82) |
  Diarrhoea C34D1: number analyzed (Participants) | 12 | 0
  Diarrhoea C34D1 | -5.56 (19.25) |
  Diarrhoea C35D1: number analyzed (Participants) | 13 | 0
  Diarrhoea C35D1 | 2.56 (16.45) |
  Diarrhoea C36D1: number analyzed (Participants) | 12 | 0
  Diarrhoea C36D1 | 0.00 (14.21) |
  Diarrhoea C37D1: number analyzed (Participants) | 11 | 0
  Diarrhoea C37D1 | 0.00 (21.08) |
  Diarrhoea C38D1: number analyzed (Participants) | 10 | 0
  Diarrhoea C38D1 | 6.67 (21.08) |
  Diarrhoea C39D1: number analyzed (Participants) | 9 | 0
  Diarrhoea C39D1 | 3.70 (20.03) |
  Diarrhoea 30 day follow up: number analyzed (Participants) | 57 | 78
  Diarrhoea 30 day follow up | -0.58 (18.36) | 1.71 (19.29)
  Diarrhoea 90 day follow up: number analyzed (Participants) | 61 | 79
  Diarrhoea 90 day follow up | 2.73 (20.45) | -1.27 (23.54)
  Financial Difficulties Baseline | 20.71 (25.99) | 19.42 (25.30)
  Financial Difficulties C2D1: number analyzed (Participants) | 208 | 217
  Financial Difficulties C2D1 | -0.64 (25.58) | -0.92 (18.68)
  Financial Difficulties C3D1: number analyzed (Participants) | 182 | 197
  Financial Difficulties C3D1 | -0.92 (25.13) | 1.18 (22.43)
  Financial Difficulties C4D1: number analyzed (Participants) | 169 | 169
  Financial Difficulties C4D1 | -2.17 (23.33) | -1.58 (22.07)
  Financial Difficulties C5D1: number analyzed (Participants) | 159 | 165
  Financial Difficulties C5D1 | -0.63 (28.92) | 0.81 (19.81)
  Financial Difficulties C6D1: number analyzed (Participants) | 149 | 146
  Financial Difficulties C6D1 | -0.89 (27.66) | 0.00 (21.80)
  Financial Difficulties C7D1: number analyzed (Participants) | 120 | 126
  Financial Difficulties C7D1 | 0.56 (24.05) | 0.26 (24.76)
  Financial Difficulties C8D1: number analyzed (Participants) | 108 | 110
  Financial Difficulties C8D1 | -0.62 (26.95) | 3.33 (23.87)
  Financial Difficulties C9D1: number analyzed (Participants) | 102 | 103
  Financial Difficulties C9D1 | 2.29 (24.94) | 1.94 (21.30)
  Financial Difficulties C10D1: number analyzed (Participants) | 85 | 79
  Financial Difficulties C10D1 | -2.75 (27.80) | 1.27 (24.13)
  Financial Difficulties C11D1: number analyzed (Participants) | 81 | 71
  Financial Difficulties C11D1 | 0.00 (27.39) | 4.69 (22.04)
  Financial Difficulties C12D1: number analyzed (Participants) | 75 | 57
  Financial Difficulties C12D1 | -0.89 (30.00) | 3.51 (22.44)
  Financial Difficulties C13D1: number analyzed (Participants) | 60 | 48
  Financial Difficulties C13D1 | -3.33 (27.92) | 4.17 (25.38)
  Financial Difficulties C14D1: number analyzed (Participants) | 55 | 44
  Financial Difficulties C14D1 | -0.61 (29.04) | 0.00 (23.84)
  Financial Difficulties C15D1: number analyzed (Participants) | 51 | 36
  Financial Difficulties C15D1 | 0.00 (29.06) | 4.63 (24.11)
  Financial Difficulties C16D1: number analyzed (Participants) | 48 | 31
  Financial Difficulties C16D1 | -2.08 (25.18) | 6.45 (26.41)
  Financial Difficulties C17D1: number analyzed (Participants) | 43 | 25
  Financial Difficulties C17D1 | -2.33 (23.45) | 1.33 (20.37)
  Financial Difficulties C18D1: number analyzed (Participants) | 41 | 21
  Financial Difficulties C18D1 | 3.25 (22.12) | 4.76 (24.23)
  Financial Difficulties C19D1: number analyzed (Participants) | 40 | 20
  Financial Difficulties C19D1 | -2.50 (21.86) | -3.33 (18.42)
  Financial Difficulties C20D1: number analyzed (Participants) | 39 | 19
  Financial Difficulties C20D1 | 0.00 (24.18) | -1.75 (20.71)
  Financial Difficulties C21D1: number analyzed (Participants) | 36 | 20
  Financial Difficulties C21D1 | 1.85 (25.13) | 3.33 (21.36)
  Financial Difficulties C22D1: number analyzed (Participants) | 31 | 17
  Financial Difficulties C22D1 | -3.23 (21.70) | 3.92 (26.04)
  Financial Difficulties C23D1: number analyzed (Participants) | 31 | 16
  Financial Difficulties C23D1 | 3.23 (23.34) | 4.17 (23.96)
  Financial Difficulties C24D1: number analyzed (Participants) | 29 | 12
  Financial Difficulties C24D1 | 1.15 (22.68) | 2.78 (26.43)
  Financial Difficulties C25D1: number analyzed (Participants) | 28 | 12
  Financial Difficulties C25D1 | 0.00 (22.22) | 8.33 (20.72)
  Financial Difficulties C26D1: number analyzed (Participants) | 26 | 9
  Financial Difficulties C26D1 | -2.56 (20.92) | -7.41 (14.70)
  Financial Difficulties C27D1: number analyzed (Participants) | 25 | 10
  Financial Difficulties C27D1 | 1.33 (17.95) | -6.67 (14.05)
  Financial Difficulties C28D1: number analyzed (Participants) | 21 | 11
  Financial Difficulties C28D1 | -4.76 (21.82) | -3.03 (17.98)
  Financial Difficulties C29D1: number analyzed (Participants) | 22 | 12
  Financial Difficulties C29D1 | 3.03 (17.55) | 0.00 (14.21)
  Financial Difficulties C30D1: number analyzed (Participants) | 20 | 0
  Financial Difficulties C30D1 | 0.00 (24.18) |
  Financial Difficulties C31D1: number analyzed (Participants) | 20 | 0
  Financial Difficulties C31D1 | 0.00 (21.63) |
  Financial Difficulties C32D1: number analyzed (Participants) | 18 | 0
  Financial Difficulties C32D1 | -5.56 (17.15) |
  Financial Difficulties C33D1: number analyzed (Participants) | 15 | 0
  Financial Difficulties C33D1 | -6.67 (13.80) |
  Financial Difficulties C34D1: number analyzed (Participants) | 12 | 0
  Financial Difficulties C34D1 | -5.56 (12.97) |
  Financial Difficulties C35D1: number analyzed (Participants) | 13 | 0
  Financial Difficulties C35D1 | -2.56 (16.45) |
  Financial Difficulties C36D1: number analyzed (Participants) | 12 | 0
  Financial Difficulties C36D1 | -2.78 (17.16) |
  Financial Difficulties C37D1: number analyzed (Participants) | 11 | 0
  Financial Difficulties C37D1 | -6.06 (13.48) |
  Financial Difficulties C38D1: number analyzed (Participants) | 10 | 0
  Financial Difficulties C38D1 | -6.67 (14.05) |
  Financial Difficulties C39D1: number analyzed (Participants) | 9 | 0
  Financial Difficulties C39D1 | -3.70 (20.03) |
  Financial Difficulties 30 day follow up: number analyzed (Participants) | 57 | 78
  Financial Difficulties 30 day follow up | 4.09 (26.03) | 9.40 (24.56)
  Financial Difficulties 90 day follow up: number analyzed (Participants) | 61 | 79
  Financial Difficulties 90 day follow up | 3.28 (24.87) | 3.80 (20.66)

11. Secondary Outcome: Change From Baseline in HRQoL Measured by the QLQ-OG25 Questionnaire Plus STO22 Belching Subscale Questionnaire
Description: OG25 evaluated gastric & gastroesophageal junction cancer-specific symptoms,had 25 items with 6 scales:dysphagia,eating restrictions,reflux,odynophagia,pain & discomfort,anxiety,and 10 single items:trouble with(taste, swallowing saliva, coughing, talking),eating in front of others,dry mouth,body image,choked when swallowing,weight loss and hair loss. STO22: gastric cancer quality of life questionnaire with 22 questions.For OG25 and STO22,items scored on(1:not at all; 2:a little, 3:quite a bit, 4:very much) and 1 question was "yes or no" for STO22.Linear transformation was used; score ranged from 0 to 100;higher score=better level of functioning or greater degree of symptoms. An item from STO22 instrument related to belching was used with OG25.
Time Frame: Baseline, on D1 from C2 through C39, 30-day follow up, 90-day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 243 | 242
Unit on a scale
  Dysphagia Baseline | 12.12 (18.27) | 12.59 (19.27)
  Dysphagia C2D1: number analyzed (Participants) | 208 | 216
  Dysphagia C2D1 | -0.37 (17.07) | -3.86 (15.69)
  Dysphagia C3D1: number analyzed (Participants) | 182 | 196
  Dysphagia C3D1 | -0.92 (15.22) | -4.59 (16.22)
  Dysphagia C4D1: number analyzed (Participants) | 166 | 169
  Dysphagia C4D1 | -2.68 (17.13) | -5.00 (17.23)
  Dysphagia C5D1: number analyzed (Participants) | 159 | 165
  Dysphagia C5D1 | -1.05 (20.30) | -5.66 (17.07)
  Dysphagia C6D1: number analyzed (Participants) | 149 | 145
  Dysphagia C6D1 | -1.42 (16.81) | -3.45 (19.00)
  Dysphagia C7D1: number analyzed (Participants) | 119 | 125
  Dysphagia C7D1 | -2.61 (16.28) | -5.16 (17.02)
  Dysphagia C8D1: number analyzed (Participants) | 108 | 109
  Dysphagia C8D1 | -2.88 (18.81) | -4.28 (17.88)
  Dysphagia C9D1: number analyzed (Participants) | 102 | 103
  Dysphagia C9D1 | -2.83 (17.67) | -5.93 (17.17)
  Dysphagia C10D1: number analyzed (Participants) | 85 | 79
  Dysphagia C10D1 | -3.27 (16.61) | -6.75 (18.70)
  Dysphagia C11D1: number analyzed (Participants) | 80 | 71
  Dysphagia C11D1 | -3.33 (16.90) | -5.95 (19.41)
  Dysphagia C12D1: number analyzed (Participants) | 75 | 57
  Dysphagia C12D1 | -3.70 (17.07) | -5.65 (16.15)
  Dysphagia C13D1: number analyzed (Participants) | 60 | 48
  Dysphagia C13D1 | -6.30 (17.64) | -4.40 (14.81)
  Dysphagia C14D1: number analyzed (Participants) | 55 | 44
  Dysphagia C14D1 | -4.24 (15.49) | -3.03 (14.25)
  Dysphagia C15D1: number analyzed (Participants) | 51 | 36
  Dysphagia C15D1 | -3.49 (14.82) | -1.54 (17.24)
  Dysphagia C16D1: number analyzed (Participants) | 48 | 31
  Dysphagia C16D1 | -2.31 (14.85) | 0.00 (12.83)
  Dysphagia C17D1: number analyzed (Participants) | 43 | 25
  Dysphagia C17D1 | -3.10 (13.13) | -1.78 (11.86)
  Dysphagia C18D1: number analyzed (Participants) | 41 | 21
  Dysphagia C18D1 | -3.25 (14.96) | -4.23 (10.82)
  Dysphagia C19D1: number analyzed (Participants) | 40 | 20
  Dysphagia C19D1 | -4.17 (13.48) | -2.78 (7.10)
  Dysphagia C20D1: number analyzed (Participants) | 39 | 19
  Dysphagia C20D1 | -4.56 (11.60) | -2.92 (11.01)
  Dysphagia C21D1: number analyzed (Participants) | 36 | 20
  Dysphagia C21D1 | -3.40 (15.22) | -3.33 (13.05)
  Dysphagia C22D1: number analyzed (Participants) | 31 | 17
  Dysphagia C22D1 | -5.38 (15.94) | -5.23 (9.72)
  Dysphagia C23D1: number analyzed (Participants) | 31 | 16
  Dysphagia C23D1 | -4.30 (14.54) | -5.56 (10.73)
  Dysphagia C24D1: number analyzed (Participants) | 29 | 12
  Dysphagia C24D1 | -4.98 (13.80) | -2.78 (11.73)
  Dysphagia C25D1: number analyzed (Participants) | 28 | 12
  Dysphagia C25D1 | -4.37 (12.95) | -3.70 (10.94)
  Dysphagia C26D1: number analyzed (Participants) | 26 | 9
  Dysphagia C26D1 | -2.99 (18.21) | 2.47 (9.26)
  Dysphagia C27D1: number analyzed (Participants) | 25 | 10
  Dysphagia C27D1 | -5.33 (12.88) | 0.00 (5.24)
  Dysphagia C28D1: number analyzed (Participants) | 21 | 11
  Dysphagia C28D1 | -4.76 (14.30) | 1.01 (5.99)
  Dysphagia C29D1: number analyzed (Participants) | 22 | 12
  Dysphagia C29D1 | -7.07 (13.95) | 1.85 (13.26)
  Dysphagia C30D1: number analyzed (Participants) | 20 | 0
  Dysphagia C30D1 | -5.00 (15.07) |
  Dysphagia C31D1: number analyzed (Participants) | 20 | 0
  Dysphagia C31D1 | -6.11 (13.72) |
  Dysphagia C32D1: number analyzed (Participants) | 18 | 0
  Dysphagia C32D1 | -7.41 (14.76) |
  Dysphagia C33D1: number analyzed (Participants) | 15 | 0
  Dysphagia C33D1 | -3.70 (16.08) |
  Dysphagia C34D1: number analyzed (Participants) | 12 | 0
  Dysphagia C34D1 | -8.33 (19.03) |
  Dysphagia C35D1: number analyzed (Participants) | 13 | 0
  Dysphagia C35D1 | -6.84 (19.53) |
  Dysphagia C36D1: number analyzed (Participants) | 12 | 0
  Dysphagia C36D1 | -9.26 (19.44) |
  Dysphagia C37D1: number analyzed (Participants) | 11 | 0
  Dysphagia C37D1 | -8.08 (14.13) |
  Dysphagia C38D1: number analyzed (Participants) | 10 | 0
  Dysphagia C38D1 | -6.67 (16.73) |
  Dysphagia C39D1: number analyzed (Participants) | 9 | 0
  Dysphagia C39D1 | -4.94 (12.56) |
  Dysphagia 30 day follow up: number analyzed (Participants) | 57 | 76
  Dysphagia 30 day follow up | 4.48 (22.60) | 0.73 (24.63)
  Dysphagia 90 day follow up: number analyzed (Participants) | 61 | 79
  Dysphagia 90 day follow up | 0.36 (12.33) | -1.83 (19.28)
  Eating Restrictions Baseline | 22.67 (25.20) | 22.51 (24.22)
  Eating Restrictions C2D1: number analyzed (Participants) | 208 | 216
  Eating Restrictions C2D1 | -1.24 (21.39) | -4.55 (20.82)
  Eating Restrictions C3D1: number analyzed (Participants) | 182 | 196
  Eating Restrictions C3D1 | -4.12 (20.26) | -6.08 (20.52)
  Eating Restrictions C4D1: number analyzed (Participants) | 166 | 169
  Eating Restrictions C4D1 | -5.52 (21.76) | -8.19 (21.18)
  Eating Restrictions C5D1: number analyzed (Participants) | 159 | 165
  Eating Restrictions C5D1 | -5.14 (23.77) | -7.22 (22.12)
  Eating Restrictions C6D1: number analyzed (Participants) | 149 | 145
  Eating Restrictions C6D1 | -3.97 (21.24) | -6.03 (23.04)
  Eating Restrictions C7D1: number analyzed (Participants) | 119 | 125
  Eating Restrictions C7D1 | -4.69 (21.03) | -5.07 (22.32)
  Eating Restrictions C8D1: number analyzed (Participants) | 108 | 109
  Eating Restrictions C8D1 | -3.70 (21.87) | -6.27 (24.35)
  Eating Restrictions C9D1: number analyzed (Participants) | 102 | 103
  Eating Restrictions C9D1 | -3.59 (22.75) | -7.52 (22.25)
  Eating Restrictions C10D1: number analyzed (Participants) | 85 | 79
  Eating Restrictions C10D1 | -4.80 (24.03) | -8.54 (26.75)
  Eating Restrictions C11D1: number analyzed (Participants) | 80 | 71
  Eating Restrictions C11D1 | -5.83 (25.96) | -9.39 (27.17)
  Eating Restrictions C12D1: number analyzed (Participants) | 75 | 57
  Eating Restrictions C12D1 | -6.22 (27.47) | -9.36 (22.33)
  Eating Restrictions C13D1: number analyzed (Participants) | 60 | 48
  Eating Restrictions C13D1 | -9.31 (28.04) | -10.59 (21.59)
  Eating Restrictions C14D1: number analyzed (Participants) | 55 | 44
  Eating Restrictions C14D1 | -6.97 (25.45) | -7.39 (22.17)
  Eating Restrictions C15D1: number analyzed (Participants) | 51 | 36
  Eating Restrictions C15D1 | -7.03 (24.46) | -6.25 (21.02)
  Eating Restrictions C16D1: number analyzed (Participants) | 48 | 31
  Eating Restrictions C16D1 | -8.68 (22.41) | -6.72 (20.23)
  Eating Restrictions C17D1: number analyzed (Participants) | 43 | 25
  Eating Restrictions C17D1 | -7.75 (22.67) | -3.33 (21.52)
  Eating Restrictions C18D1: number analyzed (Participants) | 41 | 21
  Eating Restrictions C18D1 | -7.11 (23.68) | -10.32 (21.23)
  Eating Restrictions C19D1: number analyzed (Participants) | 40 | 20
  Eating Restrictions C19D1 | -7.92 (20.06) | -9.17 (14.02)
  Eating Restrictions C20D1: number analyzed (Participants) | 39 | 19
  Eating Restrictions C20D1 | -6.41 (22.98) | -9.21 (20.95)
  Eating Restrictions C21D1: number analyzed (Participants) | 36 | 20
  Eating Restrictions C21D1 | -5.32 (20.52) | -10.00 (19.61)
  Eating Restrictions C22D1: number analyzed (Participants) | 31 | 17
  Eating Restrictions C22D1 | -7.26 (23.93) | -12.25 (22.46)
  Eating Restrictions C23D1: number analyzed (Participants) | 31 | 16
  Eating Restrictions C23D1 | -6.18 (20.07) | -12.50 (19.95)
  Eating Restrictions C24D1: number analyzed (Participants) | 29 | 12
  Eating Restrictions C24D1 | -6.03 (21.12) | -6.25 (20.45)
  Eating Restrictions C25D1: number analyzed (Participants) | 28 | 12
  Eating Restrictions C25D1 | -5.95 (23.34) | -8.33 (18.46)
  Eating Restrictions C26D1: number analyzed (Participants) | 26 | 9
  Eating Restrictions C26D1 | -7.37 (25.31) | -2.78 (17.68)
  Eating Restrictions C27D1: number analyzed (Participants) | 25 | 10
  Eating Restrictions C27D1 | -7.67 (22.30) | -3.33 (13.72)
  Eating Restrictions C28D1: number analyzed (Participants) | 21 | 11
  Eating Restrictions C28D1 | -6.35 (24.71) | 2.27 (7.54)
  Eating Restrictions C29D1: number analyzed (Participants) | 22 | 12
  Eating Restrictions C29D1 | -10.23 (19.57) | -3.47 (19.29)
  Eating Restrictions C30D1: number analyzed (Participants) | 20 | 0
  Eating Restrictions C30D1 | -5.42 (22.01) |
  Eating Restrictions C31D1: number analyzed (Participants) | 20 | 0
  Eating Restrictions C31D1 | -10.42 (20.75) |
  Eating Restrictions C32D1: number analyzed (Participants) | 18 | 0
  Eating Restrictions C32D1 | -9.26 (23.90) |
  Eating Restrictions C33D1: number analyzed (Participants) | 15 | 0
  Eating Restrictions C33D1 | -7.78 (13.90) |
  Eating Restrictions C34D1: number analyzed (Participants) | 12 | 0
  Eating Restrictions C34D1 | -17.36 (25.74) |
  Eating Restrictions C35D1: number analyzed (Participants) | 13 | 0
  Eating Restrictions C35D1 | -11.54 (26.25) |
  Eating Restrictions C36D1: number analyzed (Participants) | 12 | 0
  Eating Restrictions C36D1 | -15.97 (25.24) |
  Eating Restrictions C37D1: number analyzed (Participants) | 11 | 0
  Eating Restrictions C37D1 | -12.12 (15.08) |
  Eating Restrictions C38D1: number analyzed (Participants) | 10 | 0
  Eating Restrictions C38D1 | -17.50 (21.68) |
  Eating Restrictions C39D1: number analyzed (Participants) | 9 | 0
  Eating Restrictions C39D1 | -7.41 (13.47) |
  Eating Restrictions 30 day follow up: number analyzed (Participants) | 57 | 76
  Eating Restrictions 30 day follow up | 0.15 (27.57) | 0.88 (23.47)
  Eating Restrictions 90 day follow up: number analyzed (Participants) | 61 | 79
  Eating Restrictions 90 day follow up | -2.19 (22.77) | -0.42 (23.19)
  Reflux Baseline | 13.17 (20.28) | 16.11 (22.25)
  Reflux C2D1: number analyzed (Participants) | 208 | 216
  Reflux C2D1 | -1.04 (20.79) | -4.01 (18.66)
  Reflux C3D1: number analyzed (Participants) | 182 | 196
  Reflux C3D1 | -0.09 (21.71) | -4.17 (18.36)
  Reflux C4D1: number analyzed (Participants) | 166 | 169
  Reflux C4D1 | -0.70 (22.80) | -5.82 (21.53)
  Reflux C5D1: number analyzed (Participants) | 159 | 165
  Reflux C5D1 | -0.84 (22.17) | -7.88 (19.87)
  Reflux C6D1: number analyzed (Participants) | 149 | 145
  Reflux C6D1 | -0.11 (22.39) | -7.01 (20.57)
  Reflux C7D1: number analyzed (Participants) | 119 | 125
  Reflux C7D1 | -1.68 (20.40) | -6.67 (21.48)
  Reflux C8D1: number analyzed (Participants) | 108 | 109
  Reflux C8D1 | -1.08 (23.04) | -9.17 (21.81)
  Reflux C9D1: number analyzed (Participants) | 102 | 103
  Reflux C9D1 | -0.82 (27.49) | -11.00 (20.82)
  Reflux C10D1: number analyzed (Participants) | 85 | 79
  Reflux C10D1 | -1.57 (23.80) | -10.34 (22.69)
  Reflux C11D1: number analyzed (Participants) | 80 | 71
  Reflux C11D1 | -3.13 (21.23) | -11.03 (24.23)
  Reflux C12D1: number analyzed (Participants) | 75 | 57
  Reflux C12D1 | -4.44 (22.48) | -8.48 (23.60)
  Reflux C13D1: number analyzed (Participants) | 60 | 48
  Reflux C13D1 | -3.33 (28.26) | -9.03 (24.78)
  Reflux C14D1: number analyzed (Participants) | 55 | 44
  Reflux C14D1 | -1.82 (22.38) | -8.71 (20.80)
  Reflux C15D1: number analyzed (Participants) | 51 | 36
  Reflux C15D1 | -3.92 (18.13) | -7.41 (24.70)
  Reflux C16D1: number analyzed (Participants) | 48 | 31
  Reflux C16D1 | -3.13 (23.23) | -4.84 (20.27)
  Reflux C17D1: number analyzed (Participants) | 43 | 25
  Reflux C17D1 | -5.81 (22.09) | -2.67 (21.34)
  Reflux C18D1: number analyzed (Participants) | 41 | 21
  Reflux C18D1 | -3.25 (23.04) | -3.17 (23.93)
  Reflux C19D1: number analyzed (Participants) | 40 | 20
  Reflux C19D1 | -2.92 (22.61) | -1.67 (13.13)
  Reflux C20D1: number analyzed (Participants) | 39 | 19
  Reflux C20D1 | 0.00 (20.94) | -4.39 (24.75)
  Reflux C21D1: number analyzed (Participants) | 36 | 20
  Reflux C21D1 | 0.46 (24.07) | -2.50 (27.72)
  Reflux C22D1: number analyzed (Participants) | 31 | 17
  Reflux C22D1 | -5.38 (17.94) | -1.96 (26.93)
  Reflux C23D1: number analyzed (Participants) | 31 | 16
  Reflux C23D1 | -4.30 (18.74) | -4.17 (24.72)
  Reflux C24D1: number analyzed (Participants) | 29 | 12
  Reflux C24D1 | -2.30 (19.78) | -6.94 (26.07)
  Reflux C25D1: number analyzed (Participants) | 28 | 12
  Reflux C25D1 | -1.19 (19.74) | -4.17 (25.75)
  Reflux C26D1: number analyzed (Participants) | 26 | 9
  Reflux C26D1 | -1.28 (16.95) | 3.70 (18.22)
  Reflux C27D1: number analyzed (Participants) | 25 | 10
  Reflux C27D1 | -1.33 (17.29) | 1.67 (12.30)
  Reflux C28D1: number analyzed (Participants) | 21 | 11
  Reflux C28D1 | 0.00 (17.48) | 3.03 (16.36)
  Reflux C29D1: number analyzed (Participants) | 22 | 12
  Reflux C29D1 | -3.03 (14.21) | -1.39 (8.58)
  Reflux C30D1: number analyzed (Participants) | 20 | 0
  Reflux C30D1 | -0.83 (13.76) |
  Reflux C31D1: number analyzed (Participants) | 20 | 0
  Reflux C31D1 | -1.67 (16.13) |
  Reflux C32D1: number analyzed (Participants) | 18 | 0
  Reflux C32D1 | 0.00 (18.96) |
  Reflux C33D1: number analyzed (Participants) | 15 | 0
  Reflux C33D1 | -3.33 (14.36) |
  Reflux C34D1: number analyzed (Participants) | 12 | 0
  Reflux C34D1 | -4.17 (18.97) |
  Reflux C35D1: number analyzed (Participants) | 13 | 0
  Reflux C35D1 | 1.28 (19.79) |
  Reflux C36D1: number analyzed (Participants) | 12 | 0
  Reflux C36D1 | -4.17 (21.47) |
  Reflux C37D1: number analyzed (Participants) | 11 | 0
  Reflux C37D1 | -4.55 (18.40) |
  Reflux C38D1: number analyzed (Participants) | 10 | 0
  Reflux C38D1 | 0.00 (20.79) |
  Reflux C39D1: number analyzed (Participants) | 9 | 0
  Reflux C39D1 | 7.41 (12.11) |
  Reflux 30 day follow up: number analyzed (Participants) | 57 | 76
  Reflux 30 day follow up | 1.46 (26.03) | 0.44 (26.10)
  Reflux 90 day follow up: number analyzed (Participants) | 61 | 79
  Reflux 90 day follow up | 2.19 (19.83) | -1.69 (21.28)
  Odynophagia Baseline | 15.64 (22.78) | 17.29 (24.69)
  Odynophagia C2D1: number analyzed (Participants) | 208 | 216
  Odynophagia C2D1 | -2.80 (21.46) | -4.63 (22.20)
  Odynophagia C3D1: number analyzed (Participants) | 182 | 196
  Odynophagia C3D1 | -3.94 (19.38) | -6.04 (20.37)
  Odynophagia C4D1: number analyzed (Participants) | 166 | 169
  Odynophagia C4D1 | -5.22 (21.93) | -8.19 (21.14)
  Odynophagia C5D1: number analyzed (Participants) | 159 | 165
  Odynophagia C5D1 | -4.19 (22.58) | -7.58 (23.75)
  Odynophagia C6D1: number analyzed (Participants) | 149 | 145
  Odynophagia C6D1 | -2.80 (20.54) | -5.98 (22.96)
  Odynophagia C7D1: number analyzed (Participants) | 119 | 125
  Odynophagia C7D1 | -3.92 (19.73) | -5.33 (24.19)
  Odynophagia C8D1: number analyzed (Participants) | 108 | 109
  Odynophagia C8D1 | -4.32 (21.54) | -7.19 (23.83)
  Odynophagia C9D1: number analyzed (Participants) | 102 | 103
  Odynophagia C9D1 | -2.94 (22.30) | -7.93 (24.35)
  Odynophagia C10D1: number analyzed (Participants) | 85 | 79
  Odynophagia C10D1 | -5.10 (24.26) | -8.02 (28.35)
  Odynophagia C11D1: number analyzed (Participants) | 80 | 71
  Odynophagia C11D1 | -4.17 (25.78) | -9.62 (27.26)
  Odynophagia C12D1: number analyzed (Participants) | 75 | 57
  Odynophagia C12D1 | -6.67 (25.70) | -7.60 (22.29)
  Odynophagia C13D1: number analyzed (Participants) | 60 | 48
  Odynophagia C13D1 | -8.06 (26.66) | -7.99 (25.50)
  Odynophagia C14D1: number analyzed (Participants) | 55 | 44
  Odynophagia C14D1 | -7.58 (24.18) | -5.68 (24.10)
  Odynophagia C15D1: number analyzed (Participants) | 51 | 36
  Odynophagia C15D1 | -7.84 (23.18) | -3.24 (27.55)
  Odynophagia C16D1: number analyzed (Participants) | 48 | 31
  Odynophagia C16D1 | -9.37 (21.99) | 0.00 (23.17)
  Odynophagia C17D1: number analyzed (Participants) | 43 | 25
  Odynophagia C17D1 | -11.63 (21.37) | -2.67 (24.38)
  Odynophagia C18D1: number analyzed (Participants) | 41 | 21
  Odynophagia C18D1 | -9.76 (22.66) | -5.56 (23.77)
  Odynophagia C19D1: number analyzed (Participants) | 40 | 20
  Odynophagia C19D1 | -9.58 (18.45) | -2.50 (13.55)
  Odynophagia C20D1: number analyzed (Participants) | 39 | 19
  Odynophagia C20D1 | -7.26 (21.56) | -7.02 (25.65)
  Odynophagia C21D1: number analyzed (Participants) | 36 | 20
  Odynophagia C21D1 | -5.09 (18.61) | -7.50 (22.60)
  Odynophagia C22D1: number analyzed (Participants) | 31 | 17
  Odynophagia C22D1 | -5.91 (19.51) | -5.88 (27.60)
  Odynophagia C23D1: number analyzed (Participants) | 31 | 16
  Odynophagia C23D1 | -7.53 (21.01) | -7.29 (29.17)
  Odynophagia C24D1: number analyzed (Participants) | 29 | 12
  Odynophagia C24D1 | -6.90 (21.14) | -11.11 (29.59)
  Odynophagia C25D1: number analyzed (Participants) | 28 | 12
  Odynophagia C25D1 | -7.14 (18.39) | -9.72 (30.53)
  Odynophagia C26D1: number analyzed (Participants) | 26 | 9
  Odynophagia C26D1 | -7.69 (23.68) | -1.85 (13.03)
  Odynophagia C27D1: number analyzed (Participants) | 25 | 10
  Odynophagia C27D1 | -7.33 (18.05) | -1.67 (14.59)
  Odynophagia C28D1: number analyzed (Participants) | 21 | 11
  Odynophagia C28D1 | -9.52 (17.93) | -1.52 (11.68)
  Odynophagia C29D1: number analyzed (Participants) | 22 | 12
  Odynophagia C29D1 | -10.61 (18.22) | -1.39 (8.58)
  Odynophagia C30D1: number analyzed (Participants) | 20 | 0
  Odynophagia C30D1 | -9.17 (21.95) |
  Odynophagia C31D1: number analyzed (Participants) | 20 | 0
  Odynophagia C31D1 | -12.50 (19.40) |
  Odynophagia C32D1: number analyzed (Participants) | 18 | 0
  Odynophagia C32D1 | -11.11 (19.80) |
  Odynophagia C33D1: number analyzed (Participants) | 15 | 0
  Odynophagia C33D1 | -10.00 (15.17) |
  Odynophagia C34D1: number analyzed (Participants) | 12 | 0
  Odynophagia C34D1 | -16.67 (20.10) |
  Odynophagia C35D1: number analyzed (Participants) | 13 | 0
  Odynophagia C35D1 | -17.95 (20.93) |
  Odynophagia C36D1: number analyzed (Participants) | 12 | 0
  Odynophagia C36D1 | -18.06 (24.06) |
  Odynophagia C37D1: number analyzed (Participants) | 11 | 0
  Odynophagia C37D1 | -10.61 (15.41) |
  Odynophagia C38D1: number analyzed (Participants) | 10 | 0
  Odynophagia C38D1 | -11.67 (15.81) |
  Odynophagia C39D1: number analyzed (Participants) | 9 | 0
  Odynophagia C39D1 | -16.67 (14.43) |
  Odynophagia 30 day follow up: number analyzed (Participants) | 57 | 76
  Odynophagia 30 day follow up | 1.75 (29.66) | 2.19 (27.53)
  Odynophagia 90 day follow up: number analyzed (Participants) | 61 | 79
  Odynophagia 90 day follow up | -0.27 (18.63) | -0.21 (23.19)
  Pain and Discomfort Baseline | 23.53 (23.88) | 25.38 (25.42)
  Pain and Discomfort C2D1: number analyzed (Participants) | 208 | 216
  Pain and Discomfort C2D1 | -4.25 (23.38) | -6.94 (24.18)
  Pain and Discomfort C3D1: number analyzed (Participants) | 182 | 196
  Pain and Discomfort C3D1 | -6.59 (22.14) | -8.25 (21.97)
  Pain and Discomfort C4D1: number analyzed (Participants) | 166 | 169
  Pain and Discomfort C4D1 | -7.33 (24.99) | -11.34 (24.08)
  Pain and Discomfort C5D1: number analyzed (Participants) | 159 | 165
  Pain and Discomfort C5D1 | -7.44 (20.43) | -11.41 (26.21)
  Pain and Discomfort C6D1: number analyzed (Participants) | 149 | 145
  Pain and Discomfort C6D1 | -5.82 (25.48) | -9.31 (27.28)
  Pain and Discomfort C7D1: number analyzed (Participants) | 119 | 125
  Pain and Discomfort C7D1 | -8.54 (23.95) | -9.20 (24.54)
  Pain and Discomfort C8D1: number analyzed (Participants) | 108 | 109
  Pain and Discomfort C8D1 | -7.10 (23.04) | -9.94 (25.87)
  Pain and Discomfort C9D1: number analyzed (Participants) | 102 | 103
  Pain and Discomfort C9D1 | -5.07 (24.57) | -8.09 (26.08)
  Pain and Discomfort C10D1: number analyzed (Participants) | 85 | 79
  Pain and Discomfort C10D1 | -8.24 (26.80) | -8.23 (28.48)
  Pain and Discomfort C11D1: number analyzed (Participants) | 80 | 71
  Pain and Discomfort C11D1 | -7.71 (30.00) | -8.22 (28.99)
  Pain and Discomfort C12D1: number analyzed (Participants) | 75 | 57
  Pain and Discomfort C12D1 | -6.44 (27.52) | -5.85 (25.49)
  Pain and Discomfort C13D1: number analyzed (Participants) | 60 | 48
  Pain and Discomfort C13D1 | -11.39 (27.19) | -8.33 (29.97)
  Pain and Discomfort C14D1: number analyzed (Participants) | 55 | 44
  Pain and Discomfort C14D1 | -9.39 (25.21) | -3.79 (27.81)
  Pain and Discomfort C15D1: number analyzed (Participants) | 51 | 36
  Pain and Discomfort C15D1 | -8.82 (24.12) | -4.17 (29.11)
  Pain and Discomfort C16D1: number analyzed (Participants) | 48 | 31
  Pain and Discomfort C16D1 | -12.15 (24.73) | -5.38 (28.35)
  Pain and Discomfort C17D1: number analyzed (Participants) | 43 | 25
  Pain and Discomfort C17D1 | -9.69 (25.00) | -6.00 (28.41)
  Pain and Discomfort C18D1: number analyzed (Participants) | 41 | 21
  Pain and Discomfort C18D1 | -11.79 (22.44) | -6.35 (28.61)
  Pain and Discomfort C19D1: number analyzed (Participants) | 40 | 20
  Pain and Discomfort C19D1 | -5.83 (22.82) | -5.00 (17.18)
  Pain and Discomfort C20D1: number analyzed (Participants) | 39 | 19
  Pain and Discomfort C20D1 | -5.56 (19.99) | -7.02 (26.83)
  Pain and Discomfort C21D1: number analyzed (Participants) | 36 | 20
  Pain and Discomfort C21D1 | -7.41 (20.10) | -10.00 (23.82)
  Pain and Discomfort C22D1: number analyzed (Participants) | 31 | 17
  Pain and Discomfort C22D1 | -8.06 (21.89) | -5.88 (31.70)
  Pain and Discomfort C23D1: number analyzed (Participants) | 31 | 16
  Pain and Discomfort C23D1 | -10.22 (20.04) | -8.33 (29.81)
  Pain and Discomfort C24D1: number analyzed (Participants) | 29 | 12
  Pain and Discomfort C24D1 | -8.62 (21.19) | -8.33 (29.73)
  Pain and Discomfort C25D1: number analyzed (Participants) | 28 | 12
  Pain and Discomfort C25D1 | -11.90 (23.07) | -9.72 (32.14)
  Pain and Discomfort C26D1: number analyzed (Participants) | 26 | 9
  Pain and Discomfort C26D1 | -7.69 (26.76) | -1.85 (28.19)
  Pain and Discomfort C27D1: number analyzed (Participants) | 25 | 10
  Pain and Discomfort C27D1 | -12.00 (21.79) | -3.33 (15.32)
  Pain and Discomfort C28D1: number analyzed (Participants) | 21 | 11
  Pain and Discomfort C28D1 | -11.90 (22.45) | 3.03 (22.13)
  Pain and Discomfort C29D1: number analyzed (Participants) | 22 | 12
  Pain and Discomfort C29D1 | -12.88 (21.16) | -1.39 (11.14)
  Pain and Discomfort C30D1: number analyzed (Participants) | 20 | 0
  Pain and Discomfort C30D1 | -10.83 (24.35) |
  Pain and Discomfort C31D1: number analyzed (Participants) | 20 | 0
  Pain and Discomfort C31D1 | -15.00 (22.23) |
  Pain and Discomfort C32D1: number analyzed (Participants) | 18 | 0
  Pain and Discomfort C32D1 | -17.59 (18.50) |
  Pain and Discomfort C33D1: number analyzed (Participants) | 15 | 0
  Pain and Discomfort C33D1 | -13.33 (21.08) |
  Pain and Discomfort C34D1: number analyzed (Participants) | 12 | 0
  Pain and Discomfort C34D1 | -20.83 (23.70) |
  Pain and Discomfort C35D1: number analyzed (Participants) | 13 | 0
  Pain and Discomfort C35D1 | -21.79 (21.93) |
  Pain and Discomfort C36D1: number analyzed (Participants) | 12 | 0
  Pain and Discomfort C36D1 | -19.44 (17.16) |
  Pain and Discomfort C37D1: number analyzed (Participants) | 11 | 0
  Pain and Discomfort C37D1 | -13.64 (20.84) |
  Pain and Discomfort C38D1: number analyzed (Participants) | 10 | 0
  Pain and Discomfort C38D1 | -13.33 (33.15) |
  Pain and Discomfort C39D1: number analyzed (Participants) | 9 | 0
  Pain and Discomfort C39D1 | -22.22 (18.63) |
  Pain and Discomfort 30 day follow up: number analyzed (Participants) | 57 | 76
  Pain and Discomfort 30 day follow up | 0.88 (29.45) | 1.32 (27.99)
  Pain and Discomfort 90 day follow up: number analyzed (Participants) | 61 | 79
  Pain and Discomfort 90 day follow up | -1.37 (26.75) | -2.95 (23.08)
  Anxiety Baseline | 38.96 (28.31) | 42.05 (28.30)
  Anxiety C2D1: number analyzed (Participants) | 208 | 216
  Anxiety C2D1 | -3.93 (25.15) | -7.02 (25.23)
  Anxiety C3D1: number analyzed (Participants) | 182 | 196
  Anxiety C3D1 | -3.02 (24.93) | -6.04 (25.63)
  Anxiety C4D1: number analyzed (Participants) | 166 | 169
  Anxiety C4D1 | -4.12 (24.65) | -7.20 (26.96)
  Anxiety C5D1: number analyzed (Participants) | 159 | 165
  Anxiety C5D1 | -2.73 (26.24) | -6.77 (27.66)
  Anxiety C6D1: number analyzed (Participants) | 149 | 145
  Anxiety C6D1 | -6.04 (23.43) | -8.51 (29.14)
  Anxiety C7D1: number analyzed (Participants) | 119 | 125
  Anxiety C7D1 | -3.64 (23.28) | -8.80 (26.23)
  Anxiety C8D1: number analyzed (Participants) | 108 | 109
  Anxiety C8D1 | -4.32 (25.21) | -8.87 (29.79)
  Anxiety C9D1: number analyzed (Participants) | 102 | 103
  Anxiety C9D1 | -5.23 (25.80) | -6.96 (26.04)
  Anxiety C10D1: number analyzed (Participants) | 85 | 79
  Anxiety C10D1 | -7.45 (28.11) | -11.60 (32.40)
  Anxiety C11D1: number analyzed (Participants) | 80 | 71
  Anxiety C11D1 | -7.29 (28.54) | -8.69 (31.35)
  Anxiety C12D1: number analyzed (Participants) | 75 | 57
  Anxiety C12D1 | -10.00 (29.38) | -8.19 (31.67)
  Anxiety C13D1: number analyzed (Participants) | 60 | 48
  Anxiety C13D1 | -7.78 (30.76) | -6.60 (31.08)
  Anxiety C14D1: number analyzed (Participants) | 55 | 44
  Anxiety C14D1 | -7.88 (28.30) | -5.68 (31.53)
  Anxiety C15D1: number analyzed (Participants) | 51 | 36
  Anxiety C15D1 | -8.50 (28.55) | -6.02 (33.13)
  Anxiety C16D1: number analyzed (Participants) | 48 | 31
  Anxiety C16D1 | -15.62 (27.38) | -3.76 (37.44)
  Anxiety C17D1: number analyzed (Participants) | 43 | 25
  Anxiety C17D1 | -6.98 (24.19) | -6.67 (34.69)
  Anxiety C18D1: number analyzed (Participants) | 41 | 21
  Anxiety C18D1 | -7.32 (28.64) | -10.32 (37.07)
  Anxiety C19D1: number analyzed (Participants) | 40 | 20
  Anxiety C19D1 | -8.33 (25.88) | -2.50 (27.72)
  Anxiety C20D1: number analyzed (Participants) | 39 | 19
  Anxiety C20D1 | -9.83 (24.99) | -8.77 (35.73)
  Anxiety C21D1: number analyzed (Participants) | 36 | 20
  Anxiety C21D1 | -9.26 (29.93) | -11.67 (35.91)
  Anxiety C22D1: number analyzed (Participants) | 31 | 17
  Anxiety C22D1 | -4.84 (27.28) | -7.84 (40.45)
  Anxiety C23D1: number analyzed (Participants) | 31 | 16
  Anxiety C23D1 | -10.22 (26.76) | -10.42 (35.42)
  Anxiety C24D1: number analyzed (Participants) | 29 | 12
  Anxiety C24D1 | -9.77 (28.00) | -9.72 (41.72)
  Anxiety C25D1: number analyzed (Participants) | 28 | 12
  Anxiety C25D1 | -10.71 (24.52) | -11.11 (40.41)
  Anxiety C26D1: number analyzed (Participants) | 26 | 9
  Anxiety C26D1 | -7.69 (25.49) | 3.70 (34.13)
  Anxiety C27D1: number analyzed (Participants) | 25 | 10
  Anxiety C27D1 | -9.33 (30.08) | 6.67 (29.61)
  Anxiety C28D1: number analyzed (Participants) | 21 | 11
  Anxiety C28D1 | -10.32 (31.83) | 1.52 (29.30)
  Anxiety C29D1: number analyzed (Participants) | 22 | 12
  Anxiety C29D1 | -6.82 (33.20) | 1.39 (37.24)
  Anxiety C30D1: number analyzed (Participants) | 20 | 0
  Anxiety C30D1 | -5.00 (26.55) |
  Anxiety C31D1: number analyzed (Participants) | 20 | 0
  Anxiety C31D1 | -7.50 (28.34) |
  Anxiety C32D1: number analyzed (Participants) | 18 | 0
  Anxiety C32D1 | -10.19 (32.91) |
  Anxiety C33D1: number analyzed (Participants) | 15 | 0
  Anxiety C33D1 | -4.44 (30.52) |
  Anxiety C34D1: number analyzed (Participants) | 12 | 0
  Anxiety C34D1 | -13.89 (27.37) |
  Anxiety C35D1: number analyzed (Participants) | 13 | 0
  Anxiety C35D1 | -10.26 (25.04) |
  Anxiety C36D1: number analyzed (Participants) | 12 | 0
  Anxiety C36D1 | -12.50 (26.71) |
  Anxiety C37D1: number analyzed (Participants) | 11 | 0
  Anxiety C37D1 | -25.76 (20.23) |
  Anxiety C38D1: number analyzed (Participants) | 10 | 0
  Anxiety C38D1 | -18.33 (22.84) |
  Anxiety C39D1: number analyzed (Participants) | 9 | 0
  Anxiety C39D1 | -14.81 (34.81) |
  Anxiety 30 day follow up: number analyzed (Participants) | 57 | 76
  Anxiety 30 day follow up | 2.34 (31.25) | 3.51 (26.15)
  Anxiety 90 day follow up: number analyzed (Participants) | 61 | 79
  Anxiety 90 day follow up | 0.27 (27.47) | -4.22 (31.29)
  Eating in Front of Others Baseline | 10.70 (21.53) | 10.51 (22.36)
  Eating in Front of Others C2D1: number analyzed (Participants) | 208 | 216
  Eating in Front of Others C2D1 | -3.21 (18.25) | -3.09 (19.04)
  Eating in Front of Others C3D1: number analyzed (Participants) | 182 | 196
  Eating in Front of Others C3D1 | -2.01 (18.26) | -3.06 (19.15)
  Eating in Front of Others C4D1: number analyzed (Participants) | 166 | 169
  Eating in Front of Others C4D1 | -3.01 (16.34) | -7.10 (21.57)
  Eating in Front of Others C5D1: number analyzed (Participants) | 159 | 165
  Eating in Front of Others C5D1 | -1.68 (15.82) | -5.45 (23.37)
  Eating in Front of Others C6D1: number analyzed (Participants) | 149 | 145
  Eating in Front of Others C6D1 | -0.22 (15.25) | -4.83 (21.51)
  Eating in Front of Others C7D1: number analyzed (Participants) | 119 | 125
  Eating in Front of Others C7D1 | -0.84 (18.13) | -4.53 (20.45)
  Eating in Front of Others C8D1: number analyzed (Participants) | 108 | 109
  Eating in Front of Others C8D1 | -2.47 (18.63) | -5.81 (21.20)
  Eating in Front of Others C9D1: number analyzed (Participants) | 102 | 103
  Eating in Front of Others C9D1 | -1.63 (21.69) | -5.50 (21.44)
  Eating in Front of Others C10D1: number analyzed (Participants) | 85 | 79
  Eating in Front of Others C10D1 | -2.35 (23.45) | -6.33 (20.03)
  Eating in Front of Others C11D1: number analyzed (Participants) | 80 | 71
  Eating in Front of Others C11D1 | -2.92 (19.98) | -4.69 (19.76)
  Eating in Front of Others C12D1: number analyzed (Participants) | 75 | 57
  Eating in Front of Others C12D1 | -3.11 (20.63) | -4.09 (14.18)
  Eating in Front of Others C13D1: number analyzed (Participants) | 60 | 48
  Eating in Front of Others C13D1 | -5.56 (21.41) | 0.00 (16.84)
  Eating in Front of Others C14D1: number analyzed (Participants) | 55 | 44
  Eating in Front of Others C14D1 | -4.85 (20.71) | -4.55 (13.62)
  Eating in Front of Others C15D1: number analyzed (Participants) | 51 | 36
  Eating in Front of Others C15D1 | -8.50 (21.95) | -0.93 (9.71)
  Eating in Front of Others C16D1: number analyzed (Participants) | 48 | 31
  Eating in Front of Others C16D1 | -6.94 (18.14) | -1.08 (16.06)
  Eating in Front of Others C17D1: number analyzed (Participants) | 43 | 25
  Eating in Front of Others C17D1 | -6.20 (19.59) | 0.00 (16.67)
  Eating in Front of Others C18D1: number analyzed (Participants) | 41 | 21
  Eating in Front of Others C18D1 | -8.13 (19.41) | -3.17 (14.55)
  Eating in Front of Others C19D1: number analyzed (Participants) | 40 | 20
  Eating in Front of Others C19D1 | -10.83 (21.86) | -1.67 (7.45)
  Eating in Front of Others C20D1: number analyzed (Participants) | 39 | 19
  Eating in Front of Others C20D1 | -8.55 (19.82) | 0.00 (19.25)
  Eating in Front of Others C21D1: number analyzed (Participants) | 36 | 20
  Eating in Front of Others C21D1 | -8.33 (20.12) | -3.33 (14.91)
  Eating in Front of Others C22D1: number analyzed (Participants) | 31 | 17
  Eating in Front of Others C22D1 | -6.45 (18.09) | -3.92 (16.17)
  Eating in Front of Others C23D1: number analyzed (Participants) | 31 | 16
  Eating in Front of Others C23D1 | -7.53 (18.68) | -6.25 (18.13)
  Eating in Front of Others C24D1: number analyzed (Participants) | 29 | 12
  Eating in Front of Others C24D1 | -3.45 (18.57) | -5.56 (19.25)
  Eating in Front of Others C25D1: number analyzed (Participants) | 28 | 12
  Eating in Front of Others C25D1 | -2.38 (20.14) | -5.56 (19.25)
  Eating in Front of Others C26D1: number analyzed (Participants) | 26 | 9
  Eating in Front of Others C26D1 | -6.41 (18.90) | -3.70 (11.11)
  Eating in Front of Others C27D1: number analyzed (Participants) | 25 | 10
  Eating in Front of Others C27D1 | -2.67 (19.05) | 0.00 (0.00)
  Eating in Front of Others C28D1: number analyzed (Participants) | 21 | 11
  Eating in Front of Others C28D1 | -4.76 (26.43) | -3.03 (10.05)
  Eating in Front of Others C29D1: number analyzed (Participants) | 22 | 12
  Eating in Front of Others C29D1 | -9.09 (21.04) | 2.78 (9.62)
  Eating in Front of Others C30D1: number analyzed (Participants) | 20 | 0
  Eating in Front of Others C30D1 | -6.67 (23.20) |
  Eating in Front of Others C31D1: number analyzed (Participants) | 20 | 0
  Eating in Front of Others C31D1 | -10.00 (21.90) |
  Eating in Front of Others C32D1: number analyzed (Participants) | 18 | 0
  Eating in Front of Others C32D1 | -7.41 (24.40) |
  Eating in Front of Others C33D1: number analyzed (Participants) | 15 | 0
  Eating in Front of Others C33D1 | -8.89 (23.46) |
  Eating in Front of Others C34D1: number analyzed (Participants) | 12 | 0
  Eating in Front of Others C34D1 | -16.67 (22.47) |
  Eating in Front of Others C35D1: number analyzed (Participants) | 13 | 0
  Eating in Front of Others C35D1 | -5.13 (22.96) |
  Eating in Front of Others C36D1: number analyzed (Participants) | 12 | 0
  Eating in Front of Others C36D1 | -11.11 (21.71) |
  Eating in Front of Others C37D1: number analyzed (Participants) | 11 | 0
  Eating in Front of Others C37D1 | -12.12 (22.47) |
  Eating in Front of Others C38D1: number analyzed (Participants) | 10 | 0
  Eating in Front of Others C38D1 | -16.67 (23.57) |
  Eating in Front of Others C39D1: number analyzed (Participants) | 9 | 0
  Eating in Front of Others C39D1 | -7.41 (14.70) |
  Eating in Front of Others 30 day follow up: number analyzed (Participants) | 57 | 76
  Eating in Front of Others 30 day follow up | 2.92 (23.81) | 1.75 (24.28)
  Eating in Front of Others 90 day follow up: number analyzed (Participants) | 61 | 79
  Eating in Front of Others 90 day follow up | 3.28 (18.96) | 2.53 (16.69)
  Dry Mouth Baseline | 19.20 (24.74) | 16.87 (23.79)
  Dry Mouth C2D1: number analyzed (Participants) | 208 | 216
  Dry Mouth C2D1 | -0.32 (23.40) | 2.16 (23.30)
  Dry Mouth C3D1: number analyzed (Participants) | 182 | 196
  Dry Mouth C3D1 | -0.55 (23.89) | 4.93 (26.44)
  Dry Mouth C4D1: number analyzed (Participants) | 166 | 169
  Dry Mouth C4D1 | -2.01 (25.08) | 4.34 (28.30)
  Dry Mouth C5D1: number analyzed (Participants) | 159 | 165
  Dry Mouth C5D1 | -1.05 (26.89) | 1.41 (27.88)
  Dry Mouth C6D1: number analyzed (Participants) | 149 | 145
  Dry Mouth C6D1 | 0.89 (27.93) | 3.91 (27.64)
  Dry Mouth C7D1: number analyzed (Participants) | 119 | 125
  Dry Mouth C7D1 | -0.28 (27.62) | 0.53 (28.08)
  Dry Mouth C8D1: number analyzed (Participants) | 108 | 109
  Dry Mouth C8D1 | -1.85 (25.71) | 3.98 (29.65)
  Dry Mouth C9D1: number analyzed (Participants) | 102 | 103
  Dry Mouth C9D1 | 0.00 (28.92) | 2.27 (28.49)
  Dry Mouth C10D1: number analyzed (Participants) | 85 | 79
  Dry Mouth C10D1 | -5.88 (28.72) | -2.11 (27.39)
  Dry Mouth C11D1: number analyzed (Participants) | 80 | 71
  Dry Mouth C11D1 | -4.58 (26.38) | -2.35 (26.02)
  Dry Mouth C12D1: number analyzed (Participants) | 75 | 57
  Dry Mouth C12D1 | -5.78 (26.49) | 1.17 (25.17)
  Dry Mouth C13D1: number analyzed (Participants) | 60 | 48
  Dry Mouth C13D1 | -5.00 (26.63) | -2.08 (27.85)
  Dry Mouth C14D1: number analyzed (Participants) | 55 | 44
  Dry Mouth C14D1 | -7.27 (26.21) | -2.27 (26.31)
  Dry Mouth C15D1: number analyzed (Participants) | 51 | 36
  Dry Mouth C15D1 | -5.88 (24.68) | 0.00 (21.08)
  Dry Mouth C16D1: number analyzed (Participants) | 48 | 31
  Dry Mouth C16D1 | -7.64 (25.02) | 1.08 (16.06)
  Dry Mouth C17D1: number analyzed (Participants) | 43 | 25
  Dry Mouth C17D1 | -6.20 (19.59) | 4.00 (17.53)
  Dry Mouth C18D1: number analyzed (Participants) | 41 | 21
  Dry Mouth C18D1 | -5.69 (19.58) | 4.76 (15.94)
  Dry Mouth C19D1: number analyzed (Participants) | 40 | 20
  Dry Mouth C19D1 | -9.17 (25.02) | 3.33 (14.91)
  Dry Mouth C20D1: number analyzed (Participants) | 39 | 19
  Dry Mouth C20D1 | -8.55 (21.24) | 3.51 (24.58)
  Dry Mouth C21D1: number analyzed (Participants) | 36 | 20
  Dry Mouth C21D1 | -5.56 (24.56) | 3.33 (18.42)
  Dry Mouth C22D1: number analyzed (Participants) | 31 | 17
  Dry Mouth C22D1 | -9.68 (23.08) | 7.84 (18.74)
  Dry Mouth C23D1: number analyzed (Participants) | 31 | 16
  Dry Mouth C23D1 | -7.53 (23.90) | 2.08 (14.75)
  Dry Mouth C24D1: number analyzed (Participants) | 29 | 12
  Dry Mouth C24D1 | -6.90 (24.20) | 5.56 (27.83)
  Dry Mouth C25D1: number analyzed (Participants) | 28 | 12
  Dry Mouth C25D1 | -10.71 (22.32) | 2.78 (17.16)
  Dry Mouth C26D1: number analyzed (Participants) | 26 | 9
  Dry Mouth C26D1 | -8.97 (27.58) | 0.00 (16.67)
  Dry Mouth C27D1: number analyzed (Participants) | 25 | 10
  Dry Mouth C27D1 | -6.67 (21.52) | 3.33 (18.92)
  Dry Mouth C28D1: number analyzed (Participants) | 21 | 11
  Dry Mouth C28D1 | -4.76 (26.43) | 0.00 (14.91)
  Dry Mouth C29D1: number analyzed (Participants) | 22 | 12
  Dry Mouth C29D1 | -6.06 (28.43) | -2.78 (17.16)
  Dry Mouth C30D1: number analyzed (Participants) | 20 | 0
  Dry Mouth C30D1 | -5.00 (24.84) |
  Dry Mouth C31D1: number analyzed (Participants) | 20 | 0
  Dry Mouth C31D1 | -8.33 (28.36) |
  Dry Mouth C32D1: number analyzed (Participants) | 18 | 0
  Dry Mouth C32D1 | -11.11 (30.25) |
  Dry Mouth C33D1: number analyzed (Participants) | 15 | 0
  Dry Mouth C33D1 | -15.56 (21.33) |
  Dry Mouth C34D1: number analyzed (Participants) | 12 | 0
  Dry Mouth C34D1 | -22.22 (21.71) |
  Dry Mouth C35D1: number analyzed (Participants) | 13 | 0
  Dry Mouth C35D1 | -17.95 (25.88) |
  Dry Mouth C36D1: number analyzed (Participants) | 12 | 0
  Dry Mouth C36D1 | -16.67 (17.41) |
  Dry Mouth C37D1: number analyzed (Participants) | 11 | 0
  Dry Mouth C37D1 | -18.18 (31.14) |
  Dry Mouth C38D1: number analyzed (Participants) | 10 | 0
  Dry Mouth C38D1 | -20.00 (32.20) |
  Dry Mouth C39D1: number analyzed (Participants) | 9 | 0
  Dry Mouth C39D1 | -22.22 (33.33) |
  Dry Mouth 30 day follow up: number analyzed (Participants) | 57 | 76
  Dry Mouth 30 day follow up | -4.68 (26.31) | 5.70 (26.88)
  Dry Mouth 90 day follow up: number analyzed (Participants) | 61 | 79
  Dry Mouth 90 day follow up | 3.83 (25.16) | 6.75 (28.43)
  Trouble with Taste Baseline | 9.47 (21.58) | 7.47 (18.50)
  Trouble with Taste C2D1: number analyzed (Participants) | 208 | 216
  Trouble with Taste C2D1 | 3.85 (22.85) | 2.47 (20.69)
  Trouble with Taste C3D1: number analyzed (Participants) | 182 | 196
  Trouble with Taste C3D1 | 7.33 (25.41) | 5.27 (20.55)
  Trouble with Taste C4D1: number analyzed (Participants) | 166 | 169
  Trouble with Taste C4D1 | 5.62 (24.24) | 5.52 (24.31)
  Trouble with Taste C5D1: number analyzed (Participants) | 159 | 165
  Trouble with Taste C5D1 | 8.18 (26.71) | 8.08 (25.01)
  Trouble with Taste C6D1: number analyzed (Participants) | 149 | 145
  Trouble with Taste C6D1 | 12.30 (27.77) | 11.72 (27.65)
  Trouble with Taste C7D1: number analyzed (Participants) | 119 | 125
  Trouble with Taste C7D1 | 10.92 (28.82) | 9.33 (25.96)
  Trouble with Taste C8D1: number analyzed (Participants) | 108 | 109
  Trouble with Taste C8D1 | 10.49 (25.23) | 10.40 (28.58)
  Trouble with Taste C9D1: number analyzed (Participants) | 102 | 103
  Trouble with Taste C9D1 | 8.17 (29.83) | 6.47 (25.16)
  Trouble with Taste C10D1: number analyzed (Participants) | 85 | 79
  Trouble with Taste C10D1 | 7.06 (29.59) | 2.95 (26.25)
  Trouble with Taste C11D1: number analyzed (Participants) | 80 | 71
  Trouble with Taste C11D1 | 2.92 (27.14) | 4.23 (26.39)
  Trouble with Taste C12D1: number analyzed (Participants) | 75 | 57
  Trouble with Taste C12D1 | 2.22 (26.47) | 0.00 (21.82)
  Trouble with Taste C13D1: number analyzed (Participants) | 60 | 48
  Trouble with Taste C13D1 | 0.56 (32.18) | 3.47 (19.74)
  Trouble with Taste C14D1: number analyzed (Participants) | 55 | 44
  Trouble with Taste C14D1 | 1.82 (25.99) | 1.52 (22.68)
  Trouble with Taste C15D1: number analyzed (Participants) | 51 | 36
  Trouble with Taste C15D1 | 0.00 (27.49) | 1.85 (23.83)
  Trouble with Taste C16D1: number analyzed (Participants) | 48 | 31
  Trouble with Taste C16D1 | 1.39 (25.69) | 3.23 (15.76)
  Trouble with Taste C17D1: number analyzed (Participants) | 43 | 25
  Trouble with Taste C17D1 | 1.55 (24.07) | 8.00 (14.53)
  Trouble with Taste C18D1: number analyzed (Participants) | 41 | 21
  Trouble with Taste C18D1 | 0.81 (24.14) | 4.76 (11.95)
  Trouble with Taste C19D1: number analyzed (Participants) | 40 | 20
  Trouble with Taste C19D1 | 0.83 (21.99) | 1.67 (7.45)
  Trouble with Taste C20D1: number analyzed (Participants) | 39 | 19
  Trouble with Taste C20D1 | 2.56 (22.14) | 7.02 (13.96)
  Trouble with Taste C21D1: number analyzed (Participants) | 36 | 20
  Trouble with Taste C21D1 | -0.93 (24.54) | 10.00 (15.67)
  Trouble with Taste C22D1: number analyzed (Participants) | 31 | 17
  Trouble with Taste C22D1 | -1.08 (26.50) | 5.88 (13.10)
  Trouble with Taste C23D1: number analyzed (Participants) | 31 | 16
  Trouble with Taste C23D1 | 2.15 (24.24) | 8.33 (19.25)
  Trouble with Taste C24D1: number analyzed (Participants) | 29 | 12
  Trouble with Taste C24D1 | 0.00 (19.92) | 2.78 (9.62)
  Trouble with Taste C25D1: number analyzed (Participants) | 28 | 12
  Trouble with Taste C25D1 | 2.38 (20.14) | 5.56 (12.97)
  Trouble with Taste C26D1: number analyzed (Participants) | 26 | 9
  Trouble with Taste C26D1 | -1.28 (19.96) | 11.11 (16.67)
  Trouble with Taste C27D1: number analyzed (Participants) | 25 | 10
  Trouble with Taste C27D1 | 0.00 (19.25) | 3.33 (10.54)
  Trouble with Taste C28D1: number analyzed (Participants) | 21 | 11
  Trouble with Taste C28D1 | 3.17 (23.34) | 3.03 (10.05)
  Trouble with Taste C29D1: number analyzed (Participants) | 22 | 12
  Trouble with Taste C29D1 | 4.55 (21.32) | 8.33 (15.08)
  Trouble with Taste C30D1: number analyzed (Participants) | 20 | 0
  Trouble with Taste C30D1 | 1.67 (20.16) |
  Trouble with Taste C31D1: number analyzed (Participants) | 20 | 0
  Trouble with Taste C31D1 | 1.67 (22.88) |
  Trouble with Taste C32D1: number analyzed (Participants) | 18 | 0
  Trouble with Taste C32D1 | 0.00 (22.87) |
  Trouble with Taste C33D1: number analyzed (Participants) | 15 | 0
  Trouble with Taste C33D1 | -2.22 (23.46) |
  Trouble with Taste C34D1: number analyzed (Participants) | 12 | 0
  Trouble with Taste C34D1 | -8.33 (20.72) |
  Trouble with Taste C35D1: number analyzed (Participants) | 13 | 0
  Trouble with Taste C35D1 | -2.56 (21.35) |
  Trouble with Taste C36D1: number analyzed (Participants) | 12 | 0
  Trouble with Taste C36D1 | -2.78 (22.29) |
  Trouble with Taste C37D1: number analyzed (Participants) | 11 | 0
  Trouble with Taste C37D1 | -3.03 (27.71) |
  Trouble with Taste C38D1: number analyzed (Participants) | 10 | 0
  Trouble with Taste C38D1 | -3.33 (29.19) |
  Trouble with Taste C39D1: number analyzed (Participants) | 9 | 0
  Trouble with Taste C39D1 | 0.00 (16.67) |
  Trouble with Taste 30 day follow up: number analyzed (Participants) | 57 | 76
  Trouble with Taste 30 day follow up | 4.09 (23.63) | 9.21 (29.11)
  Trouble with Taste 90 day follow up: number analyzed (Participants) | 61 | 79
  Trouble with Taste 90 day follow up | 7.65 (25.38) | 7.59 (22.61)
  Body Image Baseline | 17.97 (25.75) | 19.64 (23.99)
  Body Image C2D1: number analyzed (Participants) | 208 | 216
  Body Image C2D1 | -0.80 (22.80) | -2.31 (22.04)
  Body Image C3D1: number analyzed (Participants) | 182 | 196
  Body Image C3D1 | 1.47 (24.48) | -1.53 (23.94)
  Body Image C4D1: number analyzed (Participants) | 166 | 169
  Body Image C4D1 | 1.00 (26.32) | -0.99 (22.25)
  Body Image C5D1: number analyzed (Participants) | 159 | 165
  Body Image C5D1 | 2.52 (28.45) | 0.61 (22.83)
  Body Image C6D1: number analyzed (Participants) | 149 | 145
  Body Image C6D1 | 3.58 (24.55) | -1.38 (26.61)
  Body Image C7D1: number analyzed (Participants) | 119 | 125
  Body Image C7D1 | 0.28 (25.85) | -0.80 (25.56)
  Body Image C8D1: number analyzed (Participants) | 108 | 109
  Body Image C8D1 | 2.78 (26.62) | 0.00 (24.43)
  Body Image C9D1: number analyzed (Participants) | 102 | 103
  Body Image C9D1 | 1.31 (24.34) | -0.97 (24.01)
  Body Image C10D1: number analyzed (Participants) | 85 | 79
  Body Image C10D1 | -1.57 (29.95) | -0.42 (26.95)
  Body Image C11D1: number analyzed (Participants) | 80 | 71
  Body Image C11D1 | -5.00 (26.57) | 0.94 (26.41)
  Body Image C12D1: number analyzed (Participants) | 75 | 57
  Body Image C12D1 | -3.56 (29.29) | -2.34 (22.59)
  Body Image C13D1: number analyzed (Participants) | 60 | 48
  Body Image C13D1 | -7.22 (30.12) | 0.00 (26.63)
  Body Image C14D1: number analyzed (Participants) | 55 | 44
  Body Image C14D1 | -6.06 (27.29) | -2.27 (25.31)
  Body Image C15D1: number analyzed (Participants) | 51 | 36
  Body Image C15D1 | -5.88 (28.83) | -0.93 (28.16)
  Body Image C16D1: number analyzed (Participants) | 48 | 31
  Body Image C16D1 | -7.64 (27.71) | 1.08 (26.50)
  Body Image C17D1: number analyzed (Participants) | 43 | 25
  Body Image C17D1 | -6.20 (27.46) | -2.67 (23.41)
  Body Image C18D1: number analyzed (Participants) | 41 | 21
  Body Image C18D1 | -8.13 (25.58) | -4.76 (26.43)
  Body Image C19D1: number analyzed (Participants) | 40 | 20
  Body Image C19D1 | -6.67 (24.11) | -1.67 (13.13)
  Body Image C20D1: number analyzed (Participants) | 39 | 19
  Body Image C20D1 | -3.42 (23.93) | -3.51 (29.18)
  Body Image C21D1: number analyzed (Participants) | 36 | 20
  Body Image C21D1 | -9.26 (20.49) | -8.33 (23.88)
  Body Image C22D1: number analyzed (Participants) | 31 | 17
  Body Image C22D1 | -5.38 (24.49) | -3.92 (30.92)
  Body Image C23D1: number analyzed (Participants) | 31 | 16
  Body Image C23D1 | -8.60 (19.18) | -8.33 (28.54)
  Body Image C24D1: number analyzed (Participants) | 29 | 12
  Body Image C24D1 | -8.05 (17.03) | -5.56 (34.33)
  Body Image C25D1: number analyzed (Participants) | 28 | 12
  Body Image C25D1 | -8.33 (23.35) | -2.78 (33.21)
  Body Image C26D1: number analyzed (Participants) | 26 | 9
  Body Image C26D1 | -6.41 (23.13) | 3.70 (11.11)
  Body Image C27D1: number analyzed (Participants) | 25 | 10
  Body Image C27D1 | -6.67 (19.25) | 3.33 (10.54)
  Body Image C28D1: number analyzed (Participants) | 21 | 11
  Body Image C28D1 | -9.52 (21.46) | 6.06 (13.48)
  Body Image C29D1: number analyzed (Participants) | 22 | 12
  Body Image C29D1 | -9.09 (25.58) | 5.56 (12.97)
  Body Image C30D1: number analyzed (Participants) | 20 | 0
  Body Image C30D1 | -3.33 (21.36) |
  Body Image C31D1: number analyzed (Participants) | 20 | 0
  Body Image C31D1 | -10.00 (21.90) |
  Body Image C32D1: number analyzed (Participants) | 18 | 0
  Body Image C32D1 | -11.11 (22.87) |
  Body Image C33D1: number analyzed (Participants) | 15 | 0
  Body Image C33D1 | -15.56 (24.77) |
  Body Image C34D1: number analyzed (Participants) | 12 | 0
  Body Image C34D1 | -13.89 (17.16) |
  Body Image C35D1: number analyzed (Participants) | 13 | 0
  Body Image C35D1 | -10.26 (16.01) |
  Body Image C36D1: number analyzed (Participants) | 12 | 0
  Body Image C36D1 | -11.11 (16.41) |
  Body Image C37D1: number analyzed (Participants) | 11 | 0
  Body Image C37D1 | -15.15 (17.41) |
  Body Image C38D1: number analyzed (Participants) | 10 | 0
  Body Image C38D1 | -16.67 (17.57) |
  Body Image C39D1: number analyzed (Participants) | 9 | 0
  Body Image C39D1 | -11.11 (16.67) |
  Body Image 30 day follow up: number analyzed (Participants) | 57 | 76
  Body Image 30 day follow up | 3.51 (30.00) | 5.26 (26.70)
  Body Image 90 day follow up: number analyzed (Participants) | 61 | 79
  Body Image 90 day follow up | 7.10 (20.29) | 6.75 (29.42)
  Trouble Swallowing Saliva Baseline | 3.84 (12.64) | 5.26 (15.52)
  Trouble Swallowing Saliva C2D1: number analyzed (Participants) | 208 | 216
  Trouble Swallowing Saliva C2D1 | 0.48 (13.70) | -1.85 (14.62)
  Trouble Swallowing Saliva C3D1: number analyzed (Participants) | 182 | 196
  Trouble Swallowing Saliva C3D1 | 0.00 (13.57) | -1.19 (15.97)
  Trouble Swallowing Saliva C4D1: number analyzed (Participants) | 166 | 169
  Trouble Swallowing Saliva C4D1 | 0.20 (16.20) | -0.59 (16.05)
  Trouble Swallowing Saliva C5D1: number analyzed (Participants) | 159 | 165
  Trouble Swallowing Saliva C5D1 | 0.21 (15.23) | -2.63 (16.04)
  Trouble Swallowing Saliva C6D1: number analyzed (Participants) | 149 | 145
  Trouble Swallowing Saliva C6D1 | 2.91 (18.96) | 0.00 (18.84)
  Trouble Swallowing Saliva C7D1: number analyzed (Participants) | 119 | 125
  Trouble Swallowing Saliva C7D1 | 1.40 (18.61) | -1.33 (18.16)
  Trouble Swallowing Saliva C8D1: number analyzed (Participants) | 108 | 109
  Trouble Swallowing Saliva C8D1 | -0.62 (15.77) | -3.06 (16.06)
  Trouble Swallowing Saliva C9D1: number analyzed (Participants) | 102 | 103
  Trouble Swallowing Saliva C9D1 | 0.65 (15.54) | -3.56 (19.75)
  Trouble Swallowing Saliva C10D1: number analyzed (Participants) | 85 | 79
  Trouble Swallowing Saliva C10D1 | 0.78 (17.04) | -4.22 (20.23)
  Trouble Swallowing Saliva C11D1: number analyzed (Participants) | 80 | 71
  Trouble Swallowing Saliva C11D1 | -0.42 (13.52) | -4.69 (18.94)
  Trouble Swallowing Saliva C12D1: number analyzed (Participants) | 75 | 57
  Trouble Swallowing Saliva C12D1 | 0.00 (10.96) | -4.68 (19.35)
  Trouble Swallowing Saliva C13D1: number analyzed (Participants) | 60 | 48
  Trouble Swallowing Saliva C13D1 | 0.00 (12.27) | -2.78 (19.25)
  Trouble Swallowing Saliva C14D1: number analyzed (Participants) | 55 | 44
  Trouble Swallowing Saliva C14D1 | -1.21 (11.04) | -3.79 (25.13)
  Trouble Swallowing Saliva C15D1: number analyzed (Participants) | 51 | 36
  Trouble Swallowing Saliva C15D1 | -1.96 (14.00) | -6.48 (23.66)
  Trouble Swallowing Saliva C16D1: number analyzed (Participants) | 48 | 31
  Trouble Swallowing Saliva C16D1 | 0.00 (16.84) | -4.30 (20.62)
  Trouble Swallowing Saliva C17D1: number analyzed (Participants) | 43 | 25
  Trouble Swallowing Saliva C17D1 | -2.33 (13.40) | -6.67 (19.25)
  Trouble Swallowing Saliva C18D1: number analyzed (Participants) | 41 | 21
  Trouble Swallowing Saliva C18D1 | -2.44 (13.72) | -6.35 (22.65)
  Trouble Swallowing Saliva C19D1: number analyzed (Participants) | 40 | 20
  Trouble Swallowing Saliva C19D1 | -0.83 (15.99) | -5.00 (16.31)
  Trouble Swallowing Saliva C20D1: number analyzed (Participants) | 39 | 19
  Trouble Swallowing Saliva C20D1 | -3.42 (16.75) | -7.02 (23.78)
  Trouble Swallowing Saliva C21D1: number analyzed (Participants) | 36 | 20
  Trouble Swallowing Saliva C21D1 | 0.00 (17.82) | -5.00 (27.09)
  Trouble Swallowing Saliva C22D1: number analyzed (Participants) | 31 | 17
  Trouble Swallowing Saliva C22D1 | 0.00 (12.17) | -5.88 (24.25)
  Trouble Swallowing Saliva C23D1: number analyzed (Participants) | 31 | 16
  Trouble Swallowing Saliva C23D1 | 0.00 (12.17) | -10.42 (23.47)
  Trouble Swallowing Saliva C24D1: number analyzed (Participants) | 29 | 12
  Trouble Swallowing Saliva C24D1 | 0.00 (12.60) | -8.33 (20.72)
  Trouble Swallowing Saliva C25D1: number analyzed (Participants) | 28 | 12
  Trouble Swallowing Saliva C25D1 | 1.19 (14.29) | -13.89 (26.43)
  Trouble Swallowing Saliva C26D1: number analyzed (Participants) | 26 | 9
  Trouble Swallowing Saliva C26D1 | -1.28 (11.47) | -11.11 (23.57)
  Trouble Swallowing Saliva C27D1: number analyzed (Participants) | 25 | 10
  Trouble Swallowing Saliva C27D1 | 0.00 (13.61) | -10.00 (22.50)
  Trouble Swallowing Saliva C28D1: number analyzed (Participants) | 21 | 11
  Trouble Swallowing Saliva C28D1 | 0.00 (10.54) | -9.09 (21.56)
  Trouble Swallowing Saliva C29D1: number analyzed (Participants) | 22 | 12
  Trouble Swallowing Saliva C29D1 | 1.52 (12.50) | -8.33 (20.72)
  Trouble Swallowing Saliva C30D1: number analyzed (Participants) | 20 | 0
  Trouble Swallowing Saliva C30D1 | 0.00 (10.81) |
  Trouble Swallowing Saliva C31D1: number analyzed (Participants) | 20 | 0
  Trouble Swallowing Saliva C31D1 | 0.00 (10.81) |
  Trouble Swallowing Saliva C32D1: number analyzed (Participants) | 18 | 0
  Trouble Swallowing Saliva C32D1 | -1.85 (7.86) |
  Trouble Swallowing Saliva C33D1: number analyzed (Participants) | 15 | 0
  Trouble Swallowing Saliva C33D1 | -2.22 (8.61) |
  Trouble Swallowing Saliva C34D1: number analyzed (Participants) | 12 | 0
  Trouble Swallowing Saliva C34D1 | 0.00 (14.21) |
  Trouble Swallowing Saliva C35D1: number analyzed (Participants) | 13 | 0
  Trouble Swallowing Saliva C35D1 | 0.00 (13.61) |
  Trouble Swallowing Saliva C36D1: number analyzed (Participants) | 12 | 0
  Trouble Swallowing Saliva C36D1 | -2.78 (9.62) |
  Trouble Swallowing Saliva C37D1: number analyzed (Participants) | 11 | 0
  Trouble Swallowing Saliva C37D1 | 0.00 (14.91) |
  Trouble Swallowing Saliva C38D1: number analyzed (Participants) | 10 | 0
  Trouble Swallowing Saliva C38D1 | 0.00 (15.71) |
  Trouble Swallowing Saliva C39D1: number analyzed (Participants) | 9 | 0
  Trouble Swallowing Saliva C39D1 | 0.00 (0.00) |
  Trouble Swallowing Saliva 30 day follow up: number analyzed (Participants) | 57 | 76
  Trouble Swallowing Saliva 30 day follow up | 1.75 (20.34) | -1.75 (17.12)
  Trouble Swallowing Saliva 90 day follow up: number analyzed (Participants) | 61 | 79
  Trouble Swallowing Saliva 90 day follow up | 1.64 (16.58) | -2.95 (21.48)
  Choked When Swallowing Baseline | 5.35 (14.01) | 6.64 (17.00)
  Choked When Swallowing C2D1: number analyzed (Participants) | 208 | 216
  Choked When Swallowing C2D1 | -1.60 (13.81) | -1.54 (15.00)
  Choked When Swallowing C3D1: number analyzed (Participants) | 182 | 196
  Choked When Swallowing C3D1 | -1.10 (12.09) | -1.87 (17.92)
  Choked When Swallowing C4D1: number analyzed (Participants) | 166 | 169
  Choked When Swallowing C4D1 | -2.01 (14.07) | -1.38 (16.41)
  Choked When Swallowing C5D1: number analyzed (Participants) | 159 | 165
  Choked When Swallowing C5D1 | -1.68 (15.82) | -2.42 (17.09)
  Choked When Swallowing C6D1: number analyzed (Participants) | 149 | 145
  Choked When Swallowing C6D1 | -1.12 (15.70) | -1.84 (18.33)
  Choked When Swallowing C7D1: number analyzed (Participants) | 119 | 125
  Choked When Swallowing C7D1 | 0.56 (19.40) | -2.93 (19.41)
  Choked When Swallowing C8D1: number analyzed (Participants) | 108 | 109
  Choked When Swallowing C8D1 | -0.31 (14.76) | -3.67 (18.89)
  Choked When Swallowing C9D1: number analyzed (Participants) | 102 | 103
  Choked When Swallowing C9D1 | -0.65 (14.82) | -2.27 (19.95)
  Choked When Swallowing C10D1: number analyzed (Participants) | 85 | 79
  Choked When Swallowing C10D1 | -1.96 (14.87) | -2.95 (19.39)
  Choked When Swallowing C11D1: number analyzed (Participants) | 80 | 71
  Choked When Swallowing C11D1 | -0.83 (14.98) | -2.82 (18.47)
  Choked When Swallowing C12D1: number analyzed (Participants) | 75 | 57
  Choked When Swallowing C12D1 | -2.22 (14.84) | -1.75 (15.96)
  Choked When Swallowing C13D1: number analyzed (Participants) | 60 | 48
  Choked When Swallowing C13D1 | -3.33 (14.65) | -4.17 (18.99)
  Choked When Swallowing C14D1: number analyzed (Participants) | 55 | 44
  Choked When Swallowing C14D1 | -3.03 (11.61) | -1.52 (21.51)
  Choked When Swallowing C15D1: number analyzed (Participants) | 51 | 36
  Choked When Swallowing C15D1 | -3.92 (12.73) | 0.93 (24.54)
  Choked When Swallowing C16D1: number analyzed (Participants) | 48 | 31
  Choked When Swallowing C16D1 | -2.08 (12.69) | 1.08 (21.92)
  Choked When Swallowing C17D1: number analyzed (Participants) | 43 | 25
  Choked When Swallowing C17D1 | -1.55 (7.10) | -4.00 (22.19)
  Choked When Swallowing C18D1: number analyzed (Participants) | 41 | 21
  Choked When Swallowing C18D1 | -0.81 (11.76) | -3.17 (17.97)
  Choked When Swallowing C19D1: number analyzed (Participants) | 40 | 20
  Choked When Swallowing C19D1 | -1.67 (10.54) | -1.67 (7.45)
  Choked When Swallowing C20D1: number analyzed (Participants) | 39 | 19
  Choked When Swallowing C20D1 | -2.56 (11.81) | -3.51 (18.90)
  Choked When Swallowing C21D1: number analyzed (Participants) | 36 | 20
  Choked When Swallowing C21D1 | -1.85 (15.83) | -5.00 (16.31)
  Choked When Swallowing C22D1: number analyzed (Participants) | 31 | 17
  Choked When Swallowing C22D1 | -2.15 (11.97) | -3.92 (20.01)
  Choked When Swallowing C23D1: number analyzed (Participants) | 31 | 16
  Choked When Swallowing C23D1 | -2.15 (14.75) | -4.17 (20.64)
  Choked When Swallowing C24D1: number analyzed (Participants) | 29 | 12
  Choked When Swallowing C24D1 | -1.15 (14.04) | -5.56 (19.25)
  Choked When Swallowing C25D1: number analyzed (Participants) | 28 | 12
  Choked When Swallowing C25D1 | -3.57 (13.88) | -5.56 (19.25)
  Choked When Swallowing C26D1: number analyzed (Participants) | 26 | 9
  Choked When Swallowing C26D1 | -2.56 (13.07) | 0.00 (0.00)
  Choked When Swallowing C27D1: number analyzed (Participants) | 25 | 10
  Choked When Swallowing C27D1 | -1.33 (17.95) | 0.00 (0.00)
  Choked When Swallowing C28D1: number analyzed (Participants) | 21 | 11
  Choked When Swallowing C28D1 | 0.00 (18.26) | 0.00 (0.00)
  Choked When Swallowing C29D1: number analyzed (Participants) | 22 | 12
  Choked When Swallowing C29D1 | 1.52 (16.19) | -2.78 (9.62)
  Choked When Swallowing C30D1: number analyzed (Participants) | 20 | 0
  Choked When Swallowing C30D1 | 3.33 (18.42) |
  Choked When Swallowing C31D1: number analyzed (Participants) | 20 | 0
  Choked When Swallowing C31D1 | 1.67 (17.01) |
  Choked When Swallowing C32D1: number analyzed (Participants) | 18 | 0
  Choked When Swallowing C32D1 | 0.00 (19.80) |
  Choked When Swallowing C33D1: number analyzed (Participants) | 15 | 0
  Choked When Swallowing C33D1 | -2.22 (15.26) |
  Choked When Swallowing C34D1: number analyzed (Participants) | 12 | 0
  Choked When Swallowing C34D1 | 0.00 (20.10) |
  Choked When Swallowing C35D1: number analyzed (Participants) | 13 | 0
  Choked When Swallowing C35D1 | 2.56 (21.35) |
  Choked When Swallowing C36D1: number analyzed (Participants) | 12 | 0
  Choked When Swallowing C36D1 | 2.78 (17.16) |
  Choked When Swallowing C37D1: number analyzed (Participants) | 11 | 0
  Choked When Swallowing C37D1 | -3.03 (17.98) |
  Choked When Swallowing C38D1: number analyzed (Participants) | 10 | 0
  Choked When Swallowing C38D1 | -3.33 (18.92) |
  Choked When Swallowing C39D1: number analyzed (Participants) | 9 | 0
  Choked When Swallowing C39D1 | 0.00 (16.67) |
  Choked When Swallowing 30 day follow up: number analyzed (Participants) | 57 | 76
  Choked When Swallowing 30 day follow up | 4.09 (21.89) | -3.07 (19.00)
  Choked When Swallowing 90 day follow up: number analyzed (Participants) | 61 | 79
  Choked When Swallowing 90 day follow up | 0.00 (14.91) | -1.69 (21.94)
  Trouble with Coughing Baseline | 10.56 (17.49) | 9.82 (19.49)
  Trouble with Coughing C2D1: number analyzed (Participants) | 208 | 216
  Trouble with Coughing C2D1 | -0.48 (16.86) | -0.77 (18.59)
  Trouble with Coughing C3D1: number analyzed (Participants) | 182 | 196
  Trouble with Coughing C3D1 | -2.01 (17.92) | -0.68 (19.08)
  Trouble with Coughing C4D1: number analyzed (Participants) | 166 | 169
  Trouble with Coughing C4D1 | -1.61 (19.00) | -0.99 (20.39)
  Trouble with Coughing C5D1: number analyzed (Participants) | 159 | 165
  Trouble with Coughing C5D1 | 0.21 (19.30) | -2.63 (18.03)
  Trouble with Coughing C6D1: number analyzed (Participants) | 149 | 145
  Trouble with Coughing C6D1 | 0.22 (23.41) | -1.38 (16.61)
  Trouble with Coughing C7D1: number analyzed (Participants) | 119 | 125
  Trouble with Coughing C7D1 | -2.24 (19.76) | -1.87 (19.54)
  Trouble with Coughing C8D1: number analyzed (Participants) | 108 | 109
  Trouble with Coughing C8D1 | -0.31 (17.94) | -1.22 (20.75)
  Trouble with Coughing C9D1: number analyzed (Participants) | 102 | 103
  Trouble with Coughing C9D1 | -3.92 (20.06) | -2.91 (21.44)
  Trouble with Coughing C10D1: number analyzed (Participants) | 85 | 79
  Trouble with Coughing C10D1 | -3.53 (22.43) | -2.11 (25.79)
  Trouble with Coughing C11D1: number analyzed (Participants) | 80 | 71
  Trouble with Coughing C11D1 | -4.17 (22.73) | -4.23 (25.15)
  Trouble with Coughing C12D1: number analyzed (Participants) | 75 | 57
  Trouble with Coughing C12D1 | -2.67 (23.09) | -8.19 (22.96)
  Trouble with Coughing C13D1: number analyzed (Participants) | 60 | 48
  Trouble with Coughing C13D1 | -5.00 (25.91) | -6.94 (22.76)
  Trouble with Coughing C14D1: number analyzed (Participants) | 55 | 44
  Trouble with Coughing C14D1 | -6.06 (15.83) | -6.82 (23.38)
  Trouble with Coughing C15D1: number analyzed (Participants) | 51 | 36
  Trouble with Coughing C15D1 | -7.19 (20.35) | -7.41 (21.25)
  Trouble with Coughing C16D1: number analyzed (Participants) | 48 | 31
  Trouble with Coughing C16D1 | -4.17 (23.44) | -8.60 (19.18)
  Trouble with Coughing C17D1: number analyzed (Participants) | 43 | 25
  Trouble with Coughing C17D1 | -7.75 (22.81) | 1.33 (17.95)
  Trouble with Coughing C18D1: number analyzed (Participants) | 41 | 21
  Trouble with Coughing C18D1 | -6.50 (21.37) | -4.76 (19.11)
  Trouble with Coughing C19D1: number analyzed (Participants) | 40 | 20
  Trouble with Coughing C19D1 | -5.00 (17.78) | -1.67 (7.45)
  Trouble with Coughing C20D1: number analyzed (Participants) | 39 | 19
  Trouble with Coughing C20D1 | -3.42 (19.93) | -5.26 (22.94)
  Trouble with Coughing C21D1: number analyzed (Participants) | 36 | 20
  Trouble with Coughing C21D1 | -4.63 (19.76) | -1.67 (20.16)
  Trouble with Coughing C22D1: number analyzed (Participants) | 31 | 17
  Trouble with Coughing C22D1 | -5.38 (17.42) | -5.88 (21.20)
  Trouble with Coughing C23D1: number analyzed (Participants) | 31 | 16
  Trouble with Coughing C23D1 | -4.30 (18.74) | -6.25 (21.84)
  Trouble with Coughing C24D1: number analyzed (Participants) | 29 | 12
  Trouble with Coughing C24D1 | -3.45 (18.57) | -5.56 (23.92)
  Trouble with Coughing C25D1: number analyzed (Participants) | 28 | 12
  Trouble with Coughing C25D1 | -2.38 (17.98) | -5.56 (19.25)
  Trouble with Coughing C26D1: number analyzed (Participants) | 26 | 9
  Trouble with Coughing C26D1 | -1.28 (17.59) | -3.70 (20.03)
  Trouble with Coughing C27D1: number analyzed (Participants) | 25 | 10
  Trouble with Coughing C27D1 | -4.00 (17.53) | -3.33 (18.92)
  Trouble with Coughing C28D1: number analyzed (Participants) | 21 | 11
  Trouble with Coughing C28D1 | -1.59 (12.81) | 0.00 (21.08)
  Trouble with Coughing C29D1: number analyzed (Participants) | 22 | 12
  Trouble with Coughing C29D1 | 3.03 (22.79) | -2.78 (17.16)
  Trouble with Coughing C30D1: number analyzed (Participants) | 20 | 0
  Trouble with Coughing C30D1 | 1.67 (17.01) |
  Trouble with Coughing C31D1: number analyzed (Participants) | 20 | 0
  Trouble with Coughing C31D1 | 3.33 (21.36) |
  Trouble with Coughing C32D1: number analyzed (Participants) | 18 | 0
  Trouble with Coughing C32D1 | 3.70 (19.43) |
  Trouble with Coughing C33D1: number analyzed (Participants) | 15 | 0
  Trouble with Coughing C33D1 | -4.44 (11.73) |
  Trouble with Coughing C34D1: number analyzed (Participants) | 12 | 0
  Trouble with Coughing C34D1 | 0.00 (14.21) |
  Trouble with Coughing C35D1: number analyzed (Participants) | 13 | 0
  Trouble with Coughing C35D1 | -2.56 (16.45) |
  Trouble with Coughing C36D1: number analyzed (Participants) | 12 | 0
  Trouble with Coughing C36D1 | -5.56 (12.97) |
  Trouble with Coughing C37D1: number analyzed (Participants) | 11 | 0
  Trouble with Coughing C37D1 | -6.06 (13.48) |
  Trouble with Coughing C38D1: number analyzed (Participants) | 10 | 0
  Trouble with Coughing C38D1 | 0.00 (15.71) |
  Trouble with Coughing C39D1: number analyzed (Participants) | 9 | 0
  Trouble with Coughing C39D1 | 3.70 (11.11) |
  Trouble with Coughing 30 day follow up: number analyzed (Participants) | 57 | 76
  Trouble with Coughing 30 day follow up | 1.17 (21.79) | 1.32 (28.51)
  Trouble with Coughing 90 day follow up: number analyzed (Participants) | 61 | 79
  Trouble with Coughing 90 day follow up | 2.19 (15.95) | 1.27 (25.29)
  Trouble Talking Baseline | 3.84 (14.34) | 3.60 (12.40)
  Trouble Talking C2D1: number analyzed (Participants) | 208 | 216
  Trouble Talking C2D1 | 0.96 (13.07) | -0.31 (9.64)
  Trouble Talking C3D1: number analyzed (Participants) | 182 | 196
  Trouble Talking C3D1 | -0.18 (11.35) | -1.02 (11.65)
  Trouble Talking C4D1: number analyzed (Participants) | 166 | 169
  Trouble Talking C4D1 | -0.40 (12.71) | 0.99 (14.28)
  Trouble Talking C5D1: number analyzed (Participants) | 159 | 165
  Trouble Talking C5D1 | 1.68 (11.74) | -0.81 (11.01)
  Trouble Talking C6D1: number analyzed (Participants) | 149 | 145
  Trouble Talking C6D1 | 0.67 (13.68) | 0.46 (11.78)
  Trouble Talking C7D1: number analyzed (Participants) | 119 | 125
  Trouble Talking C7D1 | 0.84 (15.32) | -0.53 (11.19)
  Trouble Talking C8D1: number analyzed (Participants) | 108 | 109
  Trouble Talking C8D1 | 0.93 (12.45) | -1.22 (13.55)
  Trouble Talking C9D1: number analyzed (Participants) | 102 | 103
  Trouble Talking C9D1 | 0.65 (15.54) | 0.32 (13.60)
  Trouble Talking C10D1: number analyzed (Participants) | 85 | 79
  Trouble Talking C10D1 | 0.39 (14.08) | -1.27 (15.51)
  Trouble Talking C11D1: number analyzed (Participants) | 80 | 71
  Trouble Talking C11D1 | 0.42 (12.43) | -1.41 (13.14)
  Trouble Talking C12D1: number analyzed (Participants) | 75 | 57
  Trouble Talking C12D1 | -1.33 (11.55) | 0.58 (7.69)
  Trouble Talking C13D1: number analyzed (Participants) | 60 | 48
  Trouble Talking C13D1 | -2.78 (12.71) | -1.39 (15.31)
  Trouble Talking C14D1: number analyzed (Participants) | 55 | 44
  Trouble Talking C14D1 | -3.03 (11.61) | 0.00 (16.07)
  Trouble Talking C15D1: number analyzed (Participants) | 51 | 36
  Trouble Talking C15D1 | -3.27 (13.75) | -1.85 (13.67)
  Trouble Talking C16D1: number analyzed (Participants) | 48 | 31
  Trouble Talking C16D1 | 0.00 (16.84) | -1.08 (16.06)
  Trouble Talking C17D1: number analyzed (Participants) | 43 | 25
  Trouble Talking C17D1 | -4.65 (13.77) | 2.67 (13.33)
  Trouble Talking C18D1: number analyzed (Participants) | 41 | 21
  Trouble Talking C18D1 | -3.25 (12.48) | 3.17 (14.55)
  Trouble Talking C19D1: number analyzed (Participants) | 40 | 20
  Trouble Talking C19D1 | 0.00 (15.10) | 1.67 (7.45)
  Trouble Talking C20D1: number analyzed (Participants) | 39 | 19
  Trouble Talking C20D1 | -2.56 (14.07) | 1.75 (13.49)
  Trouble Talking C21D1: number analyzed (Participants) | 36 | 20
  Trouble Talking C21D1 | -0.93 (18.66) | 3.33 (18.42)
  Trouble Talking C22D1: number analyzed (Participants) | 31 | 17
  Trouble Talking C22D1 | -3.23 (13.21) | 0.00 (20.41)
  Trouble Talking C23D1: number analyzed (Participants) | 31 | 16
  Trouble Talking C23D1 | -1.08 (13.56) | -2.08 (19.12)
  Trouble Talking C24D1: number analyzed (Participants) | 29 | 12
  Trouble Talking C24D1 | -2.30 (12.38) | 0.00 (24.62)
  Trouble Talking C25D1: number analyzed (Participants) | 28 | 12
  Trouble Talking C25D1 | -1.19 (14.29) | 2.78 (17.16)
  Trouble Talking C26D1: number analyzed (Participants) | 26 | 9
  Trouble Talking C26D1 | -1.28 (14.85) | 3.70 (11.11)
  Trouble Talking C27D1: number analyzed (Participants) | 25 | 10
  Trouble Talking C27D1 | -2.67 (13.33) | 3.33 (10.54)
  Trouble Talking C28D1: number analyzed (Participants) | 21 | 11
  Trouble Talking C28D1 | -3.17 (14.55) | 3.03 (10.05)
  Trouble Talking C29D1: number analyzed (Participants) | 22 | 12
  Trouble Talking C29D1 | -1.52 (16.19) | 2.78 (9.62)
  Trouble Talking C30D1: number analyzed (Participants) | 20 | 0
  Trouble Talking C30D1 | -1.67 (17.01) |
  Trouble Talking C31D1: number analyzed (Participants) | 20 | 0
  Trouble Talking C31D1 | 0.00 (18.73) |
  Trouble Talking C32D1: number analyzed (Participants) | 18 | 0
  Trouble Talking C32D1 | -1.85 (17.98) |
  Trouble Talking C33D1: number analyzed (Participants) | 15 | 0
  Trouble Talking C33D1 | -4.44 (17.21) |
  Trouble Talking C34D1: number analyzed (Participants) | 12 | 0
  Trouble Talking C34D1 | -5.56 (19.25) |
  Trouble Talking C35D1: number analyzed (Participants) | 13 | 0
  Trouble Talking C35D1 | -5.13 (18.49) |
  Trouble Talking C36D1: number analyzed (Participants) | 12 | 0
  Trouble Talking C36D1 | -5.56 (19.25) |
  Trouble Talking C37D1: number analyzed (Participants) | 11 | 0
  Trouble Talking C37D1 | -6.06 (20.10) |
  Trouble Talking C38D1: number analyzed (Participants) | 10 | 0
  Trouble Talking C38D1 | -6.67 (21.08) |
  Trouble Talking C39D1: number analyzed (Participants) | 9 | 0
  Trouble Talking C39D1 | 0.00 (0.00) |
  Trouble Talking 30 day follow up: number analyzed (Participants) | 57 | 76
  Trouble Talking 30 day follow up | 4.68 (18.30) | 2.19 (15.72)
  Trouble Talking 90 day follow up: number analyzed (Participants) | 61 | 79
  Trouble Talking 90 day follow up | 3.83 (10.71) | 3.38 (20.39)
  Weight Loss Baseline | 23.05 (27.43) | 24.07 (28.25)
  Weight Loss C2D1: number analyzed (Participants) | 208 | 216
  Weight Loss C2D1 | 0.16 (23.28) | 0.46 (26.99)
  Weight Loss C3D1: number analyzed (Participants) | 182 | 196
  Weight Loss C3D1 | 0.92 (26.78) | 1.02 (27.20)
  Weight Loss C4D1: number analyzed (Participants) | 166 | 169
  Weight Loss C4D1 | 0.00 (28.19) | -1.18 (25.69)
  Weight Loss C5D1: number analyzed (Participants) | 159 | 165
  Weight Loss C5D1 | 2.52 (32.38) | -2.42 (26.43)
  Weight Loss C6D1: number analyzed (Participants) | 149 | 145
  Weight Loss C6D1 | -0.45 (25.99) | -5.29 (29.05)
  Weight Loss C7D1: number analyzed (Participants) | 119 | 125
  Weight Loss C7D1 | -2.52 (27.84) | -3.47 (28.02)
  Weight Loss C8D1: number analyzed (Participants) | 108 | 109
  Weight Loss C8D1 | -2.47 (26.46) | -3.67 (29.17)
  Weight Loss C9D1: number analyzed (Participants) | 102 | 103
  Weight Loss C9D1 | -5.88 (29.45) | -7.12 (29.76)
  Weight Loss C10D1: number analyzed (Participants) | 85 | 79
  Weight Loss C10D1 | -7.06 (32.57) | -5.91 (28.12)
  Weight Loss C11D1: number analyzed (Participants) | 80 | 71
  Weight Loss C11D1 | -9.58 (30.56) | -8.45 (25.65)
  Weight Loss C12D1: number analyzed (Participants) | 75 | 57
  Weight Loss C12D1 | -10.22 (30.50) | -10.53 (24.53)
  Weight Loss C13D1: number analyzed (Participants) | 60 | 48
  Weight Loss C13D1 | -11.67 (28.67) | -10.42 (25.87)
  Weight Loss C14D1: number analyzed (Participants) | 55 | 44
  Weight Loss C14D1 | -13.94 (26.21) | -6.82 (23.38)
  Weight Loss C15D1: number analyzed (Participants) | 51 | 36
  Weight Loss C15D1 | -12.42 (26.63) | -8.33 (30.21)
  Weight Loss C16D1: number analyzed (Participants) | 48 | 31
  Weight Loss C16D1 | -15.97 (22.79) | -8.60 (22.72)
  Weight Loss C17D1: number analyzed (Participants) | 43 | 25
  Weight Loss C17D1 | -14.73 (19.66) | -13.33 (21.52)
  Weight Loss C18D1: number analyzed (Participants) | 41 | 21
  Weight Loss C18D1 | -11.38 (25.40) | -14.29 (27.02)
  Weight Loss C19D1: number analyzed (Participants) | 40 | 20
  Weight Loss C19D1 | -16.67 (22.65) | -11.67 (16.31)
  Weight Loss C20D1: number analyzed (Participants) | 39 | 19
  Weight Loss C20D1 | -10.26 (21.84) | -12.28 (25.36)
  Weight Loss C21D1: number analyzed (Participants) | 36 | 20
  Weight Loss C21D1 | -12.96 (22.93) | -16.67 (25.36)
  Weight Loss C22D1: number analyzed (Participants) | 31 | 17
  Weight Loss C22D1 | -12.90 (23.85) | -17.65 (26.66)
  Weight Loss C23D1: number analyzed (Participants) | 31 | 16
  Weight Loss C23D1 | -10.75 (19.98) | -22.92 (29.11)
  Weight Loss C24D1: number analyzed (Participants) | 29 | 12
  Weight Loss C24D1 | -10.34 (26.88) | -13.89 (30.01)
  Weight Loss C25D1: number analyzed (Participants) | 28 | 12
  Weight Loss C25D1 | -10.71 (20.39) | -11.11 (25.95)
  Weight Loss C26D1: number analyzed (Participants) | 26 | 9
  Weight Loss C26D1 | -16.67 (25.39) | -11.11 (16.67)
  Weight Loss C27D1: number analyzed (Participants) | 25 | 10
  Weight Loss C27D1 | -12.00 (21.26) | -13.33 (23.31)
  Weight Loss C28D1: number analyzed (Participants) | 21 | 11
  Weight Loss C28D1 | -14.29 (22.54) | -6.06 (13.48)
  Weight Loss C29D1: number analyzed (Participants) | 22 | 12
  Weight Loss C29D1 | -13.64 (19.68) | -8.33 (15.08)
  Weight Loss C30D1: number analyzed (Participants) | 20 | 0
  Weight Loss C30D1 | -15.00 (20.16) |
  Weight Loss C31D1: number analyzed (Participants) | 20 | 0
  Weight Loss C31D1 | -11.67 (19.57) |
  Weight Loss C32D1: number analyzed (Participants) | 18 | 0
  Weight Loss C32D1 | -20.37 (20.26) |
  Weight Loss C33D1: number analyzed (Participants) | 15 | 0
  Weight Loss C33D1 | -15.56 (24.77) |
  Weight Loss C34D1: number analyzed (Participants) | 12 | 0
  Weight Loss C34D1 | -16.67 (26.59) |
  Weight Loss C35D1: number analyzed (Participants) | 13 | 0
  Weight Loss C35D1 | -15.38 (22.01) |
  Weight Loss C36D1: number analyzed (Participants) | 12 | 0
  Weight Loss C36D1 | -13.89 (22.29) |
  Weight Loss C37D1: number analyzed (Participants) | 11 | 0
  Weight Loss C37D1 | -18.18 (27.34) |
  Weight Loss C38D1: number analyzed (Participants) | 10 | 0
  Weight Loss C38D1 | -20.00 (23.31) |
  Weight Loss C39D1: number analyzed (Participants) | 9 | 0
  Weight Loss C39D1 | -14.81 (24.22) |
  Weight Loss 30 day follow up: number analyzed (Participants) | 57 | 76
  Weight Loss 30 day follow up | -1.75 (30.49) | 3.95 (27.74)
  Weight Loss 90 day follow up: number analyzed (Participants) | 61 | 79
  Weight Loss 90 day follow up | -1.64 (24.67) | 2.95 (30.75)
  Hair Loss Baseline | 12.09 (20.80) | 12.55 (23.56)
  Hair Loss C2D1: number analyzed (Participants) | 59 | 60
  Hair Loss C2D1 | -2.26 (18.43) | -1.67 (15.56)
  Hair Loss C3D1: number analyzed (Participants) | 54 | 49
  Hair Loss C3D1 | -3.09 (19.71) | -4.76 (23.57)
  Hair Loss C4D1: number analyzed (Participants) | 53 | 46
  Hair Loss C4D1 | -0.63 (24.01) | 0.00 (15.71)
  Hair Loss C5D1: number analyzed (Participants) | 44 | 41
  Hair Loss C5D1 | -3.03 (20.10) | -0.81 (18.99)
  Hair Loss C6D1: number analyzed (Participants) | 45 | 36
  Hair Loss C6D1 | 2.96 (23.38) | -4.63 (21.31)
  Hair Loss C7D1: number analyzed (Participants) | 30 | 29
  Hair Loss C7D1 | -3.33 (22.06) | -4.60 (17.19)
  Hair Loss C8D1: number analyzed (Participants) | 35 | 26
  Hair Loss C8D1 | -5.71 (27.40) | -8.97 (20.13)
  Hair Loss C9D1: number analyzed (Participants) | 30 | 21
  Hair Loss C9D1 | -2.22 (26.16) | -9.52 (26.13)
  Hair Loss C10D1: number analyzed (Participants) | 20 | 16
  Hair Loss C10D1 | -1.67 (25.31) | -8.33 (28.54)
  Hair Loss C11D1: number analyzed (Participants) | 20 | 11
  Hair Loss C11D1 | -1.67 (27.52) | 3.03 (17.98)
  Hair Loss C12D1: number analyzed (Participants) | 22 | 12
  Hair Loss C12D1 | -4.55 (25.81) | 0.00 (20.10)
  Hair Loss C13D1: number analyzed (Participants) | 19 | 10
  Hair Loss C13D1 | -5.26 (29.94) | -6.67 (21.08)
  Hair Loss C14D1: number analyzed (Participants) | 12 | 7
  Hair Loss C14D1 | -11.11 (29.59) | 4.76 (12.60)
  Hair Loss C15D1: number analyzed (Participants) | 11 | 7
  Hair Loss C15D1 | 6.06 (25.03) | -4.76 (12.60)
  Hair Loss C16D1: number analyzed (Participants) | 13 | 5
  Hair Loss C16D1 | -2.56 (16.45) | -6.67 (14.91)
  Hair Loss C17D1: number analyzed (Participants) | 11 | 4
  Hair Loss C17D1 | 0.00 (21.08) | 0.00 (0.00)
  Hair Loss C18D1: number analyzed (Participants) | 10 | 0
  Hair Loss C18D1 | 0.00 (22.22) |
  Hair Loss C19D1: number analyzed (Participants) | 8 | 5
  Hair Loss C19D1 | 0.00 (17.82) | -13.33 (18.26)
  Hair Loss C20D1: number analyzed (Participants) | 10 | 4
  Hair Loss C20D1 | -3.33 (18.92) | 0.00 (0.00)
  Hair Loss C21D1: number analyzed (Participants) | 10 | 0
  Hair Loss C21D1 | -3.33 (18.92) |
  Hair Loss C22D1: number analyzed (Participants) | 8 | 0
  Hair Loss C22D1 | 0.00 (17.82) |
  Hair Loss C23D1: number analyzed (Participants) | 6 | 0
  Hair Loss C23D1 | 0.00 (21.08) |
  Hair Loss C24D1: number analyzed (Participants) | 7 | 0
  Hair Loss C24D1 | -4.76 (23.00) |
  Hair Loss C25D1: number analyzed (Participants) | 6 | 0
  Hair Loss C25D1 | 0.00 (21.08) |
  Hair Loss C26D1: number analyzed (Participants) | 0 | 0
  Hair Loss C27D1: number analyzed (Participants) | 0 | 0
  Hair Loss C28D1: number analyzed (Participants) | 0 | 0
  Hair Loss C29D1: number analyzed (Participants) | 0 | 0
  Hair Loss C30D1: number analyzed (Participants) | 0 | 0
  Hair Loss C31D1: number analyzed (Participants) | 0 | 0
  Hair Loss C32D1: number analyzed (Participants) | 0 | 0
  Hair Loss C33D1: number analyzed (Participants) | 0 | 0
  Hair Loss C34D1: number analyzed (Participants) | 0 | 0
  Hair Loss C35D1: number analyzed (Participants) | 0 | 0
  Hair Loss C36D1: number analyzed (Participants) | 0 | 0
  Hair Loss C37D1: number analyzed (Participants) | 0 | 0
  Hair Loss C38D1: number analyzed (Participants) | 0 | 0
  Hair Loss C39D1: number analyzed (Participants) | 0 | 0
  Hair Loss 30 day follow up: number analyzed (Participants) | 8 | 14
  Hair Loss 30 day follow up | 8.33 (23.57) | 2.38 (30.56)
  Hair Loss 90 day follow up: number analyzed (Participants) | 17 | 22
  Hair Loss 90 day follow up | 23.53 (40.42) | 15.15 (26.68)
  Belching Baseline | 12.14 (18.62) | 14.11 (21.01)
  Belching C2D1: number analyzed (Participants) | 208 | 216
  Belching C2D1 | -1.52 (15.68) | -3.09 (14.93)
  Belching C3D1: number analyzed (Participants) | 182 | 196
  Belching C3D1 | 0.92 (17.84) | -1.87 (16.94)
  Belching C4D1: number analyzed (Participants) | 166 | 169
  Belching C4D1 | 0.20 (16.51) | -3.16 (18.81)
  Belching C5D1: number analyzed (Participants) | 159 | 165
  Belching C5D1 | 1.68 (17.81) | -5.35 (18.59)
  Belching C6D1: number analyzed (Participants) | 149 | 145
  Belching C6D1 | 0.00 (16.67) | -4.02 (20.53)
  Belching C7D1: number analyzed (Participants) | 119 | 125
  Belching C7D1 | 0.28 (17.36) | -5.07 (20.66)
  Belching C8D1: number analyzed (Participants) | 108 | 109
  Belching C8D1 | 1.54 (20.95) | -5.05 (21.46)
  Belching C9D1: number analyzed (Participants) | 102 | 103
  Belching C9D1 | 1.31 (18.27) | -9.39 (20.44)
  Belching C10D1: number analyzed (Participants) | 85 | 79
  Belching C10D1 | 0.39 (18.54) | -7.38 (19.93)
  Belching C11D1: number analyzed (Participants) | 80 | 71
  Belching C11D1 | -2.08 (17.26) | -9.62 (21.21)
  Belching C12D1: number analyzed (Participants) | 75 | 57
  Belching C12D1 | -1.78 (16.11) | -7.60 (18.65)
  Belching C13D1: number analyzed (Participants) | 60 | 48
  Belching C13D1 | -0.28 (20.00) | -7.64 (22.27)
  Belching C14D1: number analyzed (Participants) | 55 | 44
  Belching C14D1 | 0.00 (17.27) | -6.06 (20.99)
  Belching C15D1: number analyzed (Participants) | 51 | 36
  Belching C15D1 | -1.31 (16.61) | -5.56 (19.92)
  Belching C16D1: number analyzed (Participants) | 48 | 31
  Belching C16D1 | -2.78 (18.30) | -5.91 (22.17)
  Belching C17D1: number analyzed (Participants) | 43 | 25
  Belching C17D1 | -2.71 (18.87) | -5.33 (22.42)
  Belching C18D1: number analyzed (Participants) | 41 | 21
  Belching C18D1 | -2.03 (17.16) | -3.17 (27.19)
  Belching C19D1: number analyzed (Participants) | 40 | 20
  Belching C19D1 | 0.42 (15.33) | -2.50 (11.18)
  Belching C20D1: number analyzed (Participants) | 39 | 19
  Belching C20D1 | 1.28 (18.09) | -7.02 (21.74)
  Belching C21D1: number analyzed (Participants) | 36 | 20
  Belching C21D1 | -0.93 (14.33) | -5.00 (23.63)
  Belching C22D1: number analyzed (Participants) | 31 | 17
  Belching C22D1 | -0.54 (17.99) | -4.90 (28.73)
  Belching C23D1: number analyzed (Participants) | 31 | 16
  Belching C23D1 | -3.23 (16.34) | -9.38 (23.55)
  Belching C24D1: number analyzed (Participants) | 29 | 12
  Belching C24D1 | 0.00 (16.67) | -5.56 (32.05)
  Belching C25D1: number analyzed (Participants) | 28 | 12
  Belching C25D1 | 0.60 (17.26) | -8.33 (31.38)
  Belching C26D1: number analyzed (Participants) | 26 | 9
  Belching C26D1 | 1.92 (17.21) | 3.70 (20.03)
  Belching C27D1: number analyzed (Participants) | 25 | 10
  Belching C27D1 | 0.00 (15.21) | 0.00 (13.61)
  Belching C28D1: number analyzed (Participants) | 21 | 11
  Belching C28D1 | 3.97 (13.85) | 1.52 (13.85)
  Belching C29D1: number analyzed (Participants) | 22 | 12
  Belching C29D1 | 0.00 (15.43) | -1.39 (11.14)
  Belching C30D1: number analyzed (Participants) | 20 | 0
  Belching C30D1 | 0.83 (14.78) |
  Belching C31D1: number analyzed (Participants) | 20 | 0
  Belching C31D1 | 2.50 (16.47) |
  Belching C32D1: number analyzed (Participants) | 18 | 0
  Belching C32D1 | 4.63 (17.90) |
  Belching C33D1: number analyzed (Participants) | 15 | 0
  Belching C33D1 | -1.11 (14.73) |
  Belching C34D1: number analyzed (Participants) | 12 | 0
  Belching C34D1 | 0.00 (12.31) |
  Belching C35D1: number analyzed (Participants) | 13 | 0
  Belching C35D1 | 3.85 (20.59) |
  Belching C36D1: number analyzed (Participants) | 12 | 0
  Belching C36D1 | 1.39 (19.41) |
  Belching C37D1: number analyzed (Participants) | 11 | 0
  Belching C37D1 | 6.06 (11.24) |
  Belching C38D1: number analyzed (Participants) | 10 | 0
  Belching C38D1 | 1.67 (16.57) |
  Belching C39D1: number analyzed (Participants) | 9 | 0
  Belching C39D1 | 3.70 (7.35) |
  Belching 30 day follow up: number analyzed (Participants) | 57 | 76
  Belching 30 day follow up | 3.22 (21.23) | 0.66 (19.52)
  Belching 90 day follow up: number analyzed (Participants) | 61 | 79
  Belching 90 day follow up | -0.55 (15.20) | -1.90 (17.50)

12. Secondary Outcome: Change From Baseline in HRQoL Measured by Global Pain (GP)
Description: The GP instrument is a single assessment of overall pain and participants were assessed in global pain according to the following response categories: 1= no pain (anymore), 2 = less pain, 3 = no change and 4 = more pain. Low pain scores are considered a better outcome than a high pain score.
Time Frame: Baseline, on D1 from C2 through C39, 30-day follow up, 90-day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 243 | 236
Unit on a scale
  Baseline | 2.45 (2.49) | 2.64 (2.55)
  C2D1: number analyzed (Participants) | 208 | 211
  C2D1 | -0.60 (2.61) | -0.63 (2.59)
  C3D1: number analyzed (Participants) | 180 | 190
  C3D1 | -0.74 (2.30) | -0.82 (2.33)
  C4D1: number analyzed (Participants) | 166 | 167
  C4D1 | -0.63 (2.58) | -0.91 (2.68)
  C5D1: number analyzed (Participants) | 159 | 164
  C5D1 | -0.37 (2.89) | -0.79 (2.84)
  C6D1: number analyzed (Participants) | 149 | 143
  C6D1 | -0.51 (2.61) | -0.57 (3.00)
  C7D1: number analyzed (Participants) | 117 | 122
  C7D1 | -0.61 (2.65) | -0.38 (2.74)
  C8D1: number analyzed (Participants) | 106 | 109
  C8D1 | -0.59 (2.45) | -0.36 (2.48)
  C9D1: number analyzed (Participants) | 102 | 103
  C9D1 | -0.65 (2.62) | -0.36 (2.63)
  C10D1: number analyzed (Participants) | 85 | 78
  C10D1 | -0.71 (2.67) | -0.71 (2.65)
  C11D1: number analyzed (Participants) | 80 | 70
  C11D1 | -0.40 (2.96) | -0.61 (2.55)
  C12D1: number analyzed (Participants) | 75 | 57
  C12D1 | 0.08 (2.91) | -0.53 (2.41)
  C13D1: number analyzed (Participants) | 60 | 48
  C13D1 | 0.05 (3.40) | -0.63 (2.44)
  C14D1: number analyzed (Participants) | 55 | 44
  C14D1 | -0.95 (2.63) | -0.34 (2.12)
  C15D1: number analyzed (Participants) | 51 | 36
  C15D1 | -0.80 (2.62) | -0.44 (1.81)
  C16D1: number analyzed (Participants) | 48 | 31
  C16D1 | -0.19 (3.07) | 0.10 (2.23)
  C17D1: number analyzed (Participants) | 43 | 25
  C17D1 | -0.74 (2.46) | -0.20 (1.32)
  C18D1: number analyzed (Participants) | 41 | 21
  C18D1 | 0.17 (3.26) | -0.48 (1.29)
  C19D1: number analyzed (Participants) | 40 | 20
  C19D1 | -0.20 (2.53) | -0.25 (0.97)
  C20D1: number analyzed (Participants) | 39 | 19
  C20D1 | 0.05 (2.72) | 0.21 (2.90)
  C21D1: number analyzed (Participants) | 36 | 20
  C21D1 | -0.06 (2.86) | 0.50 (2.96)
  C22D1: number analyzed (Participants) | 31 | 17
  C22D1 | 0.00 (2.89) | 0.00 (2.92)
  C23D1: number analyzed (Participants) | 31 | 16
  C23D1 | -0.19 (2.17) | 0.69 (3.22)
  C24D1: number analyzed (Participants) | 29 | 12
  C24D1 | -0.45 (3.41) | -0.33 (1.72)
  C25D1: number analyzed (Participants) | 28 | 12
  C25D1 | -0.86 (2.17) | 0.17 (3.21)
  C26D1: number analyzed (Participants) | 26 | 9
  C26D1 | -0.58 (2.53) | 0.22 (1.86)
  C27D1: number analyzed (Participants) | 25 | 10
  C27D1 | -1.08 (2.25) | 0.80 (3.29)
  C28D1: number analyzed (Participants) | 21 | 11
  C28D1 | 0.05 (2.89) | 0.18 (1.33)
  C29D1: number analyzed (Participants) | 22 | 12
  C29D1 | -0.14 (2.25) | -0.17 (0.72)
  C30D1: number analyzed (Participants) | 20 | 0
  C30D1 | -0.45 (2.11) |
  C31D1: number analyzed (Participants) | 20 | 0
  C31D1 | -0.45 (2.24) |
  C32D1: number analyzed (Participants) | 18 | 0
  C32D1 | -0.50 (2.71) |
  C33D1: number analyzed (Participants) | 15 | 0
  C33D1 | 0.07 (3.24) |
  C34D1: number analyzed (Participants) | 12 | 0
  C34D1 | -0.67 (3.20) |
  C35D1: number analyzed (Participants) | 13 | 0
  C35D1 | -0.69 (2.84) |
  C36D1: number analyzed (Participants) | 12 | 0
  C36D1 | -1.42 (1.56) |
  C37D1: number analyzed (Participants) | 11 | 0
  C37D1 | 0.18 (3.06) |
  C38D1: number analyzed (Participants) | 10 | 0
  C38D1 | 0.00 (3.53) |
  C39D1: number analyzed (Participants) | 9 | 0
  C39D1 | -0.89 (1.27) |
  30 day follow up: number analyzed (Participants) | 57 | 73
  30 day follow up | 0.74 (3.34) | 0.56 (2.63)
  90 day follow up: number analyzed (Participants) | 61 | 77
  90 day follow up | 0.08 (3.34) | 0.62 (2.81)

13. Secondary Outcome: Change From Baseline in HRQoL Measured by the EuroQOL Five Dimensions Questionnaire 5L (EQ-5D-5L) Questionnaire
Description: EQ-5D-5L is a standardized instrument for use as a measure of health outcomes consisting of 6 items that cover 5 main domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a general visual analog scale for health status. It was developed by the EuroQol Group for use as a generic, preference-based measure of health outcomes. Each dimension comprises 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). A unique EQ-5D-5L health state is defined by combining 1 level from each of the 5 dimensions. This questionnaire also records the respondent's self-rated health status on a vertical graduated (0 = the worst health a participant can imagine to 100 = the best health a participant can imagine) visual analogue scale. Responses to the 5 items will also be converted to a weighted health state index (utility score) based on values derived from general population samples.
Time Frame: Baseline, on D1 from C2 through C39, 30-day follow up, 90-day follow up
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | CAPOX+ Zolbetuximab | CAPOX+ Placebo
Number analyzed (Participants) | 243 | 243
Unit on a scale
  Mobility Baseline | 1.33 (0.67) | 1.33 (0.67)
  Mobility C2D1: number analyzed (Participants) | 208 | 218
  Mobility C2D1 | 0.02 (0.60) | 0.06 (0.67)
  Mobility C3D1: number analyzed (Participants) | 183 | 198
  Mobility C3D1 | -0.01 (0.61) | 0.05 (0.65)
  Mobility C4D1: number analyzed (Participants) | 169 | 171
  Mobility C4D1 | -0.01 (0.62) | 0.02 (0.76)
  Mobility C5D1: number analyzed (Participants) | 159 | 167
  Mobility C5D1 | 0.05 (0.65) | 0.00 (0.78)
  Mobility C6D1: number analyzed (Participants) | 149 | 147
  Mobility C6D1 | 0.04 (0.77) | 0.03 (0.86)
  Mobility C7D1: number analyzed (Participants) | 121 | 127
  Mobility C7D1 | 0.02 (0.72) | 0.02 (0.70)
  Mobility C8D1: number analyzed (Participants) | 109 | 111
  Mobility C8D1 | 0.20 (0.81) | 0.05 (0.78)
  Mobility C9D1: number analyzed (Participants) | 102 | 104
  Mobility C9D1 | 0.18 (0.78) | 0.06 (0.75)
  Mobility C10D1: number analyzed (Participants) | 85 | 80
  Mobility C10D1 | 0.08 (0.74) | 0.13 (0.74)
  Mobility C11D1: number analyzed (Participants) | 81 | 72
  Mobility C11D1 | 0.12 (0.68) | 0.15 (0.87)
  Mobility C12D1: number analyzed (Participants) | 75 | 58
  Mobility C12D1 | 0.08 (0.65) | 0.02 (0.66)
  Mobility C13D1: number analyzed (Participants) | 60 | 49
  Mobility C13D1 | 0.08 (0.74) | 0.10 (0.85)
  Mobility C14D1: number analyzed (Participants) | 56 | 45
  Mobility C14D1 | -0.05 (0.64) | 0.11 (0.53)
  Mobility C15D1: number analyzed (Participants) | 51 | 37
  Mobility C15D1 | -0.04 (0.69) | 0.03 (0.55)
  Mobility C16D1: number analyzed (Participants) | 48 | 32
  Mobility C16D1 | 0.02 (0.64) | 0.06 (0.56)
  Mobility C17D1: number analyzed (Participants) | 43 | 26
  Mobility C17D1 | 0.00 (0.72) | 0.08 (0.48)
  Mobility C18D1: number analyzed (Participants) | 41 | 22
  Mobility C18D1 | 0.07 (0.52) | 0.09 (0.43)
  Mobility C19D1: number analyzed (Participants) | 40 | 21
  Mobility C19D1 | 0.03 (0.53) | 0.00 (0.32)
  Mobility C20D1: number analyzed (Participants) | 39 | 20
  Mobility C20D1 | 0.10 (0.55) | 0.10 (0.55)
  Mobility C21D1: number analyzed (Participants) | 36 | 21
  Mobility C21D1 | 0.03 (0.51) | -0.14 (0.48)
  Mobility C22D1: number analyzed (Participants) | 31 | 18
  Mobility C22D1 | 0.03 (0.55) | -0.11 (0.58)
  Mobility C23D1: number analyzed (Participants) | 31 | 17
  Mobility C23D1 | 0.00 (0.58) | -0.12 (0.60)
  Mobility C24D1: number analyzed (Participants) | 29 | 13
  Mobility C24D1 | 0.07 (0.53) | -0.15 (0.69)
  Mobility C25D1: number analyzed (Participants) | 28 | 13
  Mobility C25D1 | 0.21 (0.63) | -0.08 (0.76)
  Mobility C26D1: number analyzed (Participants) | 26 | 10
  Mobility C26D1 | 0.15 (0.54) | 0.10 (0.32)
  Mobility C27D1: number analyzed (Participants) | 25 | 11
  Mobility C27D1 | 0.08 (0.76) | -0.09 (0.30)
  Mobility C28D1: number analyzed (Participants) | 21 | 11
  Mobility C28D1 | 0.24 (0.89) | 0.09 (0.30)
  Mobility C29D1: number analyzed (Participants) | 22 | 12
  Mobility C29D1 | 0.05 (0.65) | -0.08 (0.51)
  Mobility C30D1: number analyzed (Participants) | 20 | 0
  Mobility C30D1 | 0.10 (0.64) |
  Mobility C31D1: number analyzed (Participants) | 20 | 0
  Mobility C31D1 | 0.00 (0.56) |
  Mobility C32D1: number analyzed (Participants) | 18 | 0
  Mobility C32D1 | 0.06 (0.54) |
  Mobility C33D1: number analyzed (Participants) | 15 | 0
  Mobility C33D1 | 0.00 (0.76) |
  Mobility C34D1: number analyzed (Participants) | 12 | 0
  Mobility C34D1 | -0.08 (0.79) |
  Mobility C35D1: number analyzed (Participants) | 13 | 0
  Mobility C35D1 | -0.08 (0.76) |
  Mobility C36D1: number analyzed (Participants) | 12 | 0
  Mobility C36D1 | -0.08 (0.51) |
  Mobility C37D1: number analyzed (Participants) | 11 | 0
  Mobility C37D1 | 0.00 (0.63) |
  Mobility C38D1: number analyzed (Participants) | 10 | 0
  Mobility C38D1 | 0.00 (0.67) |
  Mobility C39D1: number analyzed (Participants) | 9 | 0
  Mobility C39D1 | 0.22 (0.83) |
  Mobility 30 day follow up: number analyzed (Participants) | 58 | 78
  Mobility 30 day follow up | 0.47 (0.96) | 0.36 (0.98)
  Mobility 90 day follow up: number analyzed (Participants) | 63 | 80
  Mobility 90 day follow up | 0.32 (0.76) | 0.43 (0.90)
  Self-Care Baseline | 1.12 (0.39) | 1.18 (0.56)
  Self-Care C2D1: number analyzed (Participants) | 208 | 218
  Self-Care C2D1 | 0.05 (0.48) | 0.07 (0.67)
  Self-Care C3D1: number analyzed (Participants) | 183 | 198
  Self-Care C3D1 | 0.02 (0.44) | 0.03 (0.60)
  Self-Care C4D1: number analyzed (Participants) | 169 | 171
  Self-Care C4D1 | 0.05 (0.46) | 0.02 (0.64)
  Self-Care C5D1: number analyzed (Participants) | 159 | 167
  Self-Care C5D1 | 0.05 (0.55) | 0.07 (0.72)
  Self-Care C6D1: number analyzed (Participants) | 149 | 147
  Self-Care C6D1 | 0.05 (0.51) | 0.09 (0.63)
  Self-Care C7D1: number analyzed (Participants) | 121 | 127
  Self-Care C7D1 | 0.07 (0.60) | 0.02 (0.70)
  Self-Care C8D1: number analyzed (Participants) | 109 | 111
  Self-Care C8D1 | 0.10 (0.64) | 0.05 (0.62)
  Self-Care C9D1: number analyzed (Participants) | 102 | 104
  Self-Care C9D1 | 0.15 (0.79) | 0.10 (0.58)
  Self-Care C10D1: number analyzed (Participants) | 85 | 80
  Self-Care C10D1 | 0.11 (0.66) | 0.10 (0.65)
  Self-Care C11D1: number analyzed (Participants) | 81 | 72
  Self-Care C11D1 | 0.09 (0.64) | 0.06 (0.69)
  Self-Care C12D1: number analyzed (Participants) | 75 | 58
  Self-Care C12D1 | 0.09 (0.64) | 0.10 (0.55)
  Self-Care C13D1: number analyzed (Participants) | 60 | 49
  Self-Care C13D1 | 0.05 (0.62) | 0.12 (0.56)
  Self-Care C14D1: number analyzed (Participants) | 56 | 45
  Self-Care C14D1 | 0.04 (0.50) | 0.11 (0.61)
  Self-Care C15D1: number analyzed (Participants) | 51 | 37
  Self-Care C15D1 | 0.00 (0.49) | 0.05 (0.52)
  Self-Care C16D1: number analyzed (Participants) | 48 | 32
  Self-Care C16D1 | 0.00 (0.62) | 0.09 (0.59)
  Self-Care C17D1: number analyzed (Participants) | 43 | 26
  Self-Care C17D1 | 0.02 (0.64) | 0.04 (0.53)
  Self-Care C18D1: number analyzed (Participants) | 41 | 22
  Self-Care C18D1 | 0.10 (0.49) | -0.05 (0.49)
  Self-Care C19D1: number analyzed (Participants) | 40 | 21
  Self-Care C19D1 | 0.00 (0.32) | -0.10 (0.44)
  Self-Care C20D1: number analyzed (Participants) | 39 | 20
  Self-Care C20D1 | 0.00 (0.32) | 0.05 (0.60)
  Self-Care C21D1: number analyzed (Participants) | 36 | 21
  Self-Care C21D1 | 0.03 (0.38) | -0.10 (0.44)
  Self-Care C22D1: number analyzed (Participants) | 31 | 18
  Self-Care C22D1 | 0.00 (0.37) | 0.00 (0.59)
  Self-Care C23D1: number analyzed (Participants) | 31 | 17
  Self-Care C23D1 | 0.06 (0.36) | -0.12 (0.49)
  Self-Care C24D1: number analyzed (Participants) | 29 | 13
  Self-Care C24D1 | 0.07 (0.26) | -0.08 (0.64)
  Self-Care C25D1: number analyzed (Participants) | 28 | 13
  Self-Care C25D1 | 0.11 (0.31) | -0.08 (0.64)
  Self-Care C26D1: number analyzed (Participants) | 26 | 10
  Self-Care C26D1 | 0.12 (0.33) | -0.20 (0.63)
  Self-Care C27D1: number analyzed (Participants) | 25 | 11
  Self-Care C27D1 | 0.08 (0.28) | -0.18 (0.60)
  Self-Care C28D1: number analyzed (Participants) | 21 | 11
  Self-Care C28D1 | 0.10 (0.44) | -0.18 (0.60)
  Self-Care C29D1: number analyzed (Participants) | 22 | 12
  Self-Care C29D1 | 0.14 (0.47) | -0.17 (0.58)
  Self-Care C30D1: number analyzed (Participants) | 20 | 0
  Self-Care C30D1 | 0.10 (0.45) |
  Self-Care C31D1: number analyzed (Participants) | 20 | 0
  Self-Care C31D1 | 0.10 (0.45) |
  Self-Care C32D1: number analyzed (Participants) | 18 | 0
  Self-Care C32D1 | 0.06 (0.54) |
  Self-Care C33D1: number analyzed (Participants) | 15 | 0
  Self-Care C33D1 | 0.13 (0.35) |
  Self-Care C34D1: number analyzed (Participants) | 12 | 0
  Self-Care C34D1 | 0.08 (0.29) |
  Self-Care C35D1: number analyzed (Participants) | 13 | 0
  Self-Care C35D1 | 0.08 (0.28) |
  Self-Care C36D1: number analyzed (Participants) | 12 | 0
  Self-Care C36D1 | 0.08 (0.29) |
  Self-Care C37D1: number analyzed (Participants) | 11 | 0
  Self-Care C37D1 | 0.27 (0.47) |
  Self-Care C38D1: number analyzed (Participants) | 10 | 0
  Self-Care C38D1 | 0.20 (0.42) |
  Self-Care C39D1: number analyzed (Participants) | 9 | 0
  Self-Care C39D1 | 0.22 (0.67) |
  Self-Care 30 day follow up: number analyzed (Participants) | 58 | 78
  Self-Care 30 day follow up | 0.34 (0.89) | 0.38 (0.81)
  Self-Care 90 day follow up: number analyzed (Participants) | 63 | 80
  Self-Care 90 day follow up | 0.30 (0.82) | 0.25 (0.82)
  Usual Activities Baseline | 1.40 (0.72) | 1.49 (0.81)
  Usual Activities C2D1: number analyzed (Participants) | 208 | 218
  Usual Activities C2D1 | 0.08 (0.81) | 0.06 (0.86)
  Usual Activities C3D1: number analyzed (Participants) | 183 | 198
  Usual Activities C3D1 | 0.02 (0.66) | 0.04 (0.77)
  Usual Activities C4D1: number analyzed (Participants) | 169 | 171
  Usual Activities C4D1 | 0.01 (0.76) | -0.01 (0.78)
  Usual Activities C5D1: number analyzed (Participants) | 159 | 167
  Usual Activities C5D1 | 0.10 (0.86) | 0.01 (0.89)
  Usual Activities C6D1: number analyzed (Participants) | 149 | 147
  Usual Activities C6D1 | 0.05 (0.71) | -0.03 (0.81)
  Usual Activities C7D1: number analyzed (Participants) | 121 | 127
  Usual Activities C7D1 | 0.05 (0.81) | -0.01 (0.83)
  Usual Activities C8D1: number analyzed (Participants) | 109 | 111
  Usual Activities C8D1 | 0.19 (0.76) | 0.07 (0.82)
  Usual Activities C9D1: number analyzed (Participants) | 102 | 104
  Usual Activities C9D1 | 0.19 (0.78) | -0.03 (0.82)
  Usual Activities C10D1: number analyzed (Participants) | 85 | 80
  Usual Activities C10D1 | 0.06 (0.75) | 0.03 (0.89)
  Usual Activities C11D1: number analyzed (Participants) | 81 | 72
  Usual Activities C11D1 | 0.11 (0.72) | -0.04 (0.74)
  Usual Activities C12D1: number analyzed (Participants) | 75 | 58
  Usual Activities C12D1 | 0.04 (0.71) | -0.03 (0.94)
  Usual Activities C13D1: number analyzed (Participants) | 60 | 49
  Usual Activities C13D1 | 0.02 (0.79) | 0.02 (0.80)
  Usual Activities C14D1: number analyzed (Participants) | 56 | 45
  Usual Activities C14D1 | 0.02 (0.73) | 0.00 (0.64)
  Usual Activities C15D1: number analyzed (Participants) | 51 | 37
  Usual Activities C15D1 | 0.10 (0.67) | -0.14 (0.67)
  Usual Activities C16D1: number analyzed (Participants) | 48 | 32
  Usual Activities C16D1 | 0.04 (0.65) | -0.06 (0.56)
  Usual Activities C17D1: number analyzed (Participants) | 43 | 26
  Usual Activities C17D1 | 0.00 (0.65) | -0.08 (0.63)
  Usual Activities C18D1: number analyzed (Participants) | 41 | 22
  Usual Activities C18D1 | 0.15 (0.57) | -0.14 (0.77)
  Usual Activities C19D1: number analyzed (Participants) | 40 | 21
  Usual Activities C19D1 | 0.13 (0.61) | -0.38 (0.67)
  Usual Activities C20D1: number analyzed (Participants) | 39 | 20
  Usual Activities C20D1 | 0.13 (0.57) | -0.25 (0.79)
  Usual Activities C21D1: number analyzed (Participants) | 36 | 21
  Usual Activities C21D1 | 0.17 (0.51) | -0.24 (0.70)
  Usual Activities C22D1: number analyzed (Participants) | 31 | 18
  Usual Activities C22D1 | 0.06 (0.44) | -0.22 (0.65)
  Usual Activities C23D1: number analyzed (Participants) | 31 | 17
  Usual Activities C23D1 | 0.06 (0.51) | -0.24 (0.66)
  Usual Activities C24D1: number analyzed (Participants) | 29 | 13
  Usual Activities C24D1 | 0.17 (0.47) | -0.38 (0.87)
  Usual Activities C25D1: number analyzed (Participants) | 28 | 13
  Usual Activities C25D1 | 0.25 (0.52) | -0.15 (0.99)
  Usual Activities C26D1: number analyzed (Participants) | 26 | 10
  Usual Activities C26D1 | 0.12 (0.43) | -0.30 (0.67)
  Usual Activities C27D1: number analyzed (Participants) | 25 | 11
  Usual Activities C27D1 | 0.12 (0.44) | -0.36 (0.67)
  Usual Activities C28D1: number analyzed (Participants) | 21 | 11
  Usual Activities C28D1 | 0.29 (0.56) | -0.18 (0.75)
  Usual Activities C29D1: number analyzed (Participants) | 22 | 12
  Usual Activities C29D1 | 0.14 (0.56) | -0.33 (0.65)
  Usual Activities C30D1: number analyzed (Participants) | 20 | 0
  Usual Activities C30D1 | 0.15 (0.59) |
  Usual Activities C31D1: number analyzed (Participants) | 20 | 0
  Usual Activities C31D1 | 0.05 (0.51) |
  Usual Activities C32D1: number analyzed (Participants) | 18 | 0
  Usual Activities C32D1 | 0.11 (0.76) |
  Usual Activities C33D1: number analyzed (Participants) | 15 | 0
  Usual Activities C33D1 | -0.07 (0.59) |
  Usual Activities C34D1: number analyzed (Participants) | 12 | 0
  Usual Activities C34D1 | -0.08 (0.67) |
  Usual Activities C35D1: number analyzed (Participants) | 13 | 0
  Usual Activities C35D1 | 0.08 (0.86) |
  Usual Activities C36D1: number analyzed (Participants) | 12 | 0
  Usual Activities C36D1 | -0.08 (0.67) |
  Usual Activities C37D1: number analyzed (Participants) | 11 | 0
  Usual Activities C37D1 | 0.00 (0.77) |
  Usual Activities C38D1: number analyzed (Participants) | 10 | 0
  Usual Activities C38D1 | 0.10 (0.57) |
  Usual Activities C39D1: number analyzed (Participants) | 9 | 0
  Usual Activities C39D1 | 0.22 (0.44) |
  Usual Activities 30 day follow up: number analyzed (Participants) | 58 | 78
  Usual Activities 30 day follow up | 0.57 (1.16) | 0.40 (0.93)
  Usual Activities 90 day follow up: number analyzed (Participants) | 63 | 80
  Usual Activities 90 day follow up | 0.41 (0.87) | 0.29 (0.94)
  Pain/Discomfort Baseline | 1.86 (0.86) | 1.84 (0.84)
  Pain/Discomfort C2D1: number analyzed (Participants) | 208 | 218
  Pain/Discomfort C2D1 | -0.17 (0.86) | -0.13 (0.88)
  Pain/Discomfort C3D1: number analyzed (Participants) | 183 | 198
  Pain/Discomfort C3D1 | -0.21 (0.76) | -0.16 (0.75)
  Pain/Discomfort C4D1: number analyzed (Participants) | 169 | 171
  Pain/Discomfort C4D1 | -0.26 (0.87) | -0.29 (0.91)
  Pain/Discomfort C5D1: number analyzed (Participants) | 159 | 167
  Pain/Discomfort C5D1 | -0.23 (0.87) | -0.26 (0.90)
  Pain/Discomfort C6D1: number analyzed (Participants) | 149 | 147
  Pain/Discomfort C6D1 | -0.18 (0.82) | -0.22 (0.99)
  Pain/Discomfort C7D1: number analyzed (Participants) | 121 | 127
  Pain/Discomfort C7D1 | -0.26 (0.87) | -0.20 (0.83)
  Pain/Discomfort C8D1: number analyzed (Participants) | 109 | 111
  Pain/Discomfort C8D1 | -0.23 (0.86) | -0.19 (0.89)
  Pain/Discomfort C9D1: number analyzed (Participants) | 102 | 104
  Pain/Discomfort C9D1 | -0.14 (0.75) | -0.18 (0.86)
  Pain/Discomfort C10D1: number analyzed (Participants) | 85 | 80
  Pain/Discomfort C10D1 | -0.19 (0.87) | -0.18 (0.91)
  Pain/Discomfort C11D1: number analyzed (Participants) | 81 | 72
  Pain/Discomfort C11D1 | -0.28 (0.93) | -0.11 (0.96)
  Pain/Discomfort C12D1: number analyzed (Participants) | 75 | 58
  Pain/Discomfort C12D1 | -0.19 (0.83) | -0.09 (0.90)
  Pain/Discomfort C13D1: number analyzed (Participants) | 60 | 49
  Pain/Discomfort C13D1 | -0.25 (0.84) | 0.04 (0.89)
  Pain/Discomfort C14D1: number analyzed (Participants) | 56 | 45
  Pain/Discomfort C14D1 | -0.36 (0.82) | -0.02 (0.78)
  Pain/Discomfort C15D1: number analyzed (Participants) | 51 | 37
  Pain/Discomfort C15D1 | -0.27 (0.80) | 0.00 (0.88)
  Pain/Discomfort C16D1: number analyzed (Participants) | 48 | 32
  Pain/Discomfort C16D1 | -0.35 (0.86) | -0.03 (0.86)
  Pain/Discomfort C17D1: number analyzed (Participants) | 43 | 26
  Pain/Discomfort C17D1 | -0.26 (0.73) | 0.08 (0.98)
  Pain/Discomfort C18D1: number analyzed (Participants) | 41 | 22
  Pain/Discomfort C18D1 | -0.15 (0.69) | 0.00 (0.93)
  Pain/Discomfort C19D1: number analyzed (Participants) | 40 | 21
  Pain/Discomfort C19D1 | -0.15 (0.80) | -0.05 (0.50)
  Pain/Discomfort C20D1: number analyzed (Participants) | 39 | 20
  Pain/Discomfort C20D1 | -0.05 (0.72) | -0.15 (0.99)
  Pain/Discomfort C21D1: number analyzed (Participants) | 36 | 21
  Pain/Discomfort C21D1 | -0.22 (0.72) | -0.05 (0.80)
  Pain/Discomfort C22D1: number analyzed (Participants) | 31 | 18
  Pain/Discomfort C22D1 | -0.16 (0.78) | -0.28 (0.89)
  Pain/Discomfort C23D1: number analyzed (Participants) | 31 | 17
  Pain/Discomfort C23D1 | -0.16 (0.73) | -0.18 (1.01)
  Pain/Discomfort C24D1: number analyzed (Participants) | 29 | 13
  Pain/Discomfort C24D1 | -0.14 (0.79) | 0.00 (1.08)
  Pain/Discomfort C25D1: number analyzed (Participants) | 28 | 13
  Pain/Discomfort C25D1 | -0.14 (0.85) | 0.00 (1.08)
  Pain/Discomfort C26D1: number analyzed (Participants) | 26 | 10
  Pain/Discomfort C26D1 | -0.19 (0.75) | 0.20 (0.63)
  Pain/Discomfort C27D1: number analyzed (Participants) | 25 | 11
  Pain/Discomfort C27D1 | -0.16 (0.80) | 0.00 (0.45)
  Pain/Discomfort C28D1: number analyzed (Participants) | 21 | 11
  Pain/Discomfort C28D1 | -0.29 (0.85) | 0.18 (0.75)
  Pain/Discomfort C29D1: number analyzed (Participants) | 22 | 12
  Pain/Discomfort C29D1 | -0.14 (0.77) | -0.08 (0.67)
  Pain/Discomfort C30D1: number analyzed (Participants) | 20 | 0
  Pain/Discomfort C30D1 | -0.30 (0.73) |
  Pain/Discomfort C31D1: number analyzed (Participants) | 20 | 0
  Pain/Discomfort C31D1 | -0.40 (0.68) |
  Pain/Discomfort C32D1: number analyzed (Participants) | 18 | 0
  Pain/Discomfort C32D1 | -0.33 (0.84) |
  Pain/Discomfort C33D1: number analyzed (Participants) | 15 | 0
  Pain/Discomfort C33D1 | -0.40 (0.74) |
  Pain/Discomfort C34D1: number analyzed (Participants) | 12 | 0
  Pain/Discomfort C34D1 | -0.33 (0.78) |
  Pain/Discomfort C35D1: number analyzed (Participants) | 13 | 0
  Pain/Discomfort C35D1 | -0.23 (0.60) |
  Pain/Discomfort C36D1: number analyzed (Participants) | 12 | 0
  Pain/Discomfort C36D1 | -0.42 (0.67) |
  Pain/Discomfort C37D1: number analyzed (Participants) | 11 | 0
  Pain/Discomfort C37D1 | -0.27 (0.65) |
  Pain/Discomfort C38D1: number analyzed (Participants) | 10 | 0
  Pain/Discomfort C38D1 | -0.30 (0.95) |
  Pain/Discomfort C39D1: number analyzed (Participants) | 9 | 0
  Pain/Discomfort C39D1 | -0.44 (0.53) |
  Pain/Discomfort 30 day follow up: number analyzed (Participants) | 58 | 78
  Pain/Discomfort 30 day follow up | 0.29 (1.14) | 0.32 (0.95)
  Pain/Discomfort 90 day follow up: number analyzed (Participants) | 63 | 80
  Pain/Discomfort 90 day follow up | -0.03 (0.92) | 0.10 (0.94)
  Anxiety/Depression Baseline | 1.65 (0.82) | 1.64 (0.77)
  Anxiety/Depression C2D1: number analyzed (Participants) | 208 | 218
  Anxiety/Depression C2D1 | -0.01 (0.83) | -0.11 (0.79)
  Anxiety/Depression C3D1: number analyzed (Participants) | 183 | 198
  Anxiety/Depression C3D1 | -0.05 (0.68) | -0.01 (0.88)
  Anxiety/Depression C4D1: number analyzed (Participants) | 169 | 171
  Anxiety/Depression C4D1 | -0.04 (0.74) | -0.08 (0.89)
  Anxiety/Depression C5D1: number analyzed (Participants) | 159 | 167
  Anxiety/Depression C5D1 | -0.08 (0.77) | -0.07 (0.98)
  Anxiety/Depression C6D1: number analyzed (Participants) | 149 | 147
  Anxiety/Depression C6D1 | -0.07 (0.75) | 0.00 (0.88)
  Anxiety/Depression C7D1: number analyzed (Participants) | 121 | 127
  Anxiety/Depression C7D1 | -0.04 (0.80) | -0.04 (0.86)
  Anxiety/Depression C8D1: number analyzed (Participants) | 109 | 111
  Anxiety/Depression C8D1 | -0.02 (0.77) | 0.06 (0.83)
  Anxiety/Depression C9D1: number analyzed (Participants) | 102 | 104
  Anxiety/Depression C9D1 | -0.05 (0.81) | 0.03 (0.83)
  Anxiety/Depression C10D1: number analyzed (Participants) | 85 | 80
  Anxiety/Depression C10D1 | -0.13 (0.84) | 0.13 (0.86)
  Anxiety/Depression C11D1: number analyzed (Participants) | 81 | 72
  Anxiety/Depression C11D1 | -0.11 (0.81) | 0.21 (0.98)
  Anxiety/Depression C12D1: number analyzed (Participants) | 75 | 58
  Anxiety/Depression C12D1 | -0.11 (0.83) | 0.17 (0.99)
  Anxiety/Depression C13D1: number analyzed (Participants) | 60 | 49
  Anxiety/Depression C13D1 | -0.12 (0.74) | 0.20 (0.87)
  Anxiety/Depression C14D1: number analyzed (Participants) | 56 | 45
  Anxiety/Depression C14D1 | -0.07 (0.78) | 0.22 (0.85)
  Anxiety/Depression C15D1: number analyzed (Participants) | 51 | 37
  Anxiety/Depression C15D1 | -0.02 (0.62) | 0.19 (0.84)
  Anxiety/Depression C16D1: number analyzed (Participants) | 48 | 32
  Anxiety/Depression C16D1 | 0.00 (0.71) | 0.06 (0.62)
  Anxiety/Depression C17D1: number analyzed (Participants) | 43 | 26
  Anxiety/Depression C17D1 | 0.05 (0.72) | 0.15 (0.67)
  Anxiety/Depression C18D1: number analyzed (Participants) | 41 | 22
  Anxiety/Depression C18D1 | 0.12 (0.78) | 0.00 (0.69)
  Anxiety/Depression C19D1: number analyzed (Participants) | 40 | 21
  Anxiety/Depression C19D1 | -0.10 (0.78) | -0.05 (0.38)
  Anxiety/Depression C20D1: number analyzed (Participants) | 39 | 20
  Anxiety/Depression C20D1 | -0.03 (0.71) | 0.05 (0.60)
  Anxiety/Depression C21D1: number analyzed (Participants) | 36 | 21
  Anxiety/Depression C21D1 | -0.03 (0.84) | -0.05 (0.59)
  Anxiety/Depression C22D1: number analyzed (Participants) | 31 | 18
  Anxiety/Depression C22D1 | -0.10 (0.54) | 0.17 (0.71)
  Anxiety/Depression C23D1: number analyzed (Participants) | 31 | 17
  Anxiety/Depression C23D1 | -0.03 (0.71) | 0.18 (0.95)
  Anxiety/Depression C24D1: number analyzed (Participants) | 29 | 13
  Anxiety/Depression C24D1 | -0.10 (0.62) | 0.00 (0.58)
  Anxiety/Depression C25D1: number analyzed (Participants) | 28 | 13
  Anxiety/Depression C25D1 | 0.11 (1.03) | 0.15 (0.55)
  Anxiety/Depression C26D1: number analyzed (Participants) | 26 | 10
  Anxiety/Depression C26D1 | 0.00 (0.80) | 0.20 (0.42)
  Anxiety/Depression C27D1: number analyzed (Participants) | 25 | 11
  Anxiety/Depression C27D1 | 0.00 (1.04) | 0.09 (0.30)
  Anxiety/Depression C28D1: number analyzed (Participants) | 21 | 11
  Anxiety/Depression C28D1 | 0.14 (1.06) | 0.09 (0.30)
  Anxiety/Depression C29D1: number analyzed (Participants) | 22 | 12
  Anxiety/Depression C29D1 | -0.09 (0.97) | 0.25 (0.45)
  Anxiety/Depression C30D1: number analyzed (Participants) | 20 | 0
  Anxiety/Depression C30D1 | -0.10 (0.85) |
  Anxiety/Depression C31D1: number analyzed (Participants) | 20 | 0
  Anxiety/Depression C31D1 | 0.00 (1.08) |
  Anxiety/Depression C32D1: number analyzed (Participants) | 18 | 0
  Anxiety/Depression C32D1 | -0.17 (0.86) |
  Anxiety/Depression C33D1: number analyzed (Participants) | 15 | 0
  Anxiety/Depression C33D1 | -0.07 (0.88) |
  Anxiety/Depression C34D1: number analyzed (Participants) | 12 | 0
  Anxiety/Depression C34D1 | -0.42 (0.51) |
  Anxiety/Depression C35D1: number analyzed (Participants) | 13 | 0
  Anxiety/Depression C35D1 | -0.23 (0.60) |
  Anxiety/Depression C36D1: number analyzed (Participants) | 12 | 0
  Anxiety/Depression C36D1 | -0.25 (0.45) |
  Anxiety/Depression C37D1: number analyzed (Participants) | 11 | 0
  Anxiety/Depression C37D1 | -0.45 (0.52) |
  Anxiety/Depression C38D1: number analyzed (Participants) | 10 | 0
  Anxiety/Depression C38D1 | -0.60 (0.84) |
  Anxiety/Depression C39D1: number analyzed (Participants) | 9 | 0
  Anxiety/Depression C39D1 | -0.11 (0.60) |
  Anxiety/Depression 30 day follow up: number analyzed (Participants) | 58 | 78
  Anxiety/Depression 30 day follow up | 0.41 (1.27) | 0.45 (1.00)
  Anxiety/Depression 90 day follow up: number analyzed (Participants) | 63 | 80
  Anxiety/Depression 90 day follow up | 0.10 (0.76) | 0.24 (1.00)
  Visual Analog Scale Baseline | 71.50 (19.60) | 72.65 (18.73)
  Visual Analog Scale C2D1: number analyzed (Participants) | 208 | 218
  Visual Analog Scale C2D1 | 3.01 (15.83) | 1.67 (13.60)
  Visual Analog Scale C3D1: number analyzed (Participants) | 183 | 198
  Visual Analog Scale C3D1 | 2.17 (15.19) | 2.07 (14.70)
  Visual Analog Scale C4D1: number analyzed (Participants) | 169 | 171
  Visual Analog Scale C4D1 | 3.89 (16.60) | 3.27 (18.37)
  Visual Analog Scale C5D1: number analyzed (Participants) | 159 | 167
  Visual Analog Scale C5D1 | 1.50 (17.20) | 3.74 (17.32)
  Visual Analog Scale C6D1: number analyzed (Participants) | 149 | 147
  Visual Analog Scale C6D1 | 1.18 (17.61) | 1.95 (15.93)
  Visual Analog Scale C7D1: number analyzed (Participants) | 121 | 127
  Visual Analog Scale C7D1 | 3.21 (15.60) | 2.73 (19.74)
  Visual Analog Scale C8D1: number analyzed (Participants) | 109 | 111
  Visual Analog Scale C8D1 | 3.22 (19.72) | 1.73 (17.82)
  Visual Analog Scale C9D1: number analyzed (Participants) | 102 | 104
  Visual Analog Scale C9D1 | 0.96 (17.32) | 2.49 (18.01)
  Visual Analog Scale C10D1: number analyzed (Participants) | 85 | 80
  Visual Analog Scale C10D1 | 2.88 (20.07) | 1.48 (17.73)
  Visual Analog Scale C11D1: number analyzed (Participants) | 81 | 72
  Visual Analog Scale C11D1 | -1.12 (18.13) | 1.50 (18.57)
  Visual Analog Scale C12D1: number analyzed (Participants) | 75 | 58
  Visual Analog Scale C12D1 | 2.89 (21.70) | 1.36 (24.31)
  Visual Analog Scale C13D1: number analyzed (Participants) | 60 | 49
  Visual Analog Scale C13D1 | 4.30 (17.81) | 0.88 (20.52)
  Visual Analog Scale C14D1: number analyzed (Participants) | 56 | 45
  Visual Analog Scale C14D1 | 5.68 (25.25) | 2.20 (23.17)
  Visual Analog Scale C15D1: number analyzed (Participants) | 51 | 37
  Visual Analog Scale C15D1 | 4.61 (23.63) | -1.84 (19.58)
  Visual Analog Scale C16D1: number analyzed (Participants) | 48 | 32
  Visual Analog Scale C16D1 | 2.40 (18.26) | 3.44 (25.37)
  Visual Analog Scale C17D1: number analyzed (Participants) | 43 | 26
  Visual Analog Scale C17D1 | 6.07 (24.08) | 2.35 (13.65)
  Visual Analog Scale C18D1: number analyzed (Participants) | 41 | 22
  Visual Analog Scale C18D1 | 8.49 (24.62) | 4.59 (12.68)
  Visual Analog Scale C19D1: number analyzed (Participants) | 40 | 21
  Visual Analog Scale C19D1 | 5.08 (21.11) | 5.95 (10.28)
  Visual Analog Scale C20D1: number analyzed (Participants) | 39 | 20
  Visual Analog Scale C20D1 | 2.97 (25.52) | 4.15 (14.14)
  Visual Analog Scale C21D1: number analyzed (Participants) | 36 | 21
  Visual Analog Scale C21D1 | 0.69 (19.39) | 6.29 (10.93)
  Visual Analog Scale C22D1: number analyzed (Participants) | 31 | 18
  Visual Analog Scale C22D1 | 3.55 (15.24) | 3.28 (13.40)
  Visual Analog Scale C23D1: number analyzed (Participants) | 31 | 17
  Visual Analog Scale C23D1 | 3.55 (14.93) | 4.12 (16.03)
  Visual Analog Scale C24D1: number analyzed (Participants) | 29 | 13
  Visual Analog Scale C24D1 | 5.17 (16.19) | 6.85 (14.15)
  Visual Analog Scale C25D1: number analyzed (Participants) | 28 | 13
  Visual Analog Scale C25D1 | 1.43 (20.29) | 7.15 (12.08)
  Visual Analog Scale C26D1: number analyzed (Participants) | 26 | 10
  Visual Analog Scale C26D1 | 4.15 (16.83) | 1.20 (12.84)
  Visual Analog Scale C27D1: number analyzed (Participants) | 25 | 11
  Visual Analog Scale C27D1 | 0.20 (20.58) | 4.73 (4.82)
  Visual Analog Scale C28D1: number analyzed (Participants) | 21 | 11
  Visual Analog Scale C28D1 | 2.90 (18.30) | 2.36 (6.02)
  Visual Analog Scale C29D1: number analyzed (Participants) | 22 | 12
  Visual Analog Scale C29D1 | 3.73 (15.74) | 3.58 (5.95)
  Visual Analog Scale C30D1: number analyzed (Participants) | 20 | 0
  Visual Analog Scale C30D1 | 0.75 (15.87) |
  Visual Analog Scale C31D1: number analyzed (Participants) | 20 | 0
  Visual Analog Scale C31D1 | 1.60 (16.83) |
  Visual Analog Scale C32D1: number analyzed (Participants) | 18 | 0
  Visual Analog Scale C32D1 | 2.00 (15.78) |
  Visual Analog Scale C33D1: number analyzed (Participants) | 15 | 0
  Visual Analog Scale C33D1 | 6.80 (17.07) |
  Visual Analog Scale C34D1: number analyzed (Participants) | 12 | 0
  Visual Analog Scale C34D1 | 8.33 (17.91) |
  Visual Analog Scale C35D1: number analyzed (Participants) | 13 | 0
  Visual Analog Scale C35D1 | 5.77 (16.63) |
  Visual Analog Scale C36D1: number analyzed (Participants) | 12 | 0
  Visual Analog Scale C36D1 | 4.17 (17.20) |
  Visual Analog Scale C37D1: number analyzed (Participants) | 11 | 0
  Visual Analog Scale C37D1 | 10.73 (14.55) |
  Visual Analog Scale C38D1: number analyzed (Participants) | 10 | 0
  Visual Analog Scale C38D1 | 7.10 (17.70) |
  Visual Analog Scale C39D1: number analyzed (Participants) | 9 | 0
  Visual Analog Scale C39D1 | 10.22 (11.42) |
  Visual Analog Scale 30 day follow up: number analyzed (Participants) | 58 | 78
  Visual Analog Scale 30 day follow up | -7.79 (23.72) | -8.63 (20.32)
  Visual Analog Scale 90 day follow up: number analyzed (Participants) | 63 | 80
  Visual Analog Scale 90 day follow up | -5.24 (19.73) | -4.34 (19.79)

14. Secondary Outcome: Pharmacokinetics (PK) of Zolbetuximab in Serum: Trough Concentration (Ctrough)
Description: Ctrough was defined as the predose concentration at the end of dosing interval.
Time Frame: Predose on C2D1,C5D1,C9D1,C13D1,C17D1
Population: Pharmakokinetic analysis set (PKAS) consisted of the subset of the SAF for which at least 1 zolbetuximab concentration measurement was available. Participants with available data at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms/mililiter (ug/mL)
Arm/Group | CAPOX+ Zolbetuximab
Number analyzed (Participants) | 217
micrograms/mililiter (ug/mL)
  C2D1 | 38.6 (31.3)
  C5D1: number analyzed (Participants) | 160
  C5D1 | 74.1 (51.6)
  C9D1: number analyzed (Participants) | 92
  C9D1 | 99.6 (58.2)
  C13D1: number analyzed (Participants) | 52
  C13D1 | 119.0 (55.6)
  C17D1: number analyzed (Participants) | 37
  C17D1 | 147.0 (70.5)

15. Secondary Outcome: Number of Anti-drug Antibody (ADA) Positive Participants
Description: Immunogenicity will be measured by the number of participants that are ADA positive.
Time Frame: Predose on C1D1,C2D1,C5D1,C9D1,C13D1,C17D1, 30-day follow up, 90-day Follow up
Population: Participants who were Randomized to Zolbetuximab + CAPOX Arm with at least One Valid Result for ADA
Measure: Number; unit: Participants
Arm/Group | CAPOX+ Zolbetuximab
Number analyzed (Participants) | 249
Participants
  C1D1 | 4
  C2D2: number analyzed (Participants) | 212
  C2D2 | 8
  C5D1: number analyzed (Participants) | 159
  C5D1 | 2
  C9D1: number analyzed (Participants) | 92
  C9D1 | 1
  C13D1: number analyzed (Participants) | 54
  C13D1 | 0
  C17D1: number analyzed (Participants) | 38
  C17D1 | 0
  30 Day follow up: number analyzed (Participants) | 64
  30 Day follow up | 5
  90 Day follow up: number analyzed (Participants) | 46
  90 Day follow up | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality- From the start of randomization up to 61 months and 12 days Serious and non serious adverse events- From first dose up to 61 months and 12 days
Description: SAF. Participants may have repeated in the arm groups.
Groups:
- Zolbetuximab: Participants received an IV infusion (as a minimum of 2-hour infusion) of zolbetuximab at a loading dose of 800 mg/m^2 on C1D1 followed by subsequent doses of 600 mg/m^2 every 3 weeks starting from C2D1 until participant met study treatment discontinuation criteria. Each cycle was approximately 21 days.
- Capecitabine: Participants received capecitabine orally at 1000 mg/m^2 (bid) on days 1 through 14 of each cycle until the participant met study treatment discontinuation criteria. After a maximum of 8 treatments of oxaliplatin, participants may have continued to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the participant met study treatment discontinuation criteria. Each cycle was approximately 21 days.
- Oxaliplatin: Participants received an IV infusion of oxaliplatin 130 mg/m^2 on day 1 of each cycle over 2 hours for a maximum of 8 treatments. Each cycle was approximately 21 days.
- Placebo: Participants received an IV infusion (as a minimum of 2-hour infusion) of placebo matched to zolbetuximab on C1D1 followed by subsequent doses every 3 weeks starting from C2D1 until participant met study treatment discontinuation criteria. Each cycle was approximately 21 days.
Arm/Group | Zolbetuximab | Capecitabine | Oxaliplatin | Placebo
All-Cause Mortality (participants affected / at risk) | 180/254 | 387/503 | 387/503 | 207/249
Serious Adverse Events (participants affected / at risk) | 123/254 | 249/503 | 249/503 | 126/249
Other Adverse Events (participants affected / at risk) | 249/254 | 481/503 | 481/503 | 232/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolbetuximab (N=254) | Capecitabine (N=503) | Oxaliplatin (N=503) | Placebo (N=249)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 11 (15) | 11 (15) | 6 (9)
Bone marrow infiltration (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2) | 2 (3) | 2 (3) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 3 (4) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 6 (7) | 6 (7) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 5 (5) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 10 (10) | 10 (10) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (4) | 8 (9) | 8 (9) | 5 (5)
Colitis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 17 (18) | 17 (18) | 10 (11)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 5 (5) | 5 (5) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4) | 4 (4)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 4 (6) | 4 (6) | 3 (5)
Haemorrhagic ascites (Gastrointestinal disorders) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 6 (6) | 6 (6) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 5 (5) | 5 (5) | 2 (2)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (12) | 17 (18) | 17 (18) | 6 (6)
Obstruction gastric (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oesophageal-pulmonary fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (11) | 11 (18) | 11 (18) | 4 (7)
Vomiting (Gastrointestinal disorders) | 15 (21) | 26 (35) | 26 (35) | 11 (14)
Asthenia (General disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Death (General disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Fatigue (General disorders) | 3 (3) | 6 (6) | 6 (6) | 3 (3)
Gait inability (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gravitational oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 8 (8) | 8 (8) | 3 (3)
Sudden death (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Deficiency of bile secretion (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 4 (6) | 4 (6) | 2 (4)
Liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 2 (3) | 2 (3) | 1 (2)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (4) | 2 (8) | 2 (8) | 1 (4)
COVID-19 (Infections and infestations) | 3 (3) | 6 (6) | 6 (6) | 3 (3)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (3) | 1 (3) | 1 (3)
Infection (Infections and infestations) | 2 (3) | 2 (3) | 2 (3) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Peritonitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 12 (14) | 12 (14) | 6 (8)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 3 (4) | 3 (4) | 2 (2)
Septic shock (Infections and infestations) | 2 (4) | 4 (7) | 4 (7) | 2 (3)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (3) | 1 (3) | 1 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Stoma prolapse (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (4) | 3 (6) | 3 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 4 (11) | 4 (11) | 2 (9)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (5) | 2 (5) | 1 (4)
Platelet count decreased (Investigations) | 8 (28) | 14 (48) | 14 (48) | 6 (20)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (4) | 2 (8) | 2 (8) | 1 (4)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 13 (13) | 13 (13) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (3) | 2 (5) | 2 (5) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 12 (14) | 12 (14) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 2 (3) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 23 (23) | 23 (23) | 13 (13)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (3) | 2 (3) | 2 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 5 (5) | 5 (5) | 1 (1)
Choluria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (3) | 2 (3) | 1 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 7 (12) | 7 (12) | 5 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 8 (10) | 8 (10) | 7 (7)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (11) | 10 (11) | 8 (9)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 3 (4) | 2 (3)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Embolism venous (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 5 (6) | 5 (6) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolbetuximab (N=254) | Capecitabine (N=503) | Oxaliplatin (N=503) | Placebo (N=249)
Anaemia (Blood and lymphatic system disorders) | 90 (255) | 179 (480) | 179 (480) | 89 (225)
Leukopenia (Blood and lymphatic system disorders) | 17 (41) | 25 (63) | 25 (63) | 8 (22)
Neutropenia (Blood and lymphatic system disorders) | 48 (131) | 82 (212) | 82 (212) | 34 (81)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (68) | 56 (133) | 56 (133) | 29 (65)
Abdominal distension (Gastrointestinal disorders) | 15 (21) | 29 (36) | 29 (36) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 40 (54) | 91 (120) | 91 (120) | 51 (66)
Abdominal pain upper (Gastrointestinal disorders) | 24 (37) | 37 (57) | 37 (57) | 13 (20)
Constipation (Gastrointestinal disorders) | 40 (53) | 93 (121) | 93 (121) | 53 (68)
Diarrhoea (Gastrointestinal disorders) | 79 (134) | 162 (322) | 162 (322) | 83 (188)
Nausea (Gastrointestinal disorders) | 174 (503) | 297 (786) | 297 (786) | 123 (283)
Vomiting (Gastrointestinal disorders) | 164 (463) | 236 (616) | 236 (616) | 72 (153)
Asthenia (General disorders) | 34 (67) | 65 (122) | 65 (122) | 31 (55)
Fatigue (General disorders) | 34 (64) | 74 (157) | 74 (157) | 40 (93)
Malaise (General disorders) | 30 (107) | 52 (178) | 52 (178) | 22 (71)
Oedema peripheral (General disorders) | 26 (37) | 32 (45) | 32 (45) | 6 (8)
Pyrexia (General disorders) | 32 (46) | 53 (77) | 53 (77) | 21 (31)
Alanine aminotransferase increased (Investigations) | 47 (66) | 99 (165) | 99 (165) | 52 (99)
Aspartate aminotransferase increased (Investigations) | 62 (106) | 136 (246) | 136 (246) | 74 (140)
Blood alkaline phosphatase increased (Investigations) | 14 (24) | 34 (54) | 34 (54) | 20 (30)
Blood bilirubin increased (Investigations) | 24 (69) | 47 (118) | 47 (118) | 23 (49)
Neutrophil count decreased (Investigations) | 71 (374) | 129 (635) | 129 (635) | 58 (261)
Platelet count decreased (Investigations) | 60 (185) | 121 (409) | 121 (409) | 61 (224)
Weight decreased (Investigations) | 51 (72) | 76 (104) | 76 (104) | 25 (32)
White blood cell count decreased (Investigations) | 50 (207) | 90 (377) | 90 (377) | 40 (170)
Decreased appetite (Metabolism and nutrition disorders) | 103 (195) | 188 (357) | 188 (357) | 85 (162)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 57 (136) | 92 (202) | 92 (202) | 35 (66)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (17) | 25 (37) | 25 (37) | 12 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 34 (72) | 68 (143) | 68 (143) | 34 (71)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (20) | 32 (49) | 32 (49) | 17 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 28 (36) | 28 (36) | 18 (26)
Dizziness (Nervous system disorders) | 14 (21) | 26 (37) | 26 (37) | 12 (16)
Dysgeusia (Nervous system disorders) | 18 (25) | 30 (38) | 30 (38) | 12 (13)
Hypoaesthesia (Nervous system disorders) | 31 (110) | 61 (212) | 61 (212) | 30 (102)
Neuropathy peripheral (Nervous system disorders) | 12 (18) | 25 (37) | 25 (37) | 13 (19)
Neurotoxicity (Nervous system disorders) | 14 (34) | 33 (69) | 33 (69) | 19 (35)
Peripheral sensory neuropathy (Nervous system disorders) | 57 (96) | 113 (215) | 113 (215) | 56 (119)
Insomnia (Psychiatric disorders) | 28 (36) | 46 (55) | 46 (55) | 18 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 27 (32) | 27 (32) | 15 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 25 (33) | 25 (33) | 12 (17)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 43 (67) | 92 (153) | 92 (153) | 49 (86)
Hypertension (Vascular disorders) | 15 (45) | 22 (52) | 22 (52) | 7 (7)
Ascites (Gastrointestinal disorders) | 8 (11) | 21 (33) | 21 (33) | 13 (22)
Dyspepsia (Gastrointestinal disorders) | 13 (16) | 22 (26) | 22 (26) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03653507/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03653507/SAP_001.pdf